# A Phase 2 Randomized, Open-Label, Multisite Trial to Inform Public Health Strategies Involving the Use of MVA-BN Vaccine for Mpox

**DMID Protocol Number: 22-0020** 

Sponsor: Division of Microbiology and Infectious Diseases (DMID)

**Version Number: 7.0** 

May 23, 2024

# STATEMENT OF COMPLIANCE

Each institution engaged in this research will hold a current Federalwide Assurance (FWA) issued by the Office of Human Research Protection (OHRP) for federally funded research. The IRB/IEC must be registered with OHRP as applicable to the research.

The study will be carried out in accordance with the following as applicable:

- United States Code of Federal Regulations (CFR) 45 CFR Part 46: Protection of Human Subjects
- Food and Drug Administration (FDA) Regulations: 21 CFR Part 50 (Protection of Human Subjects), 21 CFR Part 54 (Financial Disclosure by Clinical Investigators), 21 CFR Part 56 (Institutional Review Boards), 21 CFR Part 11 (Electronic Records and Electronic Signatures), and 21 CFR Part 312 (Investigational New Drug Application), and/or 21 CFR 812 (Investigational Device Exemptions)
- The International Council for Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) E6(R2) Good Clinical Practice (GCP), and the Belmont Report: Ethical Principles and Guidelines for the Protection of Human Subjects of Research, Report of the National Commission for the Protection of Human Subjects of Biomedical and Behavioral Research
- The policies and procedures of National Institutes of Health (NIH) Office of Extramural Research and DMID
- The National Institute of Allergy and Infectious Diseases (NIAID) Terms of Award
- Any additional Federal, State, and Local Regulations and Guidance

The signature below provides the necessary assurance that this study will be conducted according to all stipulations of the protocol including statements regarding confidentiality, and according to local legal and regulatory requirements, US federal regulations, and ICH E6(R2) Good Clinical Practice (GCP) guidelines.

| Site Inve | stigator Signature: | |
|-----------|-------------------------|-------|
| Signed: | | Date: |
| | Print Name, Credentials | |
| | Print Title | |

DMID/NIAID/NIH 

# TABLE OF CONTENTS

| STATEMENT OF COMPLIANCE | 2 |
|--------------------------------------------------------------|----|
| TABLE OF CONTENTS | 3 |
| LIST OF TABLES | 11 |
| LIST OF FIGURES | 11 |
| 1. PROTOCOL SUMMARY | |
| 1.1 Synopsis | |
| 1.2 Schedule of Activities (SOA) | |
| 2. Introduction | 15 |
| 2.1 Study Rationale | |
| 2.2 Background | |
| 2.3 Risk/Benefit Assessment | 18 |
| 3. OBJECTIVES AND ENDPOINTS | 18 |
| 4. STUDY DESIGN | 18 |
| 4.1 Overall Design | |
| 4.1 Overall Design 4.2 Scientific Rationale for Study Design | |
| 4.3 Justification for Dose | |
| 5. STUDY POPULATION | |
| 6. STUDY PRODUCT | |
| 6.1 Study Product(s) and Administration | 19 |
| 6.1.1 Study Product Description | |
| 6.1.2 Dosing and Administration | |
| 6.1.3 Dose Escalation | |
| 6.1.4 Dose Modifications 6.1.5 Criteria for Redosing. | |
| 6.2 Preparation/Handling/Storage/Accountability | |
| 6.2.1 Acquisition and Accountability | |
| 6.2.2 Formulation, Appearance, Packaging, and Labeling | |
| 6.2.3 Product Storage and Stability | |
| 6.2.4 Preparation | |
| 6.3 Measures to Minimize Bias: Randomization and Blinding | |
| 6.3.1 Treatment Assignment Procedures | |
| 6.3.2 Randomization | |
| 6.3.3 Blinding and Masking Procedures | |
| 6.4 Study Intervention Compliance | |
| 6.5 Concomitant Therapy | |
| 7. STUDY INTERVENTION DISCONTINUATION AND PARTICIPANT | |
| DISCONTINUATION/WITHDRAWAL | 23 |
| 8. STUDY ASSESSMENTS AND PROCEDURES | 23 |

| 8.6 Adverse Events and Serious Adverse Events | 23 |
|---|---|
| 8.6.1 Definition of Adverse Events (AE) | 23 |
| 8.6.1.1 Solicited Adverse Events | |
| 8.6.1.2 Unsolicited Events | 24 |
| 8.6.2 Definition of Serious Adverse Events | |
| 8.6.3 Classification of an Adverse Event | 25 |
| 8.6.3.1 Severity of Event | 25 |
| 8.6.3.2 Relationship to Study Intervention | 25 |
| 8.6.5 Adverse Event Reporting | |
| 8.6.5.1 Investigators Reporting of AEs | 26 |
| 8.6.5.2 Special Reporting of Adverse Events | 26 |
| 8.6.6 Serious Adverse Event Reporting | |
| 8.6.6.1 Investigators Reporting of SAEs | |
| 8.6.6.2 Regulatory Reporting of SAEs | |
| 8.6.7 Reporting Events to Participants | |
| 8.6.8 Reporting of Pregnancy | |
| 8.7 Unanticipated Problems | |
| 8.7.1 Definition of Unanticipated Problems (UP) | |
| 8.7.2 Unanticipated Problem Reporting | |
| 8.7.3 Reporting Unanticipated Problems to Participants | 29 |
| 9. STATISTICAL CONSIDERATIONS | 29 |
| 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATION | NS29 |
| 10.1 Regulatory, Ethical, and Study Oversight Considerations | 29 |
| 10.1.1 Informed Consent Process | |
| 10.1.2 Study Termination and Closure | |
| 10.1.3 Confidentiality and Privacy | |
| 10.1.4 Secondary Use of Stored Specimens and Data | |
| 10.1.4.1 Samples for Secondary Research | |
| 10.1.4.2 Data Sharing for Secondary Research | |
| 10.1.5 Key Roles and Study Governance | |
| 10.1.6 Safety Oversight | |
| 10.1.0 Builty Oversight | 32 |
| 10.1.7 Clinical Monitoring | |
| | 33 |
| 10.1.7 Clinical Monitoring | 33<br>33 |
| 10.1.7 Clinical Monitoring | 33<br>33 |
| 10.1.7 Clinical Monitoring | 33<br>33<br>33 |
| 10.1.7 Clinical Monitoring | 33<br>33<br>33<br>33 |
| 10.1.7 Clinical Monitoring | 33<br>33<br>33<br>34 |
| 10.1.7 Clinical Monitoring | 33<br>33<br>33<br>34<br>34 |
| 10.1.7 Clinical Monitoring | |
| 10.1.7 Clinical Monitoring | 33<br>33<br>34<br>34<br>34<br>34 |
| 10.1.7 Clinical Monitoring 10.1.8 Quality Assurance and Quality Control 10.1.9 Data Handling and Record Keeping 10.1.9.1 Data Collection and Management Responsibilities 10.1.9.2 Data Coordinating Center / Biostatistician Responsibilities 10.1.9.3 Data Capture Methods 10.1.9.4 Study Record Retention 10.1.9.5 Source Records 10.1.10 Protocol Deviations | |
| 10.1.7 Clinical Monitoring | |
| 10.1.7 Clinical Monitoring | |

| 10.2 Additional Considerations | 36 |
|----------------------------------------------------|----|
| 10.2.1 Research Related Injuries | |
| 10.2.2 PREP Act | |
| 10.3 Abbreviations | |
| 10.4 Protocol Amendment History | |
| 11. References | 42 |
| APPENDIX A – Stage 1: Dose Sparing Study in Adults | 46 |
| TABLE OF CONTENTS | 46 |
| LIST OF TABLES | 48 |
| LIST OF FIGURES | 49 |
| 1. PROTOCOL SUMMARY | |
| 1.1 Synopsis | 50 |
| 1.2 Schedule of Activities (SOA) | |
| 1.3 Study Schema | |
| 2. INTRODUCTION | 53 |
| 2.1 Study Rationale | 53 |
| 2.2 Background | 53 |
| 2.3 Risk/Benefit Assessment | |
| 2.3.1 Known Potential Risks | |
| 2.3.2 Known Potential Benefits | 59 |
| 2.3.3 Assessment of Potential Risks and Benefits | 59 |
| 3. OBJECTIVES AND ENDPOINTS | 60 |
| 4. STUDY DESIGN | 61 |
| 4.1 Overall Design | |
| 4.2 Scientific Rationale for Study Design | |
| 4.3 Justification for Dose | |
| 5. STUDY POPULATION | |
| 5.1 Inclusion Criteria | 62 |
| 5.2 Exclusion Criteria | |
| 5.2.1 Exclusion of Specific Populations | |
| 5.3 Inclusion of Vulnerable Participants | |
| 5.4 Lifestyle Considerations | |
| 5.5 Screen Failures | |
| 5.6 Strategies for Recruitment and Retention | 64 |
| 5.6.1 Recruitment | |
| 5.6.2 Retention | |
| 5.6.3 Compensation Plan for Participants | |
| 5.6.4 Costs | 65 |
| 6. STUDY PRODUCT | 65 |
| 6.1 Study Product(s) and Administration | 65 |

| 6.1.1 | Study Product Description | 65 |
|---|---|---|
| 6.1.2 | Dosing and Administration | 65 |
| 6.1.3 | Dose Escalation | 66 |
| 6.1.4 | Dose Modifications | 66 |
| 6.1.5 | Criteria for Redosing | 66 |
| 6.2 Pre | paration/Handling/Storage/Accountability | 66 |
| 6.2.1 | Acquisition and Accountability | |
| 6.2.2 | Formulation, Appearance, Packaging, and Labeling Product: JYNNEOS (M. | ſVA- |
| BN vacc | eine) | 67 |
| 6.2.3 | Product Storage and Stability Product: JYNNEOS (MVA-BN vaccine) | 67 |
| 6.2.4 | Preparation | 67 |
| 6.3 Me | asures to Minimize Bias: Randomization and Blinding | 68 |
| 6.3.1 | Treatment Assignment Procedures | 68 |
| 6.3.2 | Randomization | 68 |
| 6.3.3 | Blinding and Masking Procedures | 68 |
| 6.4 Stu | dy Intervention Compliance | 68 |
| 6.5 Co <sub>1</sub> | ncomitant Therapy | 68 |
| 6.5.1 | Rescue Medicine | 69 |
| 7. STUDY | INTERVENTION DISCONTINUATION AND PARTICIPANT | |
| | JATION/WITHDRAWAL | 69 |
| | ting Criteria and Discontinuation of Study Intervention | |
| 7.1.1 | | 69 |
| 7.1.1. | $\mathcal{L}$ | |
| | 2 Cohort Halting Rules | |
| 7.1.2 | <b>8</b> | |
| 7.1.3 | Follow up for participants that discontinued study intervention | |
| 7.2 Los | st to Follow-Up | 71 |
| 8. STUDY | ASSESSMENTS AND PROCEDURES | 71 |
| 8.1 Scr | eening Procedures | 71 |
| 8.1.1 | Procedures to be Followed in the Event of Abnormal Clinical Laboratory To | |
| | or Abnormal Clinical Findings During Screening | |
| 8.1.2 | Sick Visit | |
| | nunogenicity Assessments | |
| 8.2.1 | Immunogenicity/Efficacy Evaluations | |
| 8.2.2 | Exploratory Assessments | |
| | ety and Other Assessments | |
| 8.3.1 | Procedures to be Followed in the Event of Abnormal Clinical Laboratory To | |
| | or Abnormal Clinical Findings During Conduct of the Trial | |
| | verse Events and Serious Adverse Events | |
| 8.4.1 | Definition of Adverse Events (AE) | |
| 8.4.1. | | |
| 8.4.1. | | |
| 8.4.2 | Definition of Serious Adverse Events | |
| 8.4.2. | | |
| 8.4.2. | | |
| 0.7.2. | 2 Definition of Suspected Schenpetted School Reverse Redections (BOSAN | ., / C |

| 8.4.3 | Classification of an Adverse Event | 76 |
|---|---|---|
| 8.4.3.1 | Severity of Event | 76 |
| 8.4.3.2 | Relationship to Study Intervention | 77 |
| 8.4.4 | Time Period and Frequency for Event Assessment and Follow-Up | 77 |
| 8.4.5 | Adverse Event Reporting | 78 |
| 8.4.5.1 | Investigators Reporting of AEs | 78 |
| 8.4.5.2 | Special Reporting of Adverse Events | 78 |
| 8.4.6 | Serious Adverse Event Reporting | 78 |
| 8.4.6.1 | Investigators Reporting of SAEs | 78 |
| 8.4.6.2 | Regulatory Reporting of SAEs | 79 |
| 8.4.7 | Reporting Events to Participants | 79 |
| 8.4.8 | Adverse Events of Special Interest (AESI) | 80 |
| 8.4.9 | Reporting of Pregnancy | 80 |
| 8.5 Una | nticipated Problems | 80 |
| 8.5.1 | Definition of Unanticipated Problems (UP) | 80 |
| 8.5.2 | Unanticipated Problem Reporting | |
| 8.5.3 | Reporting Unanticipated Problems to Participants | 81 |
| 9. STATIST | ICAL CONSIDERATIONS | |
| | stical Hypotheses | |
| | ple Size Determination | |
| | stical Analyses | |
| 9.3.1 | General Methodology | |
| | Timing of Analyses | |
| 9.3.2.1 | | |
| 9.3.2.2<br>9.3.2.3 | | |
| 9.3.2.3 | · | |
| 9.3.3 | Populations for Analyses. | |
| 9.3.4 | Baseline Characteristics and Participant Disposition | |
| 9.3.5 | Immunogenicity Analyses | |
| 9.3.6.1 | | |
| | Other Adverse Events | |
| 10. SUPPOR | TING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | 86 |
| 10.1 Reg | ulatory, Ethical, and Study Oversight Considerations | 86 |
| 10.1.1 | Informed Consent Process. | |
| 10.1.1. | | |
| (in case | e of a minor) | |
| 10.1.1. | , | |
| 10.1.2 | Study Termination and Closure | |
| 10.1.3 | Confidentiality and Privacy | |
| 10.1.4 | Secondary Use of Stored Specimens and Data | |
| 10.1.4. | | |
| 10.1.4. | | |
| 10.1.5 | Key Roles and Study Governance | |
| 10.1.6 | Safety Oversight | |

| 10.1.7 Clinical Monitoring | 92 |
|------------------------------------------------------------------|-----|
| 10.1.8 Quality Assurance and Quality Control | |
| 10.1.9 Data Handling and Record Keeping | 93 |
| 10.1.9.1 Data Collection and Management Responsibilities | |
| 10.1.9.2 Data Coordinating Center / Biostatistician Responsibili | |
| 10.1.9.3 Data Capture Methods | |
| 10.1.9.4 Study Record Retention | |
| 10.1.9.5 Source Records | |
| 10.1.10 Protocol Deviations | |
| 10.1.11 Publication and Data Sharing Policy | |
| 10.1.11.1 Human Data Sharing Plan | |
| 10.1.11.2 Genomic Data Sharing Plan | |
| 10.1.11.3 Publication | |
| 10.1.12 Conflict of Interest Policy | |
| 10.2 Additional Considerations | |
| 10.2.2 PREP Act | |
| 11. REFERENCES | 97 |
| APPENDIX B – Stage 2: Adolescent and Adult Noninferiority Study | 99 |
| TABLE OF CONTENTS | |
| 1. Introduction | 103 |
| 1.1 Study Rationale | 103 |
| 1.2 Background | |
| 1.3 Risk/Benefit Assessment | |
| 1.3.1 Known Potential Risks | 104 |
| 1.3.2 Known Potential Benefits | 107 |
| 1.3.3 Assessment of Potential Risks and Benefits | 108 |
| 2. OBJECTIVES AND ENDPOINTS | 108 |
| 3. STUDY DESIGN | 109 |
| 3.1 Overall Design | 109 |
| 3.2 Scientific Rationale for Study Design | |
| 3.3 Justification for Dose | 111 |
| 4. STUDY POPULATION | 111 |
| 4.1 Inclusion Criteria | |
| 4.2 Exclusion Criteria | |
| 4.2.1 Exclusion of Specific Populations | |
| 4.3 Inclusion of Vulnerable Participants | |
| 4.4 Lifestyle Considerations | |
| 4.5 Screen Failures | |
| 4.6 Strategies for Recruitment and Retention | |
| 4.6.2 Retention | 113 |

| _ | 4.6.4 | Compensation Plan for Participants | |
|---|---|---|---|
| _ | | 0000 | 110 |
| 5. | STUDY I | PRODUCT | 116 |
| 5. | .1 Stuc | ly Product(s) and Administration | 116 |
| ٠. | 5.1.1 | Study Product Description | |
| | 5.1.2 | Dosing and Administration | |
| | 5.1.3 | Dose Escalation. | |
| | 5.1.4 | Dose Modifications. | |
| | 5.1.5 | Criteria for Redosing. | |
| 5. | | paration/Handling/Storage/Accountability | |
| | 5.2.1 | Acquisition and Accountability | |
| | 5.2.2 | Formulation, Appearance, Packaging, and Labeling | |
| | 5.2.3 | Product Storage and Stability | |
| | 5.2.4 | Preparation | |
| 5. | .3 Mea | sures to Minimize Bias: Randomization and Blinding | 118 |
| | 5.3.1 | Treatment Assignment Procedures | |
| | 5.3.2 | Randomization | 118 |
| | 5.3.3 | Blinding and Masking Procedures | 118 |
| 5. | .4 Stud | ly Intervention Compliance | 118 |
| 5. | .5 Con | comitant Therapy | 118 |
| 6. | STUDY 1 | NTERVENTION DISCONTINUATION AND PARTICIPANT | |
| | | VATION/WITHDRAWAL | 119 |
| 6. | .1 Halt | ing Criteria and Discontinuation of Study Intervention | 119 |
| | 6.1.1 | Study Halting Criteria | |
| | 6.1.1.1 | | |
| | 6.1.1.2 | | |
| | 6.1.2 | Individual Halting Criteria | |
| _ | 6.1.3 | Follow up for participants that discontinued study intervention | |
| | | icipant Withdrawal from the Study and Replacement | |
| 6. | .5 Los | t to Follow-Up | 121 |
| 7. | STUDY A | ASSESSMENTS AND PROCEDURES | 121 |
| 7. | 1 Scre | eening Procedures | 121 |
| | 7.1.1 | Procedures to be Followed in the Event of Abnormal Clinical Laborat | |
| | | r Abnormal Clinical Findings During Screening | • |
| 7. | | Visit | |
| 7. | | itional Study Procedures in Stage 2 | |
| | 7.3.1 | Phone Visits | |
| | 7.3.2 | Photography | |
| 7. | | nunogenicity Assessments | |
| | 7.4.1 | Immunogenicity/Efficacy Evaluations | |
| | 7.4.2 | Exploratory Assessments | |
| 7. | .5 Safe | ety and Other Assessments | |
| | 7.5.1 | Alternative Schedules | |

| 7.5.2 Procedures to be Followed in the Event of Abnormal Clinical Laboratory Test | |
|---|---|
| Values or Abnormal Clinical Findings During the Trial | 126 |
| 7.6 Adverse Events and Serious Adverse Events | |
| 7.6.1.1 Definition of Medically Attended Adverse Events (MAAE) | |
| 7.6.1.2 Definition of Suspected Unexpected Serious Adverse Reactions (SUSAR) | 126 |
| 7.6.1.3 Definition of Adverse Event of Special Interest (AESI) | 126 |
| 7.6.2 Classification of an Adverse Event | |
| See main section of the protocol for a description of the classification of an AE in terms | |
| severity and causality. | |
| 7.6.3 Time Period and Frequency for Event Assessment and Follow-Up | |
| 7.6.4 Adverse Event Reporting | |
| 7.7 Unanticipated Problems | 127 |
| 8. STATISTICAL CONSIDERATIONS | . 127 |
| 8.1 Statistical Hypotheses | 127 |
| 8.2 Sample Size Determination | |
| 8.3 Statistical Analyses | |
| 8.3.1 General Methodology | 130 |
| 8.3.2 Timing of Analyses | 130 |
| 8.3.2.1 Interim Safety Analyses | 130 |
| 8.3.2.2 Interim Immunogenicity Analyses | 130 |
| 8.3.2.3 Final Analyses | 130 |
| 8.3.3 Populations for Analyses | 131 |
| 8.3.4 Baseline Characteristics and Participant Disposition | 131 |
| 8.3.5 Immunogenicity Analyses | 131 |
| 8.3.6 Safety Analyses | 132 |
| 8.3.6.1 Reactogenicity | 132 |
| 8.3.6.2 Other Adverse Events | 132 |
| 9. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | . 133 |
| 9.1 Regulatory, Ethical, and Study Oversight Considerations | 133 |
| 9.1.1 Informed Consent Process | |
| 9.1.1.1 Requirements for Permission by Parents/LARs and Assent by Children (in | |
| of a minor) | |
| 9.1.1.2 Other Informed Consent Procedures | |
| 9.1.2 Study Termination and Closure | 136 |
| 9.1.3 Confidentiality and Privacy | 136 |
| 9.1.4 Secondary Use of Stored Specimens and Data | 137 |
| 9.1.4.1 Samples for Secondary Research | 137 |
| 9.1.4.2 Data Sharing for Secondary Research | |
| 9.1.5 Key Roles and Study Governance | |
| 9.1.6 Safety Oversight | |
| 9.1.7 Clinical Monitoring | 139 |
| 9.1.8 Quality Assurance and Quality Control | 140 |
| 9.1.9 Data Handling and Record Keeping | 140 |
| 9.1.9.1 Data Collection and Management Responsibilities | 140 |
| 9.1.9.2 Data Coordinating Center / Biostatistician Responsibilities | 140 |

| 9.1.9 | 9.3 Data Capture Methods | 140 |
|--------------|------------------------------------------------|-----|
| 9.1.9 | | 141 |
| 9.1.9 | | 141 |
| 9.1.10 | | |
| 9.1.11 | | |
| | 11.1 Human Data Sharing Plan | |
| | 11.2 Genomic Data Sharing Plan | |
| 9.1. | | |
| 9.1.12 | Conflict of Interest Policy | |
| | dditional Considerations | |
| 9.2.1 | | |
| 9.2.2 | | |
| 10. Referen | nces | 145 |
| | LIST OF TABLES | |
| Гable 1 Stu | dy Schema | 13 |
| Table 2 Prio | or Subcutaneous Dosing Trials | 16 |
| Гable 3 MV | A-BN Compared to ACAM2000 | 17 |
| | or Intradermal Dosing Compared to Subcutaneous | |
| | dy Arms | |

# LIST OF FIGURES

No table of figures entries found.

# 1. PROTOCOL SUMMARY

# 1.1 Synopsis

#### Rationale

Since the first case was identified in May of 2022 in the United Kingdom, mpox (previously known as monkeypox) has rapidly spread to more than 100 non-endemic countries, marking the first time mpox has spread widely outside Central and West Africa. In the U.S., there have been 29,630 confirmed mpox cases and 20 deaths as of December 6, 2022. To prevent further spread of mpox and to mitigate this outbreak, MVA-BN vaccine is being offered to individuals at high risk of acquiring the disease which in this outbreak include gay, bisexual, and other men who have sex with men, transgender or nonbinary people and people at occupational risk of exposure to orthopoxviruses. Post-exposure prophylaxis with JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic [MVA-BN] vaccine) is also recommended for other moderate or high-risk exposures, including in young infants, even though safety and immunogenicity data are sparse in pediatric populations. While the incidence of mpox is declining in the U.S., there is still uncertainty about when this outbreak will end and whether it will establish endemicity in high-risk groups. In addition, there is a global vaccine shortage and increasing vaccine supply will take time.

This Phase 2, open-label multi-site platform trial will evaluate strategies to inform public health decisions regarding the use of JYNNEOS for mpox prevention and mitigation of outbreaks. As JYNNEOS is also used for smallpox prophylaxis, this trial will also inform public health decisions on the use of the vaccine for smallpox. The trial is divided into stages according to public health needs and scientific priorities. Public health strategies will be evaluated in separate stages of the trial and include intradermal dose sparing strategies in adults (Stage 1) and extension of the target population for JYNNEOS to include adolescents (Stage 2). This protocol may add additional arms as needed based on public health needs and priorities. The study arms will be conducted in different stages that could overlap.

Each stage of the study will have a separate protocol in an appendix (e.g., Stage 1 is described in Appendix A, Stage 2 in Appendix B, etc.). Commonalities between the stages will be included and highlighted in this main section of this protocol.

# Stage 1

Approximately 230 healthy, vaccinia-naïve adults ages 18 to 50 years, inclusive, will be enrolled to retain 210 participants assuming a 10% drop-out rate. Participants will be randomized 1:1:1 to one of three study arms (Table 1). Participants in Arms 1 and 2 will receive a 2-dose intradermal regimen of 2x10<sup>7</sup> and 1x10<sup>7</sup> MVA-BN, respectively and Arm 3 will receive the licensed 2-dose SC regimen of 1x10<sup>8</sup> MVA-BN. All vaccines will be administered on Day 1 and 29. There will be eight study visits (plus an optional screening visit) with the last visit at approximately one year after the first study vaccination. Participants reporting mpox-like illness and who have a positive MPXV diagnostic test (laboratory-confirmed mpox case) will be seen at a sick visit. Enrollment of this Stage ended on October 13, 2022.

#### Stage 2

Approximately 315 healthy, vaccinia-naïve adolescents ages 12 to 17 years, inclusive, will be enrolled in Arm 5 to retain 300 participants assuming a 5% drop-out rate (Table 1). Approximately

DMID/NIAID/NIH 

135 healthy, vaccinia-naïve adults ages 18 to 50 years, inclusive, will be enrolled in Arm 4. These adults (Arm 4) will be combined with participants from Arm 3 (adults given subcutaneous standard dose in Stage 1) and together will be the comparator group for the primary endpoint, non-inferiority testing. Participants in Arms 4 and 5 will receive the 2-dose SC regimen of 1x10<sup>8</sup> MVA-BN. All vaccines will be administered on Day 1 and 29. There will be nine study visits (plus an optional screening visit) with the last visit at approximately one year after the second study vaccination. Participants reporting a laboratory-confirmed case of mpox will be seen at a sick visit.

**Table 1 Study Schema** 

| | Arm | N | Age in years | Dose of JYNNEOS<br>(MVA-BN) | Route of Administration* |
|---|---|---|---|---|---|
| Stage 1 | 1 | 76 | 18-50 | 2 x 10 <sup>7</sup> TCID <sub>50</sub> , (0.1 mL) | Intradermal |
| Adult | 2 | 77 | | 1 x 10 <sup>7</sup> TCID <sub>50</sub> , (0.05 mL) | Intradermal |
| | 3 | 76 | | 1 x 10 <sup>8</sup> TCID <sub>50</sub> , (0.5 mL) | Subcutaneous |
| Stage 2 | 4 | 135 | 18-50 | 1 x 10 <sup>8</sup> TCID <sub>50</sub> , (0.5 mL) | Subcutaneous |
| Adult and<br>Adolescent | 5 | 315 | 12-17 | 1 x 10 <sup>8</sup> TCID <sub>50</sub> , (0.5 mL) | Subcutaneous |

<sup>\*</sup>Subcutaneous is administered in the upper arm on Day 1 and 29. Intradermal is administered in the volar aspect (inner side) of the forearm on Day 1 and Day 29.

# **Primary Objectives:**

# Stage 1 (Adult)

- To determine if peak (Day 43) humoral immune responses in adults ages 18-50 years following an ID regimen of 2 x 10<sup>7</sup> TCID<sub>50</sub> MVA-BN are non-inferior to the licensed regimen of 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN administered SC.
- To determine if peak (Day 43) humoral immune responses in adults ages 18-50 years following an ID regimen of 1 x 10<sup>7</sup> TCID<sub>50</sub> MVA-BN are non-inferior to the licensed regimen of 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN administered SC

## **Stage 2 (Adult and Adolescent)**

- To determine if peak (Day 43) humoral immune responses in adolescents ages 12 to 17 years following administration of a 2-dose 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN regimen administered SC are non-inferior to the response in adults ages 18 to 50 years who received the licensed 2-dose SC regimen of 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN.
- To describe safety of a 2-dose 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN regimen administered SC in adolescents ages 12 to 17 years.

For a full list of Objectives/Endpoints, see corresponding section of the protocol.

#### **Inclusion Criteria**

Inclusion criteria will remain relatively consistent between stages with differences only in the ability to give informed consent in pediatric populations. See inclusion criteria for each stage in corresponding section of the protocol.

DMID/NIAID/NIH 

#### **Exclusion Criteria**

Exclusion criteria will remain relatively consistent between stages with differences due to limited data on the safety profile in pediatric population. See exclusion criteria for each stage in corresponding section of the protocol.

#### **Study Phase**

Phase 2

#### **Study Population**

This platform trial will enroll a study population that is healthy, vaccinia-naïve, non-pregnant, and non-breastfeeding. Participants with stable chronic medical conditions including those with controlled HIV can participate. In Stage 1 and Stage 2, adults ages 18 to 50 years, inclusive, will be enrolled, and in Stage 2, adolescents ages 12 to 17 years, inclusive will also be enrolled. The study will attempt to enroll a representative study population that is demographically diverse, and for the adult study (Stage 1), that is proportional to those affected by the disease during the current mpox outbreak in the United States. In Stage 2, the study will aim to enroll a population that is representative of the U.S. population to ensure broad applicability of the study findings given that the findings will be used to inform a label change in the U.S. for use of JYNNEOS in adolescents. While adolescents are not the main population impacted by the current global outbreak, there is a risk that sexually active adolescents could be impacted if mpox were introduced into this population.

#### Sites

Up to 21 U.S. clinical research sites will be involved in the study. Not all sites will participate in all stages or in all arms.

#### **Study intervention**

JYNNEOS is live vaccine produced from the strain MVA-BN, an attenuated orthopoxvirus, that does not replicate in human cells. A 2-dose SC regimen of 1 x  $10^8$  TCID<sub>50</sub> MVA-BN given 4 weeks apart is FDA-approved and licensed as a smallpox and mpox vaccine for adults, and FDA-authorized under an emergency use authorization (EUA) for children and adolescents in the United States. In addition, the FDA authorized an EUA for use of a 2-dose ID regimen of 2 x  $10^7$  TCID<sub>50</sub> MVA-BN given 4 weeks apart in adults on August 9, 2022. In Stage 1 of this study, a 2-dose ID regimen of 1 x  $10^7$  TCID<sub>50</sub> MVA-BN, given 4 weeks apart, was evaluated as an investigational dose sparing regimen.

#### Stage 1 (Adult)

There will be three study arms in which JYNNEOS will be administered by either ID or SC injection at Day 1 and 29.

#### Stage 2 (Adult and Adolescent)

There will be two study arms in which JYNNEOS will be administered by SC injection at Day 1 and 29.

#### **Study Duration**

DMID/NIAID/NIH 

This study will take approximately 24-36 months to conduct from study activation to the last study visit of the final participant enrolled.

# **Participant Duration**

It will take approximately one year for a participant to complete their participation in the study in Stage 1 and approximately 13 months in Stage 2.

#### Safety

The trial will use study and individual pausing rules. See corresponding section for details. This trial will use a Data Safety Monitoring Board (DSMB) for objective study oversight and review of any study pause.

# 1.2 Schedule of Activities (SOA)

For the Schedule of Activities (SOA) for each study stage refer to the corresponding appendix. Refer to Manual of Procedures (MOP) for detailed description of study activities.

# 2. Introduction

# 2.1 Study Rationale

On July 23, 2022, WHO declared the 2022 mpox outbreak a public health emergency of international concern (PHEIC). Since the first case of mpox was detected in the UK in a returning traveler from Nigeria on May 6, 2022, as of December 2022 the outbreak has rapidly spread to 110 countries or locations worldwide, including 103 that are non-endemic, marking the first time mpox has spread widely outside Central and West Africa. In August, the number of confirmed mpox cases in the U.S. surpassed that of any other country<sup>2,3</sup>. To mitigate the consequences of this outbreak, JYNNEOS vaccine is being offered to individuals considered to be at high risk. However, there is a global vaccine shortage and increasing the supply will take time. This study will evaluate vaccine dose sparing strategies to extend the limited supply during this global public health crisis in Stage 1, and in Stage 2, the study will evaluate vaccine safety and immunogenicity among adolescents ages 12 to 17 years to extend eligibility to adolescent population.

# 2.2 Background

Mpox is a reemerging infectious disease caused by Monkeypox virus (MPXV), a large double-stranded DNA virus belonging to the genus *Orthopoxvirus*. MPXV is a zoonotic orthopoxvirus, primarily transmitted to humans via contact with infected animals, and causing disease similar to smallpox, although with substantially lower mortality. MPXV is endemic to West and Central Africa, where the incidence of human mpox cases has increased as much as 20-fold since the end of the smallpox vaccination campaign in 1980. Outbreaks in non-endemic countries have been related to the exotic pet trade and international travel. Prior to the current global mpox outbreak, secondary human-to-human transmission in non-endemic countries was rare, and documented only twice since 2018, both cases involving travelers returning from Nigeria. The first case involved transmission between the index patient and a healthcare provider and second case

DMID/NIAID/NIH 

involved transmission to another adult and an infant within the household of the index case. <sup>14,15</sup> Mpox reemerged in Nigeria in 2017 after more than 40 years with no reported cases. <sup>16,17</sup>

On May 18, 2022, the first U.S. case of mpox was detected as part of the larger global 2022 mpox outbreak.<sup>18</sup> The U.S. was the fourth non-endemic country to detect a case in a returning traveler. On August 4, the U.S. Department of Health and Human Services declared the U.S. mpox outbreak to be a public health emergency with 7,510 confirmed cases of mpox detected in all U.S. states, D.C, and Puerto Rico.<sup>19</sup> As of December 22, 2022, there have been 83,424 confirmed mpox cases in 110 locations and countries; most cases have been from 103 non-endemic areas including 29,740 confirmed cases and 20 deaths in the United States.<sup>2</sup>

Vaccination is being used as a mitigation strategy in the current mpox outbreak for those exposed to and those deemed to be at higher risk of being exposed to mpox. There is one FDA-approved vaccine for mpox: JYNNEOS Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN). A second vaccine, ACAM2000, is likely effective but is not FDA-approved for mpox and associated with moderate risk of myocarditis and pericarditis (5.7 cases per 1,000 vaccinated) as well as encephalomyelitis, progressive vaccinia, generalized vaccinia, and ocular complications. ACAM2000 should not be given to people with a weakened immune system, eczema, cardiac disease, infants < 12 months, or pregnant women. Given these attributes, JYNNEOS is the preferred vaccine during the current outbreak and there is a limited supply of the vaccine globally with production unlikely to keep up with the growing demand as the outbreak continues to spread. Given the limited supply of MVA-BN, on August 9, 2022, the FDA issued an Emergency Use Authorization (EUA) for the emergency use of a lower (2 x 10<sup>7</sup>) ID dose of JYNNEOS for individuals 18 years of age and older determined to be at high risk for mpox infection. In addition, the EUA allowed for the emergency use of the licensed SC dose for individuals less than 18 years of age determined to be at high risk for mpox infection as JYNNEOS is licensed for use in only adults.

In the first stage of this platform trial, several potential dose sparing strategies were considered. Use of a reduced dose administered SC is unlikely to be of comparable immunogenicity to the licensed SC regimen. There were several Phase 1 and 2 trials that evaluated 2-dose regimens of MVA-BN administered SC four weeks apart (Table 2). Although the 2-dose  $5x10^7$  TCID<sub>50</sub> SC regimen may elicit GMT similar to that of ACAM2000, the GMT will likely be below that of the licensed 2-dose 1 x  $10^8$  TCID<sub>50</sub> MVA-BN regimen.

**Table 2 Prior Subcutaneous Dosing Trials** 

| Reference | | 1 X10 <sup>7</sup> | 2 X10 <sup>7</sup> | 5 X10 <sup>7</sup> | 1 X10 <sup>8</sup> | Assay |
|---|---|---|---|---|---|---|
| | | TCID <sub>50</sub> | TCID <sub>50</sub> | TCID <sub>50</sub> | TCID <sub>50</sub> | |
| Vollmar et al, | Liquid | 6.4 | | | 29.3 | IHD-J |
| Vaccine, 2006 20 | formulation | (CI not reported) | | | (CI not reported) | PRNT GMT |
| Frey at al. | Lyophilized | | 347.2 | 551.5 | 914.5 | MVA |
| Vaccine, 2007 | formulation | | (161.9, 744.7) | (321.5, 946.0) | (528.0, 1584) | PRNT GMT |
| von Krempelhuber | Lyophilized | | 5.5 | 10.3 | 19.4 | IHD-J |
| Vaccine, 2010 | formulation | | (3.2, 9.6) | (5.8, 18.4) | (11.1, 34.2) | PRNT GMT |

A single 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN dose has also been suggested for dose sparing, but in our assessment of the published literature, it is unlikely to be immunogenically equivalent to the

DMID/NIAID/NIH 

standard licensed 2-dose regimen. The pivotal Phase 3 trial demonstrated that a single dose is likely to provide a significantly lower GMT than the licensed 2-dose MVA-BN regimen, 16.9 [13.7, 20.8] as compared to 153.5 [134.3, 175.6], respectively (Table 3).

| | | MVA-BN<br>(N=185) | | | ACAM2000<br>(N=186) | | | GMTs ratio<br>MVA/ ACAM |
|---|---|---|---|---|---|---|---|---|
| Visit Week | n | GMT | 95% CI | n | GMT | 95% CI | Ratio | 95% CI |
| Plaque Reduction Neutralization Test | | | | | | | | |
| Week 0 | 185 | 1.0 | [1.0, 1.1] | 186 | 1.0 | [1.0, 1.0] | 1.008 | [0.97, 1.05] |
| Week 2 | 184 | 16.2 | [13.0, 20.1] | 184 | 16.2 | [13.1, 20.0] | 0.997 | [0.74, 1.35] |
| Week 4 | 185 | 16.9 | [13.7, 20.8] | 186 | 79.3 | [67.1, 93.8] | 0.213 | [0.16, 0.28] |
| Week 6 | 185 | 153.5 | [134 3 175 6] | 181 | 64 7 | [54 9 76 2] | 2 372 | [1 92 2 93] |

Table 3 MVA-BN Compared to ACAM2000

NIAID conducted a Phase 2 trial comparing the standard (now licensed) 2-dose 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN SC regimen (liquid formulation) and a 2-dose 2 x 10<sup>7</sup> TCID<sub>50</sub> MVA-BN ID regimen (liquid formulation) and found peak vaccinia virus, Western reserve strain (VV-WR) GMT of 49.5 (40.0, 61.3) and 59.6 (48.1, 74.0), respectively (Table 4).<sup>21</sup> The 2-dose 2 x 10<sup>7</sup> TCID<sub>50</sub> ID regimen was non-inferior to the 2-dose 1 x 10<sup>8</sup> TCID<sub>50</sub> SC regimen and utilized only one-fifth of the dose. These results are supported by a trial evaluating another MVA vaccine (ACAM3000) which showed ID vaccination at 1x10<sup>7</sup> TCID<sub>50</sub> had similar VV-WR GMT to 1x10<sup>8</sup> TCID<sub>50</sub> administered SC or IM.<sup>22</sup>

| Study Visit Day | Group | | |
|---|---|---|---|
| | Lyophilized SC 1x10 <sup>8</sup> (N=145) GMT [95% CI] | Liquid SC 1x10 <sup>8</sup><br>(N=149) GMT [95% CI] | Liquid ID 2x10 <sup>7</sup><br>(N=146) GMT [95% CI] |
| Day 0 | 7.5 [,] | 7.7 [7.4, 8.0] | 7.7 [7.4, 7.9] |
| Day 14 | 10.9 [9.9, 12.0] | 10.0 [9.0, 11.1] | 10.3 [9.3, 11.3] |
| Day 28 | 10.8 [9.9, 11.9] | 9.6 [8.7, 10.6] | 10.8 [9.9, 11.9] |
| Day 42 | 77.6 [62.3, 96.7] | 45.2 [36.4, 56.2] | 54.4 [43.7, 67.8] |
| Peak post vaccination 2 | 87.8 [71.2, 108.3] | 49.5 [40.0, 61.3] | 59.6 [48.1, 74.0] |

Table 4. Prior Intradermal Dosing Compared to Subcutaneous

Even with the EUA for intradermal MVA-BN being available, Stage 1 of this trial is designed to evaluate several unique issues:

- As vaccine supply is not anticipated to meet the demand in the next year, this trial will evaluate dose reduction strategies focused on the ID route, that is, confirming the previously studied ID dose and evaluating one tenth dose of MVA-BN (1x10<sup>7</sup>).
- This trial will also assess differences in safety and tolerability of the ID versus the licensed SC regimen as issues of tolerability have been raised by the manufacturer and some in the medical community.

While JYNNEOS is available under EUA for individuals younger than 18 years of age, this EUA will expire in January 31, 2023. An FDA approved mpox vaccine for adolescents is lacking and remains a public health need. Most reported cases in the global 2022 mpox outbreak have involved

DMID/NIAID/NIH 

men who have sex with men, with a median age of 34 years. Among global cases with age data available, 1.2% are aged 0-17 years;<sup>23</sup> in the United States, from May 17 through September 24, 2022, MPXV infections in persons under 18 years of age accounted for 0.3% of reported cases.<sup>24</sup> Among 55 adolescents aged 13-17 years, 89% were male, and the most common route of exposure was male to male sexual contact (66%). Prior to the global 2022 outbreak, mpox occurred primarily in children and adolescents in endemic countries.<sup>25,26</sup> Increased mpox transmission within adolescent populations could occur if the outbreak continues, or in future outbreaks, given the mode of transmission through skin and mucosal contact during sexual activity or other activities with close contact.

# 2.3 Risk/Benefit Assessment

For information regarding risk/benefit assessment for each study stage, see the corresponding appendix.

# 3. OBJECTIVES AND ENDPOINTS

For objectives and endpoints for each study stage, see the corresponding appendix.

# 4. STUDY DESIGN

# 4.1 Overall Design

This study is a Phase 2 randomized, open-label, non-placebo controlled, multi-site clinical trial that will evaluate two ID regimens for MVA-BN vaccine compared to the standard SC regimen in healthy, vaccinia-naïve adults 18 to 50 years of age, inclusive, (Stage 1). In Stage 2 of the study, the standard SC regimen will be evaluated in adolescents ages 12 through 17 years, inclusive, and compared to the standard SC regimen in adults ages 18 to 50, inclusive.

In Stage 1, approximately 230 adult participants will be enrolled and randomized to one of three study arms. The two dose sparing strategies include one-fifth (2 x10<sup>7</sup>) and one-tenth (1 x10<sup>7</sup>) of the standard dose of MVA-BN administered ID on Day 1 and 29 (Arm 1 and 2, respectively). The comparator arm (Arm 3) will be the 2-dose standard (1x10<sup>8</sup>) MVA-BN SC regimen. Stage 1 will enroll a 1:1:1 randomization allocation.

In Stage 2, approximately 135 healthy, vaccinia-naïve adults will be enrolled (Arm 4) and will be given the standard, licensed regimen of 1x10<sup>8</sup> MVA-BN administered SC on Day 1 and 29 and will be combined with adults from Arm 3 (Stage 1) to be the comparator for the primary endpoint, non-inferiority testing. Approximately 315 healthy, vaccinia-naïve adolescents will be enrolled and given 1x10<sup>8</sup> MVA-BN administered SC on Days 1 and 29 (Arm 5). The study will have a set target enrollment of at least 25% adolescents ages 12 to 14 years to ensure that adequate numbers of younger adolescents are enrolled.

DMID/NIAID/NIH 

# 4.2 Scientific Rationale for Study Design

The rationale for each of the arms in this study is as follows:

1. MVA-BN 2 x 10<sup>7</sup> ID (1/5th dose) on Days 1, 29 (Study Arm 1) – This regimen matches the prior ID dosing and matches the dose authorized in the EUA. This regimen would allow for 5-fold increase in vaccine supply.

- 2. MVA-BN 1 x 10<sup>7</sup> ID (1/10th dose) on Days 1, 29 (Study Arm 2) This regimen would test a larger dose conservation. This regimen would allow for 10-fold increase in vaccine supply.
- 3. MVA-BN 1 x 10<sup>8</sup> SC on Days 1, 29 (Study Arms 3, 4, and 5) This regimen is the licensed dose and route. Arm 3 will be used as a comparator to ID doses of MVA BN (Arms 1 and 2, Stage 1). Arms 4 (adult) and 5 (adolescent) will be used to evaluate noninferiority of this licensed regimen among adolescents compared to adults (Stage 2).

#### 4.3 **Justification for Dose**

This study will use the FDA-approved, licensed dose 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN administered SC on Day 1 and 29 in Stage 2 of the study and as the comparator for the ID doses of MVA-BN in Stage 1. It is anticipated that the licensed, 2-dose SC regimen will be safe and immunogenic in adolescents. The ID regimens being evaluated in this study use lower doses of the licensed vaccine, and either match or are one dilution lower than the dose used in the prior ID dosing study (PMID 26143613). Therefore, it is anticipated that these doses administered ID will be safe and immunogenic.

# 5. STUDY POPULATION

For a description of the study population, eligibility criteria, lifestyle considerations, procedures for screen failures, recruitment and retention strategies for each stage see the corresponding appendix.

# 6. STUDY PRODUCT

# 6.1 Study Product(s) and Administration

# **6.1.1** Study Product Description

JYNNEOS is FDA-approved and licensed as a smallpox and mpox vaccine in the United States. The vaccine, when thawed, is a milky, light yellow to pale white colored suspension that is licensed for subcutaneous injection. JYNNEOS is a live vaccine produced from the strain Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN), an attenuated, non-replicating orthopoxvirus. MVA-BN is grown in primary Chicken Embryo Fibroblast (CEF) cells suspended in a serum-free medium containing no material of direct animal origin, harvested from the CEF cells, purified, and concentrated by several Tangential Flow Filtration (TFF) steps including benzonase digestion. Each 0.5 mL dose is formulated to contain 0.5 x 10<sup>8</sup> to 3.95 x 108 infectious units of MVA-BN live virus in 10 mM Tris (tromethamine), 140 mM sodium chloride at pH 7.7. Each 0.5 mL dose

DMID/NIAID/NIH 

may contain residual amounts of host-cell DNA ( $\leq$  20 mcg), protein ( $\leq$  500 mcg), benzonase ( $\leq$ 0.0025 mcg), gentamicin ( $\leq$ 0.163 mcg), and ciprofloxacin ( $\leq$ 0.005 mcg).

# 6.1.2 Dosing and Administration

In this trial, a licensed vaccine is being evaluated (i.e., JYNNEOS) and there is no placebo group (Table 5). In Stage 1, use of the contralateral arm was an option if there is any residual local reaction at Day 29 or if participant requests that this be done. In Stage 2, the second vaccination will be given in the contralateral arm unless the site deems that using the same arm is in the best interest of the participant in terms of safety or using the same arm (for the second injection) will enable the site to better evaluate reactogenicity (e.g., tattoo on opposite upper arm). If the second vaccination is given in the same arm as the first vaccination, the second injection should be given approximately 5 cm away from the first injection site if physically possible.

#### **Table 5 Study Arms**

Stage 1 (Adult)

| ouge I (Hum) | | | | |
|---|---|---|---|---|
| Arm | Dose of JYNNEOS (MVA-BN) | Route of Administration* | Vaccination Day | |
| | | | Day 1 | Day 29 |
| 1 | 2 x 10 <sup>7</sup> TCID <sub>50</sub> , (0.1 mL) | Intradermal | X | X |
| 2 | 1 x 10 <sup>7</sup> TCID <sub>50</sub> , (0.05 mL) | Intradermal | X | X |
| 3 | $1 \times 10^8 \text{ TCID}_{50}, (0.5 \text{ mL})$ | Subcutaneous | X | X |

**Stage 2 (Adults and Adolescent)** 

| Arm | Dose of JYNNEOS<br>(MVA-BN) | Route of Administration* | Vaccination Day | |
|---|---|---|---|---|
| | | | Day 1 | Day 29 |
| 4 (Adult) | 1 x 10 <sup>8</sup> TCID <sub>50</sub> , (0.5 mL) | Subcutaneous | X | X |
| 5 (Adolescent) | 1 x 10 <sup>8</sup> TCID <sub>50</sub> , (0.5 mL) | Subcutaneous | X | X |

<sup>\*</sup>Subcutaneous is administered in the upper arm, intradermal is administered in the volar aspect (inner side) of the forearm.

#### **6.1.3 Dose Escalation**

Not Applicable.

#### **6.1.4 Dose Modifications**

Not Applicable.

#### 6.1.5 Criteria for Redosing

If study product administration is unsuccessful, another administration will not be attempted.

# 6.2 Preparation/Handling/Storage/Accountability

# 6.2.1 Acquisition and Accountability

DMID/NIAID/NIH 

# **Product: JYNNEOS (MVA-BN vaccine)**

The JYNNEOS (MVA-BN vaccine) will be stored and provided by DMID Repository. Study product will be shipped to the clinical research site upon request and approval from DMID.

#### **Accountability**

The participating site PI is responsible for study product distribution and disposition and has ultimate responsibility for study product accountability. The participating site PI may delegate to the participating site's research pharmacist responsibility for study product accountability. The participating site's research pharmacist will be responsible for maintaining complete records and documentation of study product receipt, accountability, dispensation, storage conditions, and final disposition of the study products.

Time of vaccine administration to the participant will be recorded on the appropriate data collection form (DCF). All study product(s), including the amount of JYNNEOS (MVA-BN vaccine), and whether administered or not, must be documented on the appropriate study product accountability record or dispensing log. The sponsor's monitoring staff will verify the participating site's study product accountability records and dispensing logs per the DMID-approved clinical monitoring plan (CMP).

Once all participant dosing is complete, the pharmacy staff should retain or dispose of used study products and complete study product accountability procedures in accordance with site-specific standard operating procedures (SOPs). This applies to:

- used JYNNEOS (MVA-BN vaccine) vials
- JYNNEOS (MVA-BN vaccine) cartons

All used vials and cartons may either be sequestered from the unused supplies and retained until study conclusion or until study product accountability has occurred by the monitor and written notification stating retention is no longer required is received. Used syringes should be discarded per usual procedure.

#### **Disposition**

After the study treatment period has ended or as appropriate over the course of the study after study product accountability has been performed, guidance for disposition of unused JYNNEOS (MVA-BN vaccine) vials will be provided by DMID.

#### 6.2.2 Formulation, Appearance, Packaging, and Labeling

#### **Product: JYNNEOS (MVA-BN vaccine)**

JYNNEOS is supplied in a single-dose vial with turquoise and white label for SC injection. Each 0.5 mL dose is formulated to contain 0.5 x  $10^8$  to 3.95 x  $10^8$  infectious units of MVA-BN live virus in 10 mM Tris (tromethamine), 140 mM sodium chloride at pH 7.7. Each 0.5 mL dose may contain residual amounts of host-cell DNA ( $\leq$  20 mcg), protein ( $\leq$  500 mcg), benzonase ( $\leq$ 0.0025 mcg), gentamicin ( $\leq$ 0.163 mcg), and ciprofloxacin ( $\leq$ 0.005 mcg). JYNNEOS is a sterile vaccine formulated without preservatives. The vial stoppers are not made with natural rubber latex.

# 6.2.3 Product Storage and Stability

DMID/NIAID/NIH 

#### **Product: JYNNEOS (MVA-BN vaccine)**

JYNNEOS should be kept frozen at -25°C to -15°C (-13°F to +5°F) and stored in the original package to protect from light. JYNNEOS should not be re-frozen once a vial has been thawed. Once thawed, the vaccine may be kept at +2°C to +8°C (+36°F to +46°F) for 4 weeks. The package insert provides additional instructions for the handling and storage of JYNNEOS.

#### 6.2.4 Preparation

Each dose (0.5 mL) is supplied in a single-dose vial. Sites should allow the vaccine to thaw and reach room temperature before use (about 15 to 30 minutes). After thawing, the total time stored at +2°C to +8°C (+36°F to +46°F) should not exceed 4 weeks. Once the vial is punctured and a dose is withdrawn, if it is not used in its entirety, it should be stored at +2°C to +8°C (+36°F to +46°F) and discarded within 8 hours of the first puncture. If the unpunctured vial is initially shipped/stored at 2-8C then it is stable for up to 8 weeks. Sites should not refreeze the vaccine. JYNNEOS may be kept frozen until the expiration date.

JYNNEOS is a light yellow to pale white colored, milky suspension when thawed. Sites will visually inspect the product for particulate matter and discoloration prior to administration. If either condition is present, the vaccine will not be administered. Study product administrators will gently swirl the vial for at least 30 seconds.

For the ID injection (Arm 1), 0.1 mL of vaccine will be withdrawn from the vial into a sterile syringe and injected intradermally into the volar aspect (inner side) of the forearm.

For the ID injection (Arm 2), 0.05 mL of vaccine will be withdrawn from the vial into a sterile syringe and injected intradermally into the volar aspect of the forearm.

For the SC injection (Arms 3, 4 and 5), 0.5 mL of vaccine will be withdrawn from the vial into a sterile syringe and injected into the fatty subcutaneous tissue of the upper arm.

See the protocol-specific MOP for detailed information on the preparation, labeling, storage, and administration for each arm.

# 6.3 Measures to Minimize Bias: Randomization and Blinding

#### **6.3.1** Treatment Assignment Procedures

The randomization procedure will be described in the MOP.

#### 6.3.2 Randomization

For Stage 1, there will be a 1:1:1 randomization allocation. Randomization will not be stratified. Randomized treatment assignments will be generated by a statistician at The Emmes Company, LLC, the Data and Statistical Coordinating Center (SDCC) for this study. Participants will be registered using a web-based application developed by The Emmes Company, LLC. Upon entry

DMID/NIAID/NIH 

of demographic data and confirmation of eligibility for the trial, the participant will be enrolled and randomized. The randomization procedure will be described in more detail in the MOP.

Stage 2 is not randomized. All Stage 2 participants will receive the licensed SC regimen. For Stage 2, the aim is to enroll at least 25% adolescents ages 12 to 14 years.

## **6.3.3** Blinding and Masking Procedures

This study will not utilize blinding or masking procedures as it is an open-label, non-placebocontrolled trial. Research laboratories will be blinded to participant study arm for the purposes of immunogenicity/efficacy evaluations.

# 6.4 Study Intervention Compliance

Each dose of JYNNEOS will be administered by a member of the clinical research team that is qualified per state and institution policies to administer the study product. Administration and date, time, and location of injection will be recorded on the appropriate eCRF.

# 6.5 Concomitant Therapy

For this platform trial that evaluates use of JYNNEOS vaccine, participants in all stages will be asked to avoid use of medications that might interfere with the evaluation of the immune response to the vaccine unless clinically indicated for a medical condition diagnosed after enrollment. Specific information regarding concomitant therapy for each study stage, see the corresponding appendix.

# 7. STUDY INTERVENTION DISCONTINUATION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

For this platform trial, additional individual and study halting criteria were added for stages involving more vulnerable populations for which safety profile is largely unknown (e.g., adolescents). For each stage, see the corresponding appendix for specific information. Refer to the corresponding appendix for information regarding participants who discontinue study intervention, study withdrawal, and participants lost to follow-up.

# 8. STUDY ASSESSMENTS AND PROCEDURES

Please see Appendix A and B for Sections 8.1 through 8.5.

For information regarding study assessments and procedures for each study stage, see the corresponding appendix.

#### **8.6** Adverse Events and Serious Adverse Events

#### **8.6.1** Definition of Adverse Events (AE)

DMID/NIAID/NIH 

Adverse event means any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related (21 CFR 312.32 (a)). An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product.

Any medical condition that is present at the time the participant is screened will be considered as baseline and not reported as an AE. However, if the severity (i.e., grade) of any pre-existing medical condition increases, it should be recorded as an AE.

Adverse events can be further divided into solicited adverse events and unsolicited adverse events. Solicited adverse events are those for which the study team will specifically query the participant whether they occurred. Unsolicited adverse events are those events that the participant report occurring without being queried about the specific event.

#### **8.6.1.1** Solicited Adverse Events

Reactogenicity will be especially important to document because of prior studies demonstrating more local (measurement) reactogenicity among participants who received the ID MVA-BN vaccine injection. This study will collect the following solicited adverse events based on prior studies. This includes local (pain at the site of the injection, erythema/redness, induration/swelling, pruritis) and systemic (fever, chills, nausea, headache, fatigue, change in appetite, myalgia [exclusive of the injection site], and arthralgia) reactogenicity. In addition, there is an expectation that some participants will develop skin discoloration and nodules which will be reported as AEs and not collected on the memory aid and followed through to resolution. For this study, the following toxicity grading scale is used:

"FDA Guidance for Industry, Toxicity Grading Scale for Healthy Adults and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" as a reference.

Of note, pruritis/itching, arthralgia, chills, and change in appetite are not included in the FDA toxicity table. However, the FDA Guidance allows for addition of other signs and symptoms as follows:

Mild: No interference with activity
Moderate: Some interference with activity

Severe: Prevents daily activity
Potentially Life Threatening: ER visit or hospitalization

#### **8.6.1.2** Unsolicited Events

Unsolicited events are all AEs spontaneously reported by the participant and/or in response to an open question from study personnel or revealed by observation, physical examination, or other diagnostic procedures.

#### **8.6.2** Definition of Serious Adverse Events

An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes (21 CFR 312.32 (a)):

DMID/NIAID/NIH 

- death
- a life-threatening adverse event\*
- inpatient hospitalization or prolongation of existing hospitalization
- a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or
- a congenital anomaly/birth defect.

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, convulsions that do not result in inpatient hospitalization, etc.

\* An adverse event is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient or participant at immediate risk of death. It does not include grade 4 severity unless the adverse event might have caused death.

# 8.6.3 Classification of an Adverse Event

The determination of seriousness, severity and causality will be made by an on-site investigator or other staff as listed on the delegation log. Any potential grade 3 or 4 AE should be evaluated by someone qualified to provide a medical evaluation of AEs. This includes but is not limited to physicians, physician assistants, and nurse practitioners.

#### 8.6.3.1 Severity of Event

All AEs or SAEs will be assessed for severity, according to the toxicity grading scale, FDA Guidance for Industry, Toxicity Grading Scale for Healthy Adults and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. For adverse events (AEs) not included in the protocol-defined grading scale, the following guidelines will be used to describe severity.

<u>Mild (Grade 1)</u>: Events that are usually transient and may require only minimal or no treatment or therapeutic intervention and generally do not interfere with the participant's usual activities of daily living.

<u>Moderate (Grade 2)</u>: Events that are usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant.

<u>Severe (Grade 3)</u>: Events interrupt usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Severe events are usually incapacitating.

<u>Life-threatening (Grade 4)</u>: Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or care provided.

# **8.6.3.2** Relationship to Study Intervention

For each reported adverse event or reaction, the Principal Investigator or designee must assess the relationship of the event to the study product using the following guideline:

DMID/NIAID/NIH 

<u>Related</u> – The AE is known to occur with the study intervention, there is a reasonable possibility that the study intervention caused the AE, or there is a temporal relationship between the study intervention and event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study intervention and the AE.

<u>Not Related</u> – There is not a reasonable possibility that the administration of the study intervention caused the event, there is no temporal relationship between the study intervention and event onset, or an alternate etiology has been established.

# 8.6.5 Adverse Event Reporting

#### 8.6.5.1 Investigators Reporting of AEs

All clearly related signs, symptoms, and results of diagnostic procedures performed because of an AE should be grouped together and recorded as a single diagnosis or AE term, if available. If the AE is a laboratory abnormality that is part of a clinical condition or syndrome, it should be recorded as the syndrome or diagnosis rather than the individual laboratory abnormality. Each AE will also be described in terms of duration (start and stop date), severity, association with the study product, action(s) taken, and outcome.

AEs characterized as intermittent require documentation of onset and duration of each episode. All AEs will be assessed for severity, relatedness to study vaccine (see Section 8.6.3.1 and Section 8.6.3.2) and seriousness (see Section 8.3.2) by the study PI or sub-investigator.

All AEs will be captured on the appropriate data collection form. Information to be collected for AEs includes event term or description, date of onset, assessment of severity, relationship to study product, and alternate etiology (assessed only by those with the training and authority to make a diagnosis and listed on the Form FDA 1572 as an investigator), date of resolution, seriousness, and outcome. AEs occurring during the trial collection and reporting period will be documented appropriately regardless of relationship.

# 8.6.5.2 Special Reporting of Adverse Events

Protocol specified Adverse Events of Special Interest (AESIs) will be reported within 24 hours of the site awareness of the AESI to the DMID Pharmacovigilance Group via the mechanism described below for SAE reporting (see Section 8.6.6.1).

#### 8.6.6 Serious Adverse Event Reporting

#### 8.6.6.1 Investigators Reporting of SAEs

Any AE that meets a protocol-defined serious criterion must be submitted immediately (within 24 hours of site awareness) on an SAE form to the DMID Pharmacovigilance Group, at the following address:

DMID Pharmacovigilance Group Clinical Research Operations and Management Support (CROMS) 6500 Rock Spring Dr. Suite 650 Bethesda, MD 20817, USA

DMID/NIAID/NIH 

SAE Hot Line: 1-800-537-9979 (US) or 1-301-897-1709 (outside US) SAE FAX Number: 1-800-275-7619 (US) or 1-301-897-1710 (outside US)

SAE Email Address: PVG@dmidcroms.com

In addition to the SAE form, select SAE data fields must also be entered into the SDCC system. See the protocol-specific MOP for details regarding this procedure.

Other supporting documentation of the event may be requested by the DMID Pharmacovigilance Group and should be provided as soon as possible. The DMID Medical Monitor will review and assess the SAE for regulatory reporting and potential impact on study participant safety and protocol conduct.

At any time after completion of the study, if the site principal investigator or appropriate sub-investigator becomes aware of an SAE that is suspected to be related to study product, the site principal investigator or appropriate sub-investigator will report the event to the DMID Pharmacovigilance Group.

# **8.6.6.2** Regulatory Reporting of SAEs

Following notification from the site Principal Investigator or appropriate sub-investigator, DMID, as the IND sponsor, will report any Suspected Unexpected Serious Adverse Reaction (SUSAR) to the FDA as an IND safety report. DMID will report an AE as a suspected unexpected adverse event only if there is evidence to suggest a causal relationship between the study intervention and the AE.

The Sponsor must ensure the event meets all three of the definitions:

- Suspected adverse reaction.
- Serious.
- Unexpected.

Both serious and unexpectedness are important, but the event will be reported only if there is evidence to suggest a causal relationship between the drug and the adverse event, such as:

- A single occurrence of an event that is uncommon and known to be strongly associated with drug exposure.
- One or more occurrences of an event that is not commonly associated with drug exposure but is otherwise uncommon in the population exposed to the drug.
- On review as an aggregate analysis when the occurrence is higher than the historical control.

DMID will report to the FDA any unexpected fatal or life-threatening suspected adverse reaction as soon as possible, but in no case later than 7 calendar days after the sponsor's initial receipt of the information. If the event is not fatal or life-threatening the IND safety report will be submitted within 15 calendar days after the sponsor determines that the information qualifies for reporting as specified in 21 CFR Part 312.32. Relevant follow up information to an IND safety report will be submitted as soon as the information is available. Upon request from FDA, DMID will submit to the FDA any additional data or information that the agency deems necessary, as soon as possible, but in no case later than 15 calendar days after receiving the request.

DMID/NIAID/NIH 

DMID will submit an IND safety report to the FDA and will notify all participating site Principal Investigators (i.e., all Principal Investigators to whom the sponsor is providing drug under its IND(s) or under any Principal Investigator's IND(s) of potential serious risks from clinical studies or any other source, as soon as possible. SAEs that are not SUSARs will be reported to the FDA at least annually in a summary format which includes all SAEs.

#### **8.6.7** Reporting Events to Participants

Participants have the right to be informed of any new findings of AEs or SAEs that may affect their safety or influence their choice to participate or continue participating in the study.

#### **8.6.8** Reporting of Pregnancy

Pregnancy is not an AE. However, any pregnancy that occurs during study participation (through Day 365 Stage 1, and Day 394 for Stage 2) should be reported to the sponsor on the appropriate DCF. Pregnancy should be followed for safety and outcome. This follow-up will include pregnancy outcome (termination, pre-term birth, term birth) and newborn outcome (live birth, fetal demise, stillbirth; presence of any congenital anomalies). No in-person visits will be required for pregnancy outcome determination.

# 8.7 Unanticipated Problems

# **8.7.1 Definition of Unanticipated Problems (UP)**

The Department of Health and Human Services Office for Human Research Protections (OHRP) considers unanticipated problems (UPs) involving risks to participants or others to include, in general, any incident, experience, or outcome that meets <u>all of</u> the following criteria:

- Unexpected in terms of nature, severity, or frequency given (a) the research procedures that are described in the protocol-related documents, such as the Institutional Review Board (IRB)-approved research protocol and informed consent, parental permission and assent documents; and (b) the characteristics of the participant population being studied; and
- Related or possibly related to participation in the research ("possibly related" means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research); and
- Suggests that the research places participants or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

Incidents arising from noncompliance with study procedures should be reported as protocol deviations (see Section 8.1.1). An incident that qualifies as both a UP and a protocol deviation should be reported as both.

### 8.7.2 Unanticipated Problem Reporting

The investigator will report UPs to the study sponsor, the reviewing Institutional Review Board (IRB) and to the SDCC.

DMID/NIAID/NIH 

The UP report will include the following information:

• Protocol identifying information: protocol title and number, PI's name, and the IRB project number;

- A detailed description of the event, incident, experience, or outcome;
- An explanation of the basis for determining that the event, incident, experience, or outcome represents an UP;
- A description of any changes to the protocol or other corrective actions that have been taken or are proposed in response to the UP.

To satisfy the requirement for prompt reporting, UPs will be reported using the following timeline:

- UPs that are SAEs will be reported to the IRB and to the SDCC/study sponsor within 24 hours of the investigator becoming aware of the event.
- Any other UP will be reported to the IRB and to the SDCC/study sponsor within a timeline defined according to the relevant policies.
- UPs will be collected through the end of the study.

#### **8.7.3** Reporting Unanticipated Problems to Participants

Participants will be informed of any UPs that will potentially influence their participation in this trial.

# 9. STATISTICAL CONSIDERATIONS

For statistical considerations for each study stage, see the corresponding appendix.

# 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

# 10.1 Regulatory, Ethical, and Study Oversight Considerations

This study will be conducted in conformity with the principles set forth in The Belmont Report: Ethical Principles and Guidelines for the Protection of Human Participants of Research (US National Commission for the Protection of Human Participants of Biomedical and Behavioral Research; April 18, 1979), and the federal policy for the Protection of Human Participants codified in 45 CFR Part 46, 21 CFR Part 50 (Protection of Human Participants), and the ICH E6(R2).

An OHRP-registered IRB will review and approve this protocol, associated informed consent, parental permission and assent documents, recruitment materials, and handouts or surveys intended for the participants, prior to the recruitment, screening and enrollment of participants. The IRB review shall be in accordance with 45 CFR 46 and 21 CFR 50, 21 CFR 56 (IRBs), and other federal, state, and local regulations and policies, as applicable.

DMID/NIAID/NIH 

Each institution engaged in this research will hold a current Federalwide Assurance (FWA) issued by the Office for Human Research Protections (OHRP) for federally funded research. and provide the FWA number to DMID. Each site principal investigator will obtain IRB approval for this protocol and any amendments to be conducted at his/her research site(s).

Any amendments to the protocol or informed consent, parental permission and assent documents will be approved by the IRB before they are implemented. IRB review and approval will occur at least annually throughout enrollment and follow-up of participants, in accordance with applicable regulations and the requirements of the IRB/IEC. The participating site PI will notify the IRB of deviations from the protocol and reportable SAEs, as applicable to the IRB policy.

DMID must receive the documentation that verifies IRB/IEC approval for this protocol, informed consent, parental permission and assent documents and associated documents, prior to the recruitment, screening and enrollment of participants, and any IRB approvals for continuing review or amendments as required by DMID.

#### **10.1.1 Informed Consent Process**

For information regarding the informed consent and assent, where applicable, process for each study stage, see the corresponding appendix.

## **10.1.2** Study Termination and Closure

Section 7, Study Intervention Discontinuation and Participant Discontinuation/Withdrawal, describes the temporary halting of the study. This study may be prematurely terminated if there is sufficient reasonable cause, including but not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants
- Results of interim efficacy or futility analysis
- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable
- Regulatory authorities' determination
- Sponsor's determination

If the study is prematurely terminated, the Principal Investigator (PI) will promptly inform study participants and the Institutional Review Board (IRB) and regulatory authorities as applicable. Study participants will be contacted, as applicable, and be informed of changes to study visit schedule. The PI will assure appropriate follow-up for the participants, as necessary. The sponsor will notify regulatory authorities as applicable.

#### 10.1.3 Confidentiality and Privacy

Participant confidentiality is strictly held in trust by the participating investigators, their staff, and the sponsor(s) and their agents. This confidentiality is extended to cover clinical information relating to participants, test results of biological samples and genetic tests, and all other information generated during participation in the study. No identifiable information concerning participants in

DMID/NIAID/NIH 

the study will be released to any unauthorized third party. Participant confidentiality will be maintained when study results are published or discussed in conferences.

The study monitor, other authorized representatives of the sponsor, representatives of the Institutional Review Board (IRB), and/or regulatory agencies may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical study site will permit access to such records.

All source records including electronic data will be stored in secured systems in accordance with institutional policies and federal regulations. All study data and research specimens that leave the site (including any electronic transmission of data) will be identified only by a coded number that cannot be linked to a participant.

As this research is funded by the NIH, it is covered by NIH policy which effectively issues the research a Certificate of Confidentiality. By this policy, researchers cannot be forced to disclose or provide, in any Federal, State, or local civil, criminal, administrative, legislative, or other proceeding, the name of such individual or any such information, document, or biospecimen that contains identifiable, sensitive information about the individual and that was created or compiled for purposes of the research, unless such disclosure or use is made with the consent of the individual to whom the information, document, or biospecimen pertains.

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects, like this study, or for information that must be released in order to meet the requirements of the FDA.

A Certificate of Confidentiality does not prevent the participant from voluntarily releasing information about themselves or their involvement in this research. If any person or agency obtains a written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

The Certificate of Confidentiality does not prevent the researchers from reporting without the participant's consent, information that would identify the participant as a participant in the research project regarding matters that must be legally reported including child and elder abuse, sexual abuse, or wanting to harm themselves or others.

The release of individual private information or specimens for other research will only occur if consent was obtained from the individual or the parent(s) or LAR of the adolescent participants to whom the information, document, or biospecimen pertains, *or* for the purposes of other research that the release is in compliance with applicable Federal regulations governing the protection of human participants in research.

DMID/NIAID/NIH 

# 10.1.4 Secondary Use of Stored Specimens and Data

#### 10.1.4.1 Samples for Secondary Research

#### **Repository Research Sample**

To participate in this study, adult participants and the parent or LAR of adolescent participants will be asked for consent for storage of samples for secondary use. Samples will be stored indefinitely at a DMID-designated storage facility. Each sample will be encoded (labeled) only with a barcode and a unique tracking number to protect participant confidentiality. Secondary research with coded samples and data may occur, however, participant confidentiality will be maintained as described for this protocol. An IRB review of the secondary research using coded specimens is required.

Repository Research Samples, upon written request and approval from DMID and any approvals required by the site, may be shared for secondary research with investigators at the participating site, with researchers at other sites or other institutions, or company-designated research laboratories. The samples will not be sold or used directly for production of any commercial product. DMID will authorize shipment from the repository.

Reports from secondary research will not be kept in the participants' health records or shared with participants, unless required by law. Reports will not be sent to the specimen repository. The participant's decision for secondary research can be changed at any time by notifying the study doctors or nurses in writing. If the participant changes his/her decision, the samples will be destroyed if the samples have not been used for research or released for a specific research project.

#### 10.1.4.2 Data Sharing for Secondary Research

Data from this study may be used for secondary research. Individual participant data collected during the trial that are sufficient to reanalyzed primary and secondary endpoints will be made available after deidentification. The SAP and Analytic Code will also be made available. This data will be available following publication, with no end date. The data will be made available to researchers who provide a methodologically sound proposal. The data will be available for any purpose outlined in the approved proposal. Proposals should be directed to DMID. To gain access, data requestors will need to sign a data access agreement. The investigator may request removal of data on individual study participants from NIH data repositories in the event that a research participant withdraws or changes his or her consent. However, data that have been distributed for approved research use cannot be retrieved.

#### **10.1.5** Key Roles and Study Governance

This is a multi-site clinical trial and as such, all study team members and roles are listed in the Manual of Procedures (MOP).

# 10.1.6 Safety Oversight

For information regarding safety oversite for each study stage, see the corresponding appendix.

DMID/NIAID/NIH 

# 10.1.7 Clinical Monitoring

Clinical site monitoring is conducted to ensure that the rights and well-being of trial participants are protected, that the reported trial data are accurate, complete, and verifiable. Clinical Monitoring ensures that the conduct of the trial is in compliance with the currently approved protocol/amendment(s), International Council for Harmonisation (ICH), Good Clinical Practice, and with applicable regulatory requirement(s) and sponsor requirements.

Monitoring for this study will be overseen by NIAID/DMID and conducted by NIAID/DMID contractors. Details of clinical site monitoring are documented in a Clinical Monitoring Plan (CMP). The CMP describes in detail who will conduct the monitoring, at what frequency monitoring will be done, at what level of detail monitoring will be performed, and the distribution of monitoring reports. Monitoring visits will include, but are not limited to, review of regulatory files, investigational product administration and accountability records, eCRFs, informed consent, parental permission and assent forms, medical and laboratory reports, site study storage records, training records, and protocol and GCP compliance. Site monitors will have access to each participating site, study personnel, and all study documentation according to the NIAID or DMID-approved site monitoring plan. Study monitors will meet with site principal investigators (or designee) to discuss any problems and outstanding issues and will document site visit findings and discussions.

# 10.1.8 Quality Assurance and Quality Control

Quality control (QC) and quality assurance (QA) activities are essential to the safety of participants, and the reliability of study data. Each site participating in the study is responsible for integrating quality control checks throughout the study and implementing a QA Checklist or Clinical Quality Management Plan (CQMP). The site will conduct the following:

- 1. Routine internal QC and QA activities for the purposes of measuring, documenting and reporting study conduct, protocol adherence, human participants' protections, and reliability of the protocol-driven data collected.
- 2. Processes for addressing data quality issues (i.e., collecting, recording), and reporting findings in a timely manner.
- 3. Identify systemic issues (e.g., protocol or human participant protections non-compliance), and implementation and evaluation of Corrective and Preventative Action Plan (CAPA) procedures, if applicable.

#### 10.1.9 Data Handling and Record Keeping

## 10.1.9.1 Data Collection and Management Responsibilities

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site investigator. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported. All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data.

DMID/NIAID/NIH 

#### 10.1.9.2 Data Coordinating Center / Biostatistician Responsibilities

The data coordinating center for this study will be responsible for data management, quality review, analysis, and reporting of the study data. Adverse events and medical history will be coded according to the MedDRA dictionary. Concomitant medications will be coded according to the WHO Drug dictionary. At the end of the study, a copy of all datasets including annotated case report forms and data dictionary will be provided to DMID.

A separate Study Data Standardization Plan (SDSP) will be developed which describes the technical recommendations for the submission of human study data and related information in a standardized electronic format throughout product development.

#### 10.1.9.3 Data Capture Methods

Clinical research data, including, but not limited to, AE/SAEs, concomitant medications, medical history, physical assessments will be abstracted from the source documentation and/or collected on source document worksheet by study personnel then entered into an eCRFs via a 21 CFR Part 11-compliant internet data entry system provided by the study data coordinating center. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate.

The IND Sponsor is responsible for review of data collection tools and processes, and review of data and reports.

Study data will be collected on paper CRFs and then entered into the eCRF or data will be entered directly into the eCRF.

#### 10.1.9.4 Study Record Retention

For information regarding study record retention for each study stage, see the corresponding appendix.

#### 10.1.9.5 Source Records

Source data are all information, original records of clinical findings, observations, or other activities documented in a clinical trial necessary for the reconstruction and evaluation of the trial. Each participating site will maintain appropriate medical and research records for this trial, in compliance with ICH GCP, regulatory, and institutional requirements. Data recorded in the electronic case report form (eCRF) derived from source documents should be consistent with the data recorded on the source documents. Data entered directly into the eCRFs will be considered the source document. All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data.

Interview of participants is sufficient for obtaining medical history. Solicitation of medical records from the participant's primary care provider is not required.

DMID/NIAID/NIH 

#### 10.1.10 Protocol Deviations

A protocol deviation is any noncompliance with the clinical trial protocol, any process that is noted in the protocol and refers to details in the MOP, or GCP requirements.

The noncompliance may be either on the part of the participant, the investigator, or the study site staff. Following a deviation(s), corrective actions should be developed by the site and implemented promptly. All individual protocol deviations will be addressed in participant study records.

It is the responsibility of the site principal investigator and personnel to use continuous vigilance to identify and report deviations within five working days of identification of the protocol deviation, or within five working days of the scheduled protocol-required activity. All deviations must be promptly reported to DMID per the protocol deviation reporting procedures. Protocol deviations must be sent to the local IRB/IEC per their guidelines. The site principal investigator and personnel are responsible for knowing and adhering to their IRB requirements.

#### **10.1.11** Publication and Data Sharing Policy

## 10.1.11.1 Human Data Sharing Plan

All NIH protocols are required to have a Data Sharing Plan describe provisions for protecting the participants' privacy and the confidentiality of the data. This study will be conducted in accordance with the following publication and data sharing policies and regulations:

National Institutes of Health (NIH) Public Access Policy, which ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive <u>PubMed Central</u> upon acceptance for publication.

As of January 2018, all clinical trials supported by the NIH must be registered on ClinicalTrials.gov, no later than 21 days after the enrollment of the first participant. Results of all clinical trials supported by the NIH, generally, need to be submitted no later than 12 months following the primary completion date. As part of the result posting, a copy of this protocol and a copy of the Statistical Analysis Plan will be posted on ClinicalTrials.gov.

#### 10.1.11.2 Genomic Data Sharing Plan

Not Applicable.

#### **10.1.11.3** Publication

This study will comply with the NIH Public Access Policy, which ensures that the public has access to the published results of NIH funded research. As such, the final peer-reviewed journal manuscripts will be accessible to the public on PubMed Central no later than 12 months after publication.

#### **10.1.12** Conflict of Interest Policy

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and

DMID/NIAID/NIH 

managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct of this trial. DMID has established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

### **10.2** Additional Considerations

#### **10.2.1** Research Related Injuries

For any potential research related injury, the site principal investigator or designee will assess the participant. The site principal investigator should then determine if an injury occurred as a direct result of the tests or treatments that are done for this trial. As needed, referrals to appropriate health care facilities will be provided to the participant. No financial compensation will be provided by the NIAID, NIH, or the federal government to the participant, for any injury suffered due to participation in this trial.

#### **10.2.2 PREP Act**

The study vaccine and the efforts for this clinical trial are covered under the Public Readiness and Emergency Preparedness Act (PREP Act). The PREP Act applies under the terms of the PREP Act declaration in place for smallpox/orthopoxvirus countermeasures for activities conducted pursuant federal agreements federal to programs (ref: www.federalregister.gov/documents/2015/12/09/2015-31092/smallpox-medicalcountermeasures-amendment). JYNNEOS is used under an IND for mpox pursuant to a federal agreement/program and is therefore covered under the PREP Act. The PREP Act covers persons (such as manufacturers, distributers, program planners, and other qualified persons who prescribe, administer or dispense study product) are immune from liability from the administration, or use of a covered countermeasure, such as JYNNEOS. The PREP Act provides immunity for covered persons from liability, unless the injury was caused by willful misconduct.

The PREP Act also established the Countermeasures Injury Compensation Program (CICP) to provide compensation for serious injuries or death that occur as the direct result of the administration or use of certain countermeasures. Any requests for compensation must be filed within one year of the administration or use of the covered countermeasure. Requests for Benefits must be made to the Health Resources and Services Administration's (HRSA) Countermeasures Injury Compensation Program (http://www.hrsa.gov/cicp/) by filing a Request for Benefits Form and all required medical records and supporting documentation. Additional information on filing a Request for Benefits is available on the CICP's website at http://www.hrsa.gov/cicp/. Compensation may then be available for reasonable and necessary medical benefits, lost wages and/or death benefits to eligible individuals for certain injuries in accordance with regulations published by the Secretary of HHS (found at 42 CFR part 110).

If an individual suffers a serious physical injury or death from the administration or use of a covered countermeasure in this study, the individual, the individual's legal or personal representative, the administrator/executor of a deceased individual's estate, or certain survivors may request benefits from the CICP. A serious physical injury means an injury that warranted hospitalization (whether

DMID/NIAID/NIH 
or not the person was actually hospitalized) or that led to a significant loss of function or disability. The CICP is the payer of last resort. This means that it only covers expenses or provides benefits that other third-party payers (such as health insurance, the Department of Veterans Affairs, or Workers' Compensation programs) do not have an obligation to pay.

If the Secretary of HHS does not make a final determination on the individual's request within 240 days, or if the individual decides not to accept the compensation, the injured individual or his representative may pursue a tort claim in the US District Court for the District of Columbia, but only if the claim involves willful misconduct and meets the other requirements for suit under the PREP Act. Any award is reduced by any public or private insurance or worker's compensation available to the injured individual. Awards for non-economic damages, such as pain, suffering, physical impairment, mental anguish, and loss of consortium are also limited. If the individual accepts compensation, or if there is no willful misconduct, then the individual does not have a tort claim that can be filed in a US Federal or a State court.

DMID/NIAID/NIH 

# 10.3 Abbreviations

| AE | Adverse Event |
|--------|-----------------------------------------------------|
| AESI | Adverse Event of Special Interest |
| BLA | Biologics License Application |
| BP | Blood Pressure |
| CAPA | Corrective and Preventative Action Plan |
| CEF | Chicken Embryo Fibroblast |
| CFR | Code of Federal Regulations |
| CI | Confidence Interval |
| CICP | Countermeasures Injury Compensation Program |
| CMP | Clinical Monitoring Plan |
| CMS | Clinical Material Services |
| CQMP | Clinical Quality Management Plan |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| CSR | Clinical Study Report |
| CSIC | enmour study resport |
| DHHS | Department of Health and Human Services |
| DMID | Division of Microbiology and Infectious Diseases |
| DSMB | Data and Safety Monitoring Board |
| BSIVIB | Data and Salety Memoring Deard |
| eCRF | Electronic Case Report Form |
| EUA | Emergency Use Authorization |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Amendments Act of 2007 |
| FWA | Federalwide Assurance |
| GCP | Good Clinical Practice |
| GMFR | Geometric Mean Fold Rise |
| HHS | Health and Human Services |
| HIPAA | Health Insurance Portability and Accountability Act |
| HR | Heart Rate |
| HRSA | Health Resources and Services Administration |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| ICMJE | International Committee of Medical Journal Editors |
| ID | Intradermal |
| IEC | Independent or Institutional Ethics Committee |
| IND | Investigational New Drug Application |
| IRB | Institutional Review Board |
| ISO | International Organization for Standardization |
| ITT | Intention-To-Treat |
| LAR | Legal Authorized Representative |
| MAAE | Medically Attended Adverse Event |

| MedDRA | Medical Dictionary for Regulatory Activities |
|--------|-------------------------------------------------------|
| MITT | Modified Intent to Treat |
| MOP | Manual of Procedures |
| MPXV | Monkeypox Virus |
| N | Number (typically refers to participants) |
| NDA | New Drug Application |
| NI | Non - Inferior |
| NIAID | National Institute of Allergy and Infectious Diseases |
| NIH | National Institutes of Health |
| OHRP | Office for Human Research Protections |
| PHI | Protected Health Information |
| PI | Principal Investigator |
| PP | Per Protocol |
| PREP | Public Readiness and Emergency Preparedness Act |
| QA | Quality Assurance |
| QC | Quality Control |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SC | Subcutaneous |
| SDCC | Statistical and Data Coordinating Center |
| SDSP | Study Data Standardization Plan |
| SOA | Schedule of Activities |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TCID | Mean Tissue Culture Infectious Dose |
| TFF | Tangential Flow Filtration |
| UP | Unanticipated Problem |
| US | United States |
| WHO | World Health Organization |

# 10.4 Protocol Amendment History

| Versio | Date | Description of | Brief Rationale |
|---|---|---|---|
| n | | Change | |
| 7.0 | 5/23/2 | -Updated analysis | -Will allow for Stage 2 interim Clinial Study Report |
| | 4 | plan for Stage 2 | to be produced to inform public health needs. |
| 6.0 | 8/31/2 | -Updated interim | - Stage 1 interim data review of immunogenicity |
| | 3 | immunogenicity | may be performed after all participants have |
| | | analysis plan for | completed Day 181, rather than Day 43 |
| | | Stage 1 | -Stage 2 Objectives and Endpoints table did not list |
| | | -Corrected an error in | Day 1 as a timepoint for Vaccinia Virus specific |
| | | the Stage 2 Objectives and | PRNT assay for first Secondary Objective -Will allow for Stage 2 interim immunogenicity |
| | | Endpoints table | analysis |
| | | -Updated interim | -Guidance for disposition of unused and used study |
| | | immunogenicity | product in Stage 2 will be provided by DMID. |
| | | analysis plan for | |
| | | Stage 2 | |
| | | -Revised language in | |
| | | main section of | |
| | | protocol regarding | |
| | | study product | |
| | | disposition -Clarified Protocol | |
| | | Amendment History | |
| | | table for Version 5.0 | |
| | | -Fixed typo in Stage | |
| | | 2 SOA footnotes | |
| 5.0 | 4/13/2 | Allow Day 57 visit in | -Will allow for phone/virtual visit at Day 57 if no |
| | 023 | Stage 2 to be done by | ongoing vaccine site skin changes at Day 43 visit |
| | | phone/virtual visit in | -Per FDA approval of labeling change dated |
| | | certain scenarios. | 4/14/2023 |
| | | -Added that a Day 43 | https://www.fda.gov/media/166224/download?utm |
| | | targeted physical exam (at least | _medium=email&utm_source=govdelivery |
| | | assessment of | |
| | | vaccination site) is | |
| | | required | |
| | | -JYNNEOS MVA- | |
| | | BN vaccine thaw | |
| | | time increased from | |
| | | 12 hours to 4 weeks. | |

| | | | • |
|---|---|---|---|
| 4.0 | 2/28/2 | Adjustment of sample size and | Revisions made in response to FDA and DSMB feedback. Exclusion criteria revised to reduce |
| | | revision to exclusion criteria for Stage 2. | potential for confounding of safety data. |
| | | - | |
| 3.0 | 1/13/2 | Addition of new stage to the protocol, see Appendix B of this document. | New stage of the platform trial to evaluate safety and immunogenicity of the standard dose regimen of JYNNEOS in adolescents ages 12 to 17 years, inclusive compared to adults. |
| 2.0 | 9/22/2 | For description of changes to Version 1.0, see document on study website | Clarification of study procedures and correction of internal inconsistencies within the protocol |

## 11. REFERENCES

1. Pan American Health Organization. Mpox (monkeypox) outbreak - 2022. (https://www.paho.org/en/mpox-monkeypox-outbreak-2022#:~:text=On%2023%20July%202022%2C%20the,of%20International%20Concern%20(PHEIC)).

- 2. Centers for Disease Control and Prevention. 2022 Mpox Outbreak Global Map. (https://www.cdc.gov/poxvirus/monkeypox/response/2022/world-map.html).
- 3. Outbreak News Today. England: Monkeypox case confirmed, Patient had recent travel history from Nigeria. (https://outbreaknewstoday.com/england-monkeypox-case-confirmed-patient-had-recent-travel-history-from-nigeria-68610/).
- 4. McCollum AM, Damon IK. Human monkeypox. Clin Infect Dis 2014;58(2):260-7. DOI: 10.1093/cid/cit703.
- 5. Grant R, Nguyen LL, Breban R. Modelling human-to-human transmission of monkeypox. Bull World Health Organ 2020;98(9):638-640. DOI: 10.2471/BLT.19.242347.
- 6. Gong Q, Wang C, Chuai X, Chiu S. Monkeypox virus: a re-emergent threat to humans. Virol Sin 2022. DOI: 10.1016/j.virs.2022.07.006.
- 7. Rimoin AW, Mulembakani PM, Johnston SC, et al. Major increase in human monkeypox incidence 30 years after smallpox vaccination campaigns cease in the Democratic Republic of Congo. Proc Natl Acad Sci U S A 2010;107(37):16262-7. DOI: 10.1073/pnas.1005769107.
- 8. World Health Organization. Emergence of monkeypox in West Africa and Central Africa, 1970-2017. Wkly Epidemiol Rec 2018;93(11):125-32. (https://www.ncbi.nlm.nih.gov/pubmed/29546750).
- 9. Centers for Disease Control and Prevention. Multistate outbreak of monkeypox--Illinois, Indiana, and Wisconsin, 2003. MMWR Morb Mortal Wkly Rep 2003;52(23):537-40. (https://www.ncbi.nlm.nih.gov/pubmed/12803191).
- 10. Erez N, Achdout H, Milrot E, et al. Diagnosis of Imported Monkeypox, Israel, 2018. Emerg Infect Dis 2019;25(5):980-983. DOI: 10.3201/eid2505.190076.
- 11. Yong SEF, Ng OT, Ho ZJM, et al. Imported Monkeypox, Singapore. Emerg Infect Dis 2020;26(8):1826-1830. DOI: 10.3201/eid2608.191387.
- 12. Rao AK, Schulte J, Chen TH, et al. Monkeypox in a Traveler Returning from Nigeria Dallas, Texas, July 2021. MMWR Morb Mortal Wkly Rep 2022;71(14):509-516. DOI: 10.15585/mmwr.mm7114a1.
- 13. Vaughan A, Aarons E, Astbury J, et al. Human-to-Human Transmission of Monkeypox Virus, United Kingdom, October 2018. Emerg Infect Dis 2020;26(4):782-785. DOI: 10.3201/eid2604.191164.
- 14. Hobson G, Adamson J, Adler H, et al. Family cluster of three cases of monkeypox imported from Nigeria to the United Kingdom, May 2021. Euro Surveill 2021;26(32). DOI: 10.2807/1560-7917.ES.2021.26.32.2100745.
- 15. Mauldin MR, McCollum AM, Nakazawa YJ, et al. Exportation of Monkeypox Virus From the African Continent. J Infect Dis 2022;225(8):1367-1376. DOI: 10.1093/infdis/jiaa559.
- 16. Yinka-Ogunleye A, Aruna O, Dalhat M, et al. Outbreak of human monkeypox in Nigeria in 2017-18: a clinical and epidemiological report. Lancet Infect Dis 2019;19(8):872-879. DOI: 10.1016/S1473-3099(19)30294-4.

DMID/NIAID/NIH 

17. Durski KN, McCollum AM, Nakazawa Y, et al. Emergence of Monkeypox - West and Central Africa, 1970-2017. MMWR Morb Mortal Wkly Rep 2018;67(10):306-310. DOI: 10.15585/mmwr.mm6710a5.

- 18. Constantino AK. Health officials confirm first U.S. case of monkeypox virus this year in Massachusetts. CNBC Health & Science, 2022.
- 19. Department of Health and Human Services. Determination that a public health emergency exists. (https://aspr.hhs.gov/legal/PHE/Pages/monkeypox-4Aug22.aspx).
- 20. Vollmar J, Arndtz N, Eckl KM, et al. Safety and immunogenicity of IMVAMUNE, a promising candidate as a third generation smallpox vaccine. Vaccine 2006;24(12):2065-70. DOI: 10.1016/j.vaccine.2005.11.022.
- 21. Frey SE, Wald A, Edupuganti S, et al. Comparison of lyophilized versus liquid modified vaccinia Ankara (MVA) formulations and subcutaneous versus intradermal routes of administration in healthy vaccinia-naive subjects. Vaccine 2015;33(39):5225-34. DOI: 10.1016/j.vaccine.2015.06.075.
- 22. Wilck MB, Seaman MS, Baden LR, et al. Safety and immunogenicity of modified vaccinia Ankara (ACAM3000): effect of dose and route of administration. J Infect Dis 2010;201(9):1361-70. DOI: 10.1086/651561.
- World Health Organization. Multi-country outbreak of mpox, External situation report #11. Emergency Situational Update. Geneva, Switzerland: December 1, 2022. (https://www.who.int/publications/m/item/multi-country-outbreak-of-mpox--external-situation-report--11---1-december-2022).
- 24. Hennessee I SV, McArdle CE, et al. . Epidemiologic and Clinical Features of Children and Adolescents Aged <18 Years with Monkeypox United States, May 17–September 24, 2022. MMWR Morb Mortal Wkly Rep 2022(71):1407–1411. DOI: http://dx.doi.org/10.15585/mmwr.mm7144a4.
- 25. Hutin W, R. J., Malfait, P., Pebody, R., Loparev, V. N., Ropp, S. L., Rodriguez, M., Knight, J. C., Tshioko, F. K., Khan, A. S., Szczeniowski, M. V., & Esposito, J. J. Outbreak of Human Monkeypox, Democratic Republic of Congo, 1996 to 1997. . Emerging Infectious Diseases 2001;7(3):434–438. DOI: https://doi.org/10.3201/eid0703.017311.
- 26. Ježek Z, Szczeniowski M, Paluku KM, Mutombo M. Human Monkeypox: Clinical Features of 282 Patients. The Journal of Infectious Diseases 1987;156(2):293-298. DOI: 10.1093/infdis/156.2.293.
- 27. US Food and Drug Administration. Summary Basis for Regulatory Action (https://www.fda.gov/media/131802/download).
- 28. Overton ET, Lawrence SJ, Wagner E, et al. Immunogenicity and safety of three consecutive production lots of the non replicating smallpox vaccine MVA: A randomised, double blind, placebo controlled phase III trial. PLoS One 2018;13(4):e0195897. DOI: 10.1371/journal.pone.0195897.
- 29. US Food and Drug Administration. Fact Sheet for Healthcare Providers Administering Vaccine: Emergency Use Authorization of JYNNEOS (Smallpox and Monkeypox Vaccine, Live, Non-replicating) for Prevention of Monkeypox Disease in Individuals Determined to Be at High Risk for Monkeypox Infection. 2022.
- 30. Elizaga ML VS, Marovich MA, Sato AH, Lawrence DN, Chaitman BR, Frey SE, Keefer MC; MVA Cardiac Safety Working Group. Prospective surveillance for cardiac adverse events in healthy adults receiving modified vaccinia Ankara vaccines: a systematic review. PLoS One 2013;8(1):e54407. DOI: 10.1371/journal.pone.0054407.

DMID/NIAID/NIH 

31. Scriba TJ, Tameris, M., Mansoor, N., Smit, E., van der Merwe, L., Isaacs, F., Keyser, A., Moyo, S., Brittain, N., Lawrie, A., Gelderbloem, S., Veldsman, A., Hatherill, M., Hawkridge, A., Hill, A.V.S., Hussey, G.D., Mahomed, H., McShane, H. and Hanekom, W.A., . Modified vaccinia Ankara-expressing Ag85A, a novel tuberculosis vaccine, is safe in adolescents and children, and induces polyfunctional CD4+ T cells. . Eur J Immunol 2010;40:279-290. (https://doi.org/10.1002/eji.200939754).

- 32. Anywaine Z BH, Anzala O, Mutua G, Sirima SB, Eholie S, et al. . Safety and immunogenicity of 2-dose heterologous Ad26.ZEBOV, MVA-BN-Filo Ebola vaccination in children and adolescents in Africa: A randomised, placebo-controlled, multicentre Phase II clinical trial. PLoS Medicine 2022;19(1):e1003865. (https://doi.org/10.1371/journal.pmed.1003865).
- 33. Afolabi MO ID, Manno D, et al. Safety and immunogenicity of the two-dose heterologous Ad26.ZEBOV and MVA-BN-Filo Ebola vaccine regimen in children in Sierra Leone: a randomised, double-blind, controlled trial. Lancet Infect Dis 2022;22:110-122.
- 34. Suter M, Meisinger-Henschel C, Tzatzaris M, et al. Modified vaccinia Ankara strains with identical coding sequences actually represent complex mixtures of viruses that determine the biological properties of each strain. Vaccine 2009;27(52):7442-50. DOI: 10.1016/j.vaccine.2009.05.095.
- 35. Stittelaar KJ, Kuiken T, de Swart RL, et al. Safety of modified vaccinia virus Ankara (MVA) in immune-suppressed macaques. Vaccine 2001;19(27):3700-9. DOI: 10.1016/s0264-410x(01)00075-5.
- 36. Overton ET, Stapleton J, Frank I, et al. Safety and Immunogenicity of Modified Vaccinia Ankara-Bavarian Nordic Smallpox Vaccine in Vaccinia-Naive and Experienced Human Immunodeficiency Virus-Infected Individuals: An Open-Label, Controlled Clinical Phase II Trial. Open Forum Infect Dis 2015;2(2):ofv040. DOI: 10.1093/ofid/ofv040.
- 37. Greenberg RN, Overton ET, Haas DW, et al. Safety, immunogenicity, and surrogate markers of clinical efficacy for modified vaccinia Ankara as a smallpox vaccine in HIV-infected subjects. J Infect Dis 2013;207(5):749-58. DOI: 10.1093/infdis/jis753.
- 38. Overton ET, Lawrence SJ, Stapleton JT, et al. A randomized phase II trial to compare safety and immunogenicity of the MVA-BN smallpox vaccine at various doses in adults with a history of AIDS. Vaccine 2020;38(11):2600-2607. DOI: 10.1016/j.vaccine.2020.01.058.
- 39. von Sonnenburg F, Perona P, Darsow U, et al. Safety and immunogenicity of modified vaccinia Ankara as a smallpox vaccine in people with atopic dermatitis. Vaccine 2014;32(43):5696-702. DOI: 10.1016/j.vaccine.2014.08.022.
- 40. Greenberg RN, Hurley MY, Dinh DV, et al. A Multicenter, Open-Label, Controlled Phase II Study to Evaluate Safety and Immunogenicity of MVA Smallpox Vaccine (IMVAMUNE) in 18-40 Year Old Subjects with Diagnosed Atopic Dermatitis. PLoS One 2015;10(10):e0138348. DOI: 10.1371/journal.pone.0138348.
- 41. Cassimatis DC, Atwood JE, Engler RM, Linz PE, Grabenstein JD, Vernalis MN. Smallpox vaccination and myopericarditis: a clinical review. J Am Coll Cardiol 2004;43(9):1503-10. DOI: 10.1016/j.jacc.2003.11.053.
- 42. Department of Health and Human Services. 46.110 Expedited review procedures for certain kinds of research involving no more than minimal risk, and for minor changes in approved research.

DMID/NIAID/NIH 

- (https://www.hhs.gov/ohrp/sites/default/files/ohrp/sachrp/mtgings/2013%20March%20Mtg/approvedexpeditedreviewcategories.pdf).
- 43. von Krempelhuber A, Vollmar J, Pokorny R, et al. A randomized, double-blind, dose-finding Phase II study to evaluate immunogenicity and safety of the third generation smallpox vaccine candidate IMVAMUNE. Vaccine 2010;28(5):1209-16. DOI: 10.1016/j.vaccine.2009.11.030.
- 44. Pittman PR, Hahn M, Lee HS, et al. Phase 3 Efficacy Trial of Modified Vaccinia Ankara as a Vaccine against Smallpox. N Engl J Med 2019;381(20):1897-1908. DOI: 10.1056/NEJMoa1817307.

DMID/NIAID/NIH 

## **APPENDIX A – STAGE 1: DOSE SPARING STUDY IN ADULTS**

Stage 1 began enrollment on September 7, 2022 and completed enrollment on October 12, 2022. This appendix contains Version 2.0 dated September 22, 2022 which is also found on the study website.

# **TABLE OF CONTENTS**

| TABLE OF O | CONTENTS | 46 |
|------------|--------------------------------------------|----|
| 1.1 Sy | nopsis | 50 |
| 1.2 Sc. | hedule of Activities (SOA) | 52 |
| 1.3 Stu | ıdy Schema | 53 |
| 2. INTROI | DUCTION | 53 |
| 2.1 Stu | ıdy Rationale | 53 |
| 2.2 Ba | ckground | 53 |
| 2.3 Ris | sk/Benefit Assessment | 55 |
| 2.3.1 | Known Potential Risks | 55 |
| 2.3.2 | Known Potential Benefits | |
| 2.3.3 | Assessment of Potential Risks and Benefits | 59 |
| 3. OBJEC | TIVES AND ENDPOINTS | 60 |
| 4. STUDY | DESIGN | 61 |
| 4.1 Ov | rerall Design | 61 |
| 4.2 Sc | ientific Rationale for Study Design | 61 |
| 4.3 Jus | stification for Dose | 61 |
| 5. STUDY | POPULATION | 61 |
| 5.1 Inc | clusion Criteria | 62 |
| | clusion Criteria | |
| 5.2.1 | Exclusion of Specific Populations. | |
| | clusion of Vulnerable Participants | |
| | Festyle Considerations | |
| | reen Failures | |
| | rategies for Recruitment and Retention | 64 |
| 5.6.1 | Recruitment | |
| 5.6.2 | Retention | |
| 5.6.3 | Compensation Plan for Participants | |
| 5.6.4 | Costs | 65 |
| 6. STUDY | PRODUCT | 65 |
| | ady Product(s) and Administration | |
| 6.1.1 | Study Product Description. | |
| 6.1.2 | Dosing and Administration | |
| 6.1.3 | Dose Escalation | 66 |

| 6.1.4 | Dose Modifications | .66 |
|---|---|---|
| 6.1.5 | Criteria for Redosing | .66 |
| 6.2 Prep | paration/Handling/Storage/Accountability | .66 |
| 6.2.1 | Acquisition and Accountability | .66 |
| 6.2.2 | Formulation, Appearance, Packaging, and Labeling Product: JYNNEOS (MVA | -BN |
| vaccine) | 67 | |
| 6.2.3 | Product Storage and Stability Product: JYNNEOS (MVA-BN vaccine) | .67 |
| 6.2.4 | Preparation | |
| 6.3 Mea | asures to Minimize Bias: Randomization and Blinding | .68 |
| 6.3.1 | Treatment Assignment Procedures. | .68 |
| 6.3.2 | Randomization | .68 |
| 6.3.3 | Blinding and Masking Procedures | .68 |
| 6.4 Stud | dy Intervention Compliance | .68 |
| 6.5 Cor | comitant Therapy | |
| 6.5.1 | Rescue Medicine | .69 |
| 7. STUDY | INTERVENTION DISCONTINUATION AND PARTICIPANT | |
| | ATION/WITHDRAWAL | 69 |
| | ting Criteria and Discontinuation of Study Intervention | .69 |
| 7.1.1 | Study Halting Criteria | |
| 7.1.2 | Individual Halting Criteria | |
| 7.1.3 | Follow up for participants that discontinued study intervention | |
| 7.2 Los | t to Follow-Up | .71 |
| 8. STUDY | ASSESSMENTS AND PROCEDURES | .71 |
| 8.1 Scr | eening Procedures | 71 |
| 8.1.1 | Procedures to be Followed in the Event of Abnormal Clinical Laboratory Test V | |
| | al Clinical Findings During Screening | |
| 8.1.2 | Sick Visit | |
| | nunogenicity Assessments | |
| 8.2.1 | | |
| 8.2.2 | Exploratory Assessments | |
| | ety and Other Assessments | |
| 8.3.1 | Procedures to be Followed in the Event of Abnormal Clinical Laboratory Test V | |
| | al Clinical Findings During Conduct of the Trial | |
| | Verse Events and Serious Adverse Events | |
| 8.4.1 | Definition of Adverse Events (AE) | |
| 8.4.2 | Definition of Serious Adverse Events | |
| 8.4.3 | Classification of an Adverse Event | |
| 8.4.4 | Time Period and Frequency for Event Assessment and Follow-Up | |
| 8.4.5 | Adverse Event Reporting | |
| 8.4.6 | Serious Adverse Event Reporting | |
| 8.4.7 | Reporting Events to Participants | |
| 8.4.8 | Adverse Events of Special Interest (AESI) | |
| 8.4.9 | Reporting of Pregnancy | |
| | Reporting of Freguency | |
| 8.5 Una | inticipated Problems | 80 |

| 8.5.2 | Unanticipated Problem Reporting | 80 |
|---|---|---|
| 8.5.3 | Reporting Unanticipated Problems to Participants | 81 |
| 9. STATIS | TICAL CONSIDERATIONS | 81 |
| 9.1 Sta | tistical Hypotheses | 81 |
| | nple Size Determination | |
| | tistical Analyses | |
| 9.3.1 | General Methodology | |
| 9.3.2 | Timing of Analyses | 83 |
| 9.3.3 | Populations for Analyses | |
| 9.3.4 | Baseline Characteristics and Participant Disposition | 84 |
| 9.3.5 | Immunogenicity Analyses | 84 |
| 9.3.6 | Safety Analyses | 85 |
| 10. SUPPOR | RTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | 86 |
| | gulatory, Ethical, and Study Oversight Considerations | |
| 10.1.1 | Informed Consent Process. | |
| 10.1.2 | Study Termination and Closure | |
| 10.1.3 | Confidentiality and Privacy | |
| 10.1.4 | Secondary Use of Stored Specimens and Data | |
| 10.1.5 | Key Roles and Study Governance | |
| 10.1.6 | Safety Oversight. | |
| 10.1.7 | Clinical Monitoring. | |
| 10.1.8 | Quality Assurance and Quality Control | |
| 10.1.9<br>10.1.10 | Data Handling and Record Keeping | |
| 10.1.10 | Protocol Deviations Publication and Data Sharing Policy | |
| 10.1.11 | Conflict of Interest Policy | |
| | ditional Considerations | |
| 10.2 Au | Research Related Injuries | |
| 10.2.1 | PREP Act | |
| | ENCES | |
| ii. Referen | | |
| | LIST OF TABLES | |
| Table 1 Sche | dule of Activities (SOA) | 52 |
| | y Schema | |
| | Subcutaneous Dosing Trials | |
| | A-BN Compared to ACAM2000 | |
| | Intradermal Dosing Compared to Subcutaneous | |
| | y Arms | |
| | er calculations | |
| | dard deviation estimatesdard deviation estimates | |
| 1 auit 7. Stall | uatu ucviation estimates | o. |

# **LIST OF FIGURES**

No table of figures entries found.

## 1. PROTOCOL SUMMARY

## 1.1 Synopsis

#### Rationale

Since the first case was identified four months ago, monkeypox has rapidly spread to 85 non-endemic countries, marking the first time monkeypox has spread widely outside Central and West Africa. To prevent further spread of this outbreak, MVA-BN vaccine is being offered to individuals at high risk. However, there is a global vaccine shortage and increasing vaccine supply will take time. This study will evaluate dose sparing strategies to extend the vaccine supply during this global public health crisis.

#### **Study Design**

This study is a Phase 2 randomized, open-label, non-placebo controlled, multi-site clinical trial that will evaluate the immunogenicity and safety of two, dose sparing strategies including one- fifth  $(2x10^7)$  and one-tenth  $(1x10^7)$  of the standard dose of MVA-BN (JYNNEOS) administered intradermally (ID) on Day 1 and 29 (Arm 1 and 2, respectively), compared with the standard, licensed regimen of  $1x10^8$  MVA-BN administered subcutaneously (SC) on Day 1 and 29 (Arm 3). At least 210 healthy, vaccinia-naïve adults 18 to 50 years of age will be enrolled and randomized 1:1:1 to one of three study arms. There will be eight study visits (plus an optional screening visit) with the last visit at approximately one year after the first study vaccination.

Participants reporting monkeypox-like illness and who have a laboratory-confirmed monkeypox (i.e., a positive diagnostic test for monkeypox) will be seen at a sick visit.

## **Primary Objectives**

- To determine if peak (Day 43) humoral immune responses following an ID regimen of 2 x 10<sup>7</sup> TCID<sub>50</sub> MVA-BN are non-inferior to the licensed regimen of 1 x 10<sup>8</sup> MVA-BN administered SC.
- To determine if peak (Day 43) humoral immune responses following an ID regimen of 1 x 10<sup>7</sup> TCID<sub>50</sub> MVA-BN are non-inferior to the licensed regimen of 1 x 10<sup>8</sup> MVA-BN administered SC

For a full list of Objectives/Endpoints, see corresponding section of the protocol.

#### **Inclusion Criteria**

See inclusion criteria in corresponding section of the protocol.

#### **Exclusion Criteria**

See exclusion criteria in corresponding section of the protocol.

#### **Study Phase**

Phase 2

#### **Study Population**

DMID/NIAID/NIH 

The study population will be healthy, vaccinia-naïve, non-pregnant, non-breastfeeding adults 18 to 50 years of age. Participants with stable chronic medical conditions including those with controlled HIV infection can participate. The study will attempt to enroll a representative study population that is proportional to those affected by the disease and demographically diverse.

#### Sites

Up to 10 US clinical research sites.

#### **Study intervention**

There will be three study arms in which JYNNEOS will be administered by either ID or SC injection at Day 1 and 29. JYNNEOS is live vaccine produced from the strain Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN), an attenuated orthopoxvirus, that is non-replicating in human cells. It is FDA-approved and licensed as a smallpox and monkeypox vaccine in the United States.

#### **Study Duration**

This study will take approximately 15 months to conduct from study activation to the final participant's last study visit.

#### **Participant Duration**

It will take approximately one year for a participant to complete their participation in the study.

#### Safety

The trial will use study and individual pausing rules. See corresponding section for details. This trial will use a Data Safety Monitoring Board (DSMB) for objective oversight of the study and review for any study pause.

DMID/NIAID/NIH 

## 1.2 Schedule of Activities (SOA)

The trial will include the following activities and procedures at each study visit. Only procedures that contribute to participant eligibility and study objectives and endpoints are included. Refer to Manual of Procedures (MOP) for detailed description of study activities.

**Table 1 Schedule of Activities (SOA)** 

| Procedures | Optional<br>Screening Visit<br>Day -7 to -1 | Enrollment/Baseline<br>Visit 1 Day 1 | Visit 2<br>Day 15 +/- 3 day | Visit 3<br>Day 29 +/- 3 days | Visit 4<br>Day 43 +/- 3 days | Visit 5<br>Day 57 +/- 3 days | Visit 6 Day 90 +/- 5<br>days | Visit 7<br>Day 181 +/- 7 days | Visit 8<br>Day 365 +/- 14 days | Sick/Unscheduled<br>Visit <sup>6</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Informed consent | X | $X^1$ | | | | | | | | |
| Demographics | X | $X^1$ | | | | | | | | |
| Medical history | X | $X^1$ | X | X | X | X | X | X | X | X |
| Randomization | | X | | | | | | | | |
| Vaccine administration | | X | | X | | | | | | |
| Targeted physical exam | X | $X^1$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ |
| Vital signs | X | $X^1$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ |
| Concomitant<br>medication review | X | $X^1$ | X | Х | Х | X | $X^3$ | $X^3$ | | Х |
| SAE/ MAAEs <sup>4</sup> | | All SAE/ | MAAEs, l | Days 1 thi | ough 57 | 1 | Only rela<br>SAE/MA<br>Days 58 - | AEs | | $X^4$ |
| Unsolicited AEs <sup>4</sup> | | Day 1 thr<br>Day 57 | ough Day | 29 and D | ay 29 thro | ough | | | | $X^4$ |
| Solicited (Local and<br>Systemic) AEs | | Day 1 thr<br>Day 15 | | Day 29 tl<br>Day 43 | nrough | | | | | $X^4$ |
| Tolerability<br>Assessment | | | X | | X | | | | | |
| Pregnancy test 5 | Х | $X^1$ | | X | | | | | | |
| Blood volume per visit (ml) | | 32 | 20 | 20 | 32 | 20 | 20 | 20 | 20 | 20 |
| Blood volume total (ml) | | 32 | 52 | 72 | 104 | 124 | 144 | 164 | 184 | 204 |

<sup>&</sup>lt;sup>1</sup> If there is no screening visit, these activities should be conducted at the Day 1 visit prior to randomization. Temperature should be collected on Day 1 and 29 pre-vaccination for all participants.

DMID/NIAID/NIH 

<sup>&</sup>lt;sup>2</sup> A targeted (symptom-driven) physical exam will be done at screening (i.e., screening visit or Day 1), on Days 15, 29, and 43 (at least assessment of vaccination site and presence of skin discoloration and nodules will be done), and as needed in all other visits if interim change in medical status reported by participant. Vital signs will be done at screening and on Day 1 and 29 prior to vaccination and on an as needed basis during all other visits.

<sup>&</sup>lt;sup>3</sup> After Day 57, only concomitant medications that are associated with a related SAE or MAAE (detected through Day 181) and clinically relevant to report, will be recorded in the CRF. An exception to this rule for recording concomitant medications is for sick visits. During sick visits, concomitant medications will be collected.

<sup>&</sup>lt;sup>4</sup> If SAE/MAAE or unsolicited AE are reported during a sick visit and within the reporting window, it will be reported as AE. See more information about collection of AEs in the safety section of the protocol.

Protocol 22-0020
Appendix A
23 May 2024

## 1.3 Study Schema

Table 2 Study Schema

| Arm | Dose of JYNNEOS (MVA-BN) | Route of Administration* | e of Administration* Vaccination Day | |
|---|---|---|---|---|
| | | | Day 1 | Day 29 |
| 1 | 2 x 10 <sup>7</sup> TCID <sub>50</sub> , (0.1 mL) | Intradermal | X | X |
| 2 | $1 \times 10^7 \text{ TCID}_{50}, (0.05 \text{ mL})$ | Intradermal | X | X |
| 3 | 1 x 10 <sup>8</sup> TCID <sub>50</sub> , (0.5 mL) | Subcutaneous | X | X |

<sup>\*</sup>Subcutaneous is administered in the upper arm, intradermal is administered in the volar aspect (inner side) of the forearm.

## 2. INTRODUCTION

## 2.1 Study Rationale

On July 23, 2022, WHO declared the 2022 monkeypox outbreak a public health emergency of international concern (PHEIC). Since the first case of monkeypox was detected in the UK in a returning traveler from Nigeria on May 6, 2022, as of September 2022 the outbreak has rapidly spread to >100 countries or locations worldwide, including 96 that are non-endemic, marking the first time monkeypox has spread widely outside Central and West Africa. In August, the number of confirmed monkeypox cases in the U.S. surpassed that of any other country. To mitigate the consequences of this outbreak, monkeypox vaccine is being offered to individuals considered to be at high risk. However, there is a global vaccine shortage and increasing the supply will take time. This study will evaluate vaccine dose sparing strategies to extend the limited supply during this global public health crisis.

# 2.2 Background

Monkeypox is a reemerging infectious disease caused by Monkeypox virus (MPXV), a large double-stranded DNA virus belonging to the genus, *Orthopoxvirus*. MPXV is a zoonotic orthopoxvirus, primarily transmitted to humans via contact with infected animals, and causing disease similar to smallpox, although with substantially lower mortality. MPXV is endemic to West and Central Africa, where the incidence of human monkeypox cases has increased as much as 20-fold since the end of the smallpox vaccination campaign in 1980. Outbreaks in nonendemic countries have been related to the exotic pet trade and international travel. Prior to the current global monkeypox outbreak, secondary human-to-human transmission in nonendemic countries was rare, and documented only twice since 2018, both cases involving travelers returning from Nigeria. The first case involved transmission between the index patient and a healthcare

DMID/NIAID/NIH 

<sup>&</sup>lt;sup>5</sup> A pregnancy test will be done at the screening visit (if conducted) and on Day 1 prior to randomization. If there is no screening visit, then pregnancy test done will be done on Day 1 only. Participants of childbearing potential must have negative serum or urine pregnancy test in the 24 hours prior to Day 1 and 29 study vaccinations and results confirmed prior to randomization.

<sup>&</sup>lt;sup>6</sup> Participants reporting monkeypox-like illness and who have a laboratory-confirmed monkeypox will be seen at a sick visit. An unscheduled visit may also occur for reasons including, but not limited to, AE follow up, blood draw, or early termination final visit.

provider<sup>10</sup> and second case involved transmission to another adult and an infant within the household of the index case.<sup>11,12</sup> Monkeypox reemerged in Nigeria in 2017 after more than 40 years with no reported cases.<sup>13,14</sup>

On May 18, 2022, the first U.S. case of monkeypox was detected as part of the larger global 2022 monkeypox outbreak. The U.S. was the fourth non-endemic country to detect a case in a returning traveler. On August 4, the U.S. Department of Health and Human Services declared the U.S. monkeypox outbreak to be a public health emergency with 7,510 confirmed cases of monkeypox detected in all U.S. states, D.C, and Puerto Rico. As of August 15, 2022, there have been 36,589 confirmed monkeypox cases in 92 countries; most cases have been from 85 non-endemic countries including 11,890 confirmed cases in the United States.

Vaccination is being used as a mitigation strategy in the current monkeypox outbreak for those exposed to and those deemed to be at higher risk of being exposed to monkeypox. There is one FDA-approved vaccine for monkeypox: JYNNEOS Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN). A second vaccine, ACAM2000 is likely effective but is not FDA-approved for monkeypox and associated with moderate risk of myocarditis and pericarditis (5.7 cases per 1,000 vaccinated) as well as encephalomyelitis, progressive vaccinia, generalized vaccinia, and ocular complications. ACAM2000 should not be given to people with weakened immune system, eczema, cardiac disease, infants <12 months, or pregnant women. Given these attributes, JYNNEOS is the preferred vaccine during the current outbreak and there is a limited supply of the vaccine globally with production unlikely to keep up with the growing demand as the outbreak continues to spread. Given the limited supply of MVA-BN, dose sparing strategies have been suggested. On August 9, 2022, the U.S. Food and Drug Administration (FDA) issued an Emergency Use Authorization (EUA) for the emergency use of a lower (2 x 10<sup>7</sup>) ID dose of JYNNEOS for individuals 18 years of age and older determined to be at high risk for monkeypox infection.

There are several potential dose sparing strategies we considered. Use of a reduced dose administered SC is unlikely to be of comparable immunogenicity to the licensed SC regimen. There were several Phase 1 and 2 trials that evaluated 2-dose regimens of MVA-BN administered SC four weeks apart (Table 3). Although the 2-dose  $5 \times 10^7$  TCID<sub>50</sub> SC regimen may elicit GMT similar to ACAM2000, the GMT will likely be below that of the licensed 2-dose 1 x  $10^8$  MVA-BN regimen.

**Table 3 Prior Subcutaneous Dosing Trials** 

| Reference | | 1 X10 <sup>7</sup> | 2 X10 <sup>7</sup> | 5 X10 <sup>7</sup> | 1 X10 <sup>8</sup> | Assay |
|---|---|---|---|---|---|---|
| | | TCID <sub>50</sub> | TCID <sub>50</sub> | TCID <sub>50</sub> | TCID <sub>50</sub> | |
| Vollmar et al, | Liquid | 6.4 | | | 29.3 | IHD-J PRNT |
| Vaccine, 2006 15 | formulation | (CI not reported) | | | (CI not reported) | GMT |
| Frey at al. | Lyophilized | | 347.2 | 551.5 | 914.5 | MVA PRNT |
| Vaccine, 2007 | formulation | | (161.9, 744.7) | (321.5, 946.0) | (528.0, 1584) | GMT |
| von Krempelhuber | Lyophilized | | 5.5 | 10.3 | 19.4 | IHD-J PRNT |
| Vaccine, 2010 | formulation | | (3.2, 9.6) | (5.8, 18.4) | (11.1, 34.2) | GMT |

A single 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN dose has also been suggested for dose sparing, but in our assessment of the published literature, it is unlikely to be immunogenically equivalent to the standard licensed 2-dose regimen. The pivotal Phase 3 trial demonstrated that a single dose is likely to provide a significantly lower GMT than the licensed 2-dose MVA-BN regimen, 16.9 [13.7, 20.8] as compared to 153.5 [134.3, 175.6], respectively (Table 4).

DMID/NIAID/NIH 

Table 4 MVA-BN Compared to ACAM2000

| | | | | | | | GMTs ratio<br>MVA/ACAM | |
|---|---|---|---|---|---|---|---|---|
| Visit Week | n | GMT | 95% CI | n | GMT | 95% CI | Ratio | 95% CI |
| Plaque Reduction | on Ne | utralizat | tion Test | | | | | |
| Week 0 | 185 | 1.0 | [1.0, 1.1] | 186 | 1.0 | [1.0, 1.0] | 1.008 | [0.97, 1.05] |
| Week 2 | 184 | 16.2 | [13.0, 20.1] | 184 | 16.2 | [13.1, 20.0] | 0.997 | [0.74, 1.35] |
| Week 4 | 185 | 16.9 | [13.7, 20.8] | 186 | 79.3 | [67.1, 93.8] | 0.213 | [0.16, 0.28] |
| Week 6 | 185 | 153.5 | [134.3, 175.6] | 181 | 64.7 | [54.9, 76.2] | 2.372 | [1.92, 2.93] |

NIAID conducted a Phase 2 trial comparing the standard (now licensed) 2-dose 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN SC regimen (liquid formulation) and a 2-dose 2 x 10<sup>7</sup> TCID<sub>50</sub> MVA-BN ID regimen (liquid formulation) and found peak vaccinia virus, Western reserve strain (VV-WR) GMT of 49.5 (40.0, 61.3) and 59.6 (48.1, 74.0), respectively (Table 5). The 2-dose 2 x 10<sup>7</sup> TCID<sub>50</sub> ID regimen was non-inferior to the 2-dose 1 x 10<sup>8</sup> TCID<sub>50</sub> SC regimen and utilized only one-fifth of the dose. These results are supported by a trial evaluating another MVA vaccine (ACAM3000) which showed ID vaccination at 1x10<sup>7</sup> TCID<sub>50</sub> had similar VV-WR GMT to 1x10<sup>8</sup> TCID<sub>50</sub> administered SC or IM. To 1x10<sup>8</sup> TCID<sub>50</sub> administered SC or IM.

**Table 5 Prior Intradermal Dosing Compared to Subcutaneous** 

| Study Visit Day | Group | | |
|---|---|---|---|
| | Lyophilized SC 1x10 <sup>8</sup><br>(N=145) GMT [95% CI] | Liquid SC 1x10 <sup>8</sup> (N=149)<br>GMT [95% CI] | Liquid ID 2x10 <sup>7</sup> (N=146)<br>GMT [95% CI] |
| Day 0 | 7.5 [,] | 7.7 [7.4, 8.0] | 7.7 [7.4, 7.9] |
| Day 14 | 10.9 [9.9, 12.0] | 10.0 [9.0, 11.1] | 10.3 [9.3, 11.3] |
| Day 28 | 10.8 [9.9, 11.9] | 9.6 [8.7, 10.6] | 10.8 [9.9, 11.9] |
| Day 42 | 77.6 [62.3, 96.7] | 45.2 [36.4, 56.2] | 54.4 [43.7, 67.8] |
| Peak post vaccination 2 | 87.8 [71.2, 108.3] | 49.5 [40.0, 61.3] | 59.6 [48.1, 74.0] |

Even with the EUA for intradermal MVA-BN being available, this trial is designed to evaluate several unique issues:

- As vaccine supply is not anticipated to meet the demand in the next year, this trial will evaluate dose reduction strategies focused on the ID route, that is, confirming the previously studied ID dose and evaluating one tenth dose of MVA-BN (1x10<sup>7</sup>).
- This trial will also assess differences in safety and tolerability of the ID versus the licensed SC regimen as issues of tolerability have been raised by the manufacturer and some in the medical community.

#### 2.3 Risk/Benefit Assessment

#### 2.3.1 Known Potential Risks

DMID/NIAID/NIH 

The potential risks to the participants in the study are those related to venipuncture and reactogenicity as well as possible reactions to the vaccine.

### Venipuncture

Venipuncture may cause transient mild discomfort and/or fainting. Bruising at the site of the venipuncture may occur but can be prevented or lessened by applying pressure for several minutes after the injection. Infection at the site is possible but highly unlikely with the use of aseptic technique.

#### **Adverse Reactions**

MVA-BN administered SC was approved by the FDA as the vaccine JYNNEOS for smallpox and monkeypox on September 24, 2019.<sup>18</sup> At the time of licensure, the clinical development program for JYNNEOS included 22 studies involving 7,093 smallpox vaccine-naïve and 766 smallpox vaccine-experienced participants who received at least 1 dose of JYNNEOS and were monitored for safety for at least 6 months following the first vaccination. There were mostly local and systemic reactogenicity and rare cases of allergy/hypersensitivity observed. Within 8 days of administration of a first or second dose of JYNNEOS, the most common solicited local (injection site) reactions among 2,943 smallpox vaccine-naïve healthy adult participants included pain (84.9%), redness (60.8%), swelling (51.6%), induration (45.4%), and itching (43.1%). The most common solicited systemic adverse reactions were muscle pain (42.8%), headache (34.8%), fatigue (30.4%), nausea (17.3%), and chills (10.4%). In a large clinical trial involving 3,003 participants who received at least one dose of MVA, the majority of solicited local and systemic adverse reactions had a median duration of 1 to 6 days, and there was a similar frequency of reported adverse reactions after the first and second dose of JYNNEOS except for site pain which was more common after the first dose (79.3% versus 69.9%).<sup>19</sup>

An analysis of serious adverse events (SAEs) among the 7,093 smallpox vaccine-naïve and 766 smallpox vaccine-experienced participants who received at least 1 dose of JYNNEOS identified only four SAEs (0.05%) in which a causal relationship could not be ruled out. All were non-fatal SAEs and included Crohn's disease, sarcoidosis, extraocular muscle paresis, and throat tightness (angioedema). The trial that had the related angioedema had three other post-vaccination hypersensitivity reactions which were non-serious and judged to related to the vaccination.

As with all injectable vaccines, there is a risk of an allergic reaction or an anaphylactic event. To mitigate the risk, individuals with known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products will not be eligible to participate in the study. In addition, sites must observe participants for 30 minutes after each vaccination and will have appropriate medical treatment available to manage possible anaphylactic reactions. Participants who have an allergic reaction that is temporally associated with vaccination and that the PI believes to be related, will not receive any more study product. However, the participant will be encouraged not to withdraw from the study so that they may be followed for safety and immunogenicity until the end of the study.

#### **Intradermal Route of Administration**

In a Phase 2 clinical trial that compared the ID and SC administration of the liquid formation of MVA-BN, no participants in the Liquid SC dose group experienced a severe systemic reaction and 20.4% experienced a moderate systemic reaction following the first vaccination, and 1.9% of

DMID/NIAID/NIH 

participants experienced severe systemic reactions and 16.6% experienced moderate systemic reactions following the second vaccination. In the Liquid ID dose group, 3.1% of participants experienced a severe systemic reaction and 24.1% experienced moderate systemic reactions following the first vaccination, and 0.7% experienced a severe systemic reaction and 15.0% experienced moderate systemic reactions following the second vaccination. Fatigue was the most common systemic reaction reported in both groups after both vaccinations, reported by 35.9% in the Liquid SC dose group and 41.4% in the Liquid ID dose group after the first vaccination, and 33.1%, and 29.4% of participants in the Liquid SC, and Liquid ID dose groups, respectively after the second vaccination.

Pain at the injection site occurred in 65.4% and 91.0% of participants in the Liquid ID group and the SC group, respectively. Itchiness was the most prevalent local reaction in the Liquid ID group, reported by 89.0% of participants after either vaccination compared to 48.5% in the Liquid SC group. Vaccine site discoloration (hyperpigmentation) was seen in 122 (63.9%) participants in the Liquid ID group and all but three of these events were graded as mild (Grade 1). In contrast, only seven (4.2%) participants in the Liquid SC group had discoloration at the vaccine site and all but one event was Grade 1. Nodule formation at the vaccine site occurred at a similar frequency of participants in the Liquid ID and Liquid SC group; 35 (18.3%) and 34 (20.4%) participants developed a nodule, respectively.

The original protocol (and report) used a more conservative grading scale for erythema and induration than the FDA's current guidance document, "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials". When NIAID reanalyzed the data using the FDA's current toxicity grading scale, 12% of participants in the ID group and 7.2% in the SC group experienced moderate/severe erythema following the first vaccination, and 59.5% in the ID group and 31.2% in the SC group following the second vaccination. Systemic reactogenicity was similar across the two arms.

#### **Risk During Pregnancy**

There were four developmental toxicity studies that evaluated the effect of JYNNEOS on fetal and postnatal development and found no vaccine-related fetal malformations or adverse effects on postnatal development. JYNNEOS has not been evaluated in preclinical studies for carcinogenicity or mutagenicity.

No safety signals were observed in 29 pregnancies that occurred during the clinical development program of MVA-BN and the rate of spontaneous abortions observed was similar to the published background incidence. However, there is insufficient data to assess the vaccine risk to the pregnant woman and her fetus and because of this, woman who are pregnant will not be eligible to participate in this study and females of reproductive potential will be asked to use effective birth control through Day 57.

#### **Risk to Breast Feeding Infant**

It is not known whether JYNNEOS is excreted in human milk. Data are not available to assess the effects of JYNNEOS in the breastfed infant or on milk production/excretion. For this reason, woman who are breastfeeding will not be eligible to participate in this study.

#### Risk to Children and Adolescents

DMID/NIAID/NIH 

Safety and immunogenicity of JYNNEOS have not been established in individuals less than 18 years of age. For this reason, this study will enroll only adults 18 to 50 years of age.

#### **Risk to Individuals with Chronic Diseases**

JYNNEOS does not replicate in human cell lines and therefore the vaccine can be safely administered to immunocompromised individuals. Safety has been demonstrated in clinical trials and studies involving severely immunocompromised animals<sup>20,21</sup> and humans with HIV infection.<sup>22-24</sup> The safety of JYNNEOS in HIV-infected individuals was evaluated in an open label trial that included 351 HIV-infected smallpox vaccine-naïve participants, 131 HIV-infected participants who previously received smallpox vaccine, 88 non-HIV-infected smallpox vaccine-naïve participants, and 9 non-HIV-infected participants who had previously received a smallpox vaccine.<sup>22</sup> HIV-infected participants had CD4 counts  $\geq$  200 and  $\leq$  750 cells/µL at study entry.

Among smallpox vaccine-naïve participants, solicited local and systemic adverse reactions were reported at similar or lower frequencies in HIV-infected participants than in non-HIV-infected participants. Frequencies of other solicited local and systemic adverse reactions were similar to those reported in other trials.<sup>23,24</sup> In this study, individuals infected with HIV can participate in the study unless they had an AIDS defining illness within the last year or their viral load is not well-controlled with antiretroviral therapy (ART).

Individuals with atopic dermatitis (AD) are not able to receive replicating smallpox vaccines including ACAM2000. However, two clinical trials have shown that they can safely be given JYNNEOS.<sup>25,26</sup> The larger of the two studies was a multicenter, open-label clinical trial that evaluated the safety of JYNNEOS in 350 smallpox vaccine-naïve participants either with active or a history of AD and in 282 participants without AD.<sup>26</sup> The proportion of participants reporting solicited local and systemic adverse reactions was similar between the arms, except for redness (61.2% with AD vs. 49.3% without AD), swelling (52.2% with AD vs. 40.8% without AD), chills (15.9% with AD vs. 7.8% without AD) and headache (47.2% with AD vs. 34.8% without AD). However, most adverse events were mild to moderate in severity. In this study, individuals with AD are eligible to participate.

#### **Cardiac Adverse Events of Special Interest (AESI)**

During the 2002-2004 smallpox vaccination campaign initiated by the US Department of Defense (DoD) and Department of Health and Human Services (DHHS) to protect military personnel and civilian first-responders, there were high rates of pericarditis and myocarditis reported among those vaccinated with Dryvax. Similarly, high rates were detected after receipt of ACAM2000.<sup>27</sup> Because of this, during the clinical development of MVA-BN, participants were monitored for cardiac-related signs or symptoms through at least 6 months after the last vaccination. In 22 studies, cardiac AESIs were reported to occur in 1.3% (95/7,093) of JYNNEOS recipients and in 0.2% (3/1,206) of placebo recipients who were smallpox vaccine naïve. The higher proportion of JYNNEOS recipients who experienced cardiac AESIs was driven by cases of asymptomatic post-vaccination elevation of troponin I, the clinical significance of which is unknown.

Among the cardiac AESIs reported, there were six, non-serious cases (0.08%) deemed causally related to JYNNEOS vaccination including tachycardia, electrocardiogram (ECG) T wave inversion, unspecified ECG abnormality, ECG ST segment elevation, ECG T wave abnormality, and palpitations. These data are consistent with findings from a randomized, double-blind, placebo-

DMID/NIAID/NIH 

controlled Phase 3 trial that evaluated the immunogenicity and safety of three consecutive production lots of MVA-BN. In that trial, eight out of 3,003 (0.3%) participants who received at least one dose of MVA-BN had a cardiac AESI. Of these events, two of the eight were considered possibly related to MVA-BN vaccination; one participant had a right bundle branch block on ECG, and the other participant had clinical symptoms consistent with acute pericarditis but had a negative cardiac work-up. This same participant had positive serology to Coxsackie B virus suggesting that an acute viral infection may have been the cause of their symptoms. Given these data, we will not be monitoring for cardiac AESI during this study.

However, we will be monitoring AE, MAAE, and SAE that will allow us to detect symptomatic cardiac conditions.

#### 2.3.2 Known Potential Benefits

JYNNEOS was licensed in 2019 based on pre-clinical studies and clinical trial data showing that the vaccinia virus-specific (VV-WR) geometric mean titer (GMT) elicited by two doses of JYNNEOS was non-inferior to that elicited by ACAM2000; ACAM2000 was licensed based on non-inferiority to Dryvax. Participation in this study may result in protection against monkeypox during this current outbreak. However, participation may also provide no direct benefit to the participant if they develop antibodies to vaccinia virus and/or monkeypox virus that are not fully protective. Society may benefit from the identification of dose sparing regimens that could be used during the current global vaccine shortage. Additional supportive data on ID dosing may be used to inform the public health response to the current outbreak.

#### 2.3.3 Assessment of Potential Risks and Benefits

JYNNEOS is a licensed product with a good safety profile. This study compares the standard 2-dose licensed SC dosing regimen with two, 2-dose ID regimens that use lower doses of the vaccine. We do not anticipate that the risks of participating in the trial and receiving this licensed vaccine will outweigh the benefits of participation and the value of the information gained from conducting this study. Risk to participants will be minimized by excluding groups of individuals identified to be at greatest risk for adverse reactions following vaccination with JYNNEOS.

DMID/NIAID/NIH 

# 3. OBJECTIVES AND ENDPOINTS

| OBJECTIVES | ENDPOINTS<br>(OUTCOME MEASURES) |
|---|---|
| Primary | |
| To determine if peak (Day 43) humoral immune responses following an ID regimen of 2 x 10 <sup>7</sup> TCID <sub>50</sub> MVA- BN are non-inferior to the licensed regimen of 1 x 10 <sup>8</sup> TCID <sub>50</sub> MVA-BN administered SC | Vaccinia virus specific PRNT GMT at Day 43 |
| To determine if peak (Day 43) humoral immune responses following an ID regimen of 1 x 10 <sup>7</sup> TCID <sub>50</sub> MVA- BN are non-inferior to the licensed regimen of 1 x 10 <sup>8</sup> TCID <sub>50</sub> MVA-BN administered SC | Vaccinia virus specific PRNT GMT at Day 43 |
| Secondary | |
| To determine if individual peak humoral immune responses following each ID regimen are non-inferior to the licensed regimen administered SC | Individual peak GMT through Day 365 |
| To evaluate humoral immune responses of each ID regimen (separately) compared to licensed SC regimen each study day. | Vaccinia virus specific PRNT GMT at Study Day 1, 15, 29, 43, 57, 90, 181, and 365 |
| To evaluate the kinetics of the humoral immune responses of each ID regimen (separately) compared to licensed SC regimen through Day 365 | Vaccinia virus specific PRNT half-life (t ½) |
| To compare relative safety among study arms as assessed by systemic and local reactogenicity for 14 days after each vaccination, unsolicited adverse events for 28 days after each vaccination, and serious adverse events (SAE) and medically attended events (MAAE) from Day 1 through Day 57, and related SAE/MAAEs through Day 181 | Frequency, severity, and relatedness of solicited systemic and local AE for 14 days after each vaccination. Frequency severity, and relatedness of unsolicited AEs in each study arm for 28 days after each vaccination. Frequency and relatedness of MAAE and SAEs in each study arm. Frequency of withdrawals or discontinuation of vaccination in each study arm |
| Exploratory | |
| To evaluate other measures of the humoral immune responses for each regimen | Results from additional immunologic assays for vaccinia and other related viruses. |
| To evaluate humoral immune responses of each ID regimen (separately) compared to licensed dose administered SC to monkeypox virus. | Monkeypox virus specific PRNT GMT at Day 1 and 43. |

### 4. STUDY DESIGN

## 4.1 Overall Design

This study is a Phase 2 randomized, open-label, non-placebo controlled, multi-site clinical trial that will evaluate two ID regimens for MVA-BN vaccine compared to the standard SC regimen in healthy, vaccinia-naïve adults 18 to 50 years of age, inclusive. At least 210 participants will be enrolled and randomized to one of three study arms. The two dose sparing strategies include one-fifth  $(2 \times 10^7)$  and one-tenth  $(1 \times 10^7)$  of the standard dose of MVA-BN administered ID on Day 1 and 29 (Arm 1 and 2, respectively). The comparator arm (Arm 3) will be the 2-dose standard  $(1\times 10^8)$  MVA-BN SC regimen.

The study will enroll a 1:1:1 randomization allocation. Participants will not be stratified by clinical trial site, demographic characteristics or HIV infection status; however, these data will be collected during screening and enrollment. Each participant may be screened either in a separate visit in the 7 days prior to Day 1 or on Day 1. Participants will be followed as outlined in the Schedule of Activities. The last follow-up visit will be at about 1 year after the first vaccination.

## 4.2 Scientific Rationale for Study Design

The rationale for each of the arms in this study is as follows:

- 1. MVA-BN 2 x 10<sup>7</sup> TCID<sub>50</sub> ID (1/5th dose) on Days 1, 29 (Study Arm 1) This regimen matches the prior ID dosing and matches the dose authorized in the EUA. This regimen would allow for 5-fold increase in vaccine supply.
- 2. MVA-BN 1 x 10<sup>7</sup> TCID<sub>50</sub> ID (1/10th dose) on Days 1, 29 (Study Arm 2) This regimen would test a larger dose conservation. This regimen would allow for 10-fold increase in vaccine supply.
- 3. MVA-BN 1 x 10<sup>8</sup> TCID<sub>50</sub> SC on Days 1, 29 (Study Arm 3) This regimen is the licensed dose and route and will be used as a comparator.

## **4.3 Justification for Dose**

This study will use the FDA-approved, licensed dose 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN administered SC on Day 1 and 29 as the comparator for the ID doses of MVA-BN. The ID regimens being evaluated in this study use lower doses of the licensed vaccine, and either match or are one dilution lower than the dose used in the prior ID dosing study (PMID 26143613). Therefore, it is anticipated this range is safe and immunogenic.

## 5. STUDY POPULATION

This study will enroll healthy, non-pregnant, non-breastfeeding adults 18 to 50 years old. Participants with stable medical conditions and well-controlled HIV infection can participate. The study will aim to enroll a population that has demographic features similar to the population being affected with monkeypox, yet also reflects the larger U.S. population to ensure broad applicability of the study findings. To this end, the goal will be to enroll:

DMID/NIAID/NIH 

- at least 30% female participants,
- at least 20% African American/Black participants,
- at least 20% Hispanic participants.

These are enrollment goals and will not be a deviation if these are not ultimately met. Sites will be chosen based on projected ability to enroll the representative study population. Enrollment will be monitored and adjusted at individual sites to pursue these goals while also enrolling this study quickly to inform public health decisions.

Participant Inclusion and Exclusion Criteria must be confirmed by an investigator named on the delegation log. If there is any uncertainty, the PI should make the decision on whether a potential participant is eligible for study enrollment. No exemptions are granted on Inclusion/Exclusion Criteria.

#### 5.1 Inclusion Criteria

To be eligible to participate in this study, an individual must meet all the following criteria:

- 1. Individuals 18 50 years of age inclusive at the time of consent.
- 2. Able to read the written informed consent, states willingness to comply with all study procedures, and is anticipated to be available for all study visits.
- 3. Agreement to adhere to Lifestyle Considerations (defined in section 5.4) during the study.
- 4. Females of reproductive potential who have sexual intercourse with males must agree to use highly effective contraception for at least 1 month prior to signing ICF and through Day 57.

*Note: See MOP for definitions and list of highly effective contraception* 

5. In good general health as evidenced by medical history, physical examination, and clinical judgement of the investigator to be in stable state of health.

Note: Participants with pre-existing stable chronic medical conditions defined as conditions not requiring significant change in therapy or hospitalization for worsening disease in the 4 weeks prior to enrollment can be included at the discretion of the investigator. This includes stable, well-controlled HIV positive individuals.

6. If HIV infected individual, they must be on suppressive ART for at least 6 months, report a CD4 count of greater than 350 cells/μL and no AIDS-defining illness in the last year.

## 5.2 Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Ever received a licensed or an investigational smallpox or monkeypox vaccine.

Note: this includes Dryvax, Acam2000, LC 16 m8, MVA-based vaccine candidate or licensed vaccines, and Jynneos, Imvamune or Imvanex)

DMID/NIAID/NIH 

- 2. Any history of monkeypox, cowpox, or vaccinia infection.
- 3. Close contact of anyone known to have monkeypox in the 3 weeks prior to signing ICF
- 4. Immunocompromised as determined by the investigator
- 5. Recent or current use of any immunosuppressing medications in the 4 weeks prior to signing ICF.

Note: topical, ophthalmic, inhaled, intranasal and intraarticular corticosteroids are acceptable, but receipt of  $\geq$ 20 mg/day of prednisone or equivalent for  $\geq$ 14 consecutive days in the 4 weeks prior to signing ICF is exclusionary.

- 6. Pregnant or breast feeding.
- 7. Received or plans to receive a live vaccine in the 4 weeks prior to signing ICF and 4 weeks after each vaccination
- 8. Received or plans to receive any other vaccine in the 2 weeks prior to signing ICF through Day 43.
- 9. Received experimental therapeutic agent or vaccine in the 3 months prior to signing ICF.
- 10. Has known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products.

Note: this includes individuals with history of severe allergic reaction to gentamicin, ciprofloxacin, chicken or egg protein.

- 11. Has tattoos, scars, or other marks which would, in the opinion of the investigator, interfere with assessment of the vaccination site.
- 12. Has any medical disease or condition that, in the opinion of the participating site PI or appropriate sub-investigator, precludes study participation.

Note: this includes acute, subacute, intermittent, or chronic medical disease or condition that would place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the participant's successful completion of this trial.

#### **5.2.1** Exclusion of Specific Populations

This study will enroll healthy non-pregnant, non-breastfeeding adults 18 to 50 years old. Adults with a history of receiving smallpox vaccine as a child and those born before 1971 will be excluded as they are likely to have received smallpox vaccination during the smallpox eradication campaign. Because the effects on the fetus are not known, pregnant individuals will not be eligible for the trial (see Risk/Benefit Assessment Section). In addition, individuals who are breastfeeding will not be eligible because it is not known if JYNNEOS is excreted in the breastmilk. Adolescents and children will not be included in this trial because there is no safety or efficacy data on the ID route of administration in this population. Should the outcome of this trial be deemed acceptable, additional trials may be initiated, including those in other populations.

# 5.3 Inclusion of Vulnerable Participants

Not Applicable. This study will not enroll vulnerable participants including prisoners, cognitively

DMID/NIAID/NIH 

impaired participants, adolescents, and children.

## 5.4 Lifestyle Considerations

During this study, participants are asked to:

- Follow public health guidance on preventing monkeypox infection and notify the clinical site if exposed to an individual with monkeypox.
- Contact the clinical site immediately if they develop signs and symptoms consistent with monkeypox to schedule a study sick visit.
- Refrain from receiving a live vaccine from enrollment through Day 57.
- Refrain from receiving any other vaccine through Day 43.
- Decline participation in another study evaluating investigational vaccines through Day 181.
- Decline participation in another study evaluating an investigational MVA-based vaccine through end of trial.

Of note, participants may enroll in non-interventional, observational studies (e.g., natural history study of monkeypox). However, concurrent participation in this trial and observational studies can only occur if the recommended blood collection volumes are not exceeded.

#### 5.5 Screen Failures

After the screening evaluations have been completed, the investigator or designee is to review the inclusion/exclusion criteria and determine the participant's eligibility for the study. The following information will be collected on screen failures: demographics (age, screen number, sex, ethnicity, and race) and reason(s) for ineligibility. Participants who are found to be ineligible will be told the reason for ineligibility.

A participant may be re-screened once if a protocol eligibility criterion that is not met at the initial time of screening, will be met by rescreening at a later date (e.g., a vaccine was received within exclusionary window at first screening that would not be in the exclusionary window at a later rescreen).

# 5.6 Strategies for Recruitment and Retention

#### 5.6.1 Recruitment

Potential participants will learn about the study via IRB-approved recruitment strategies, which may include direct mailing, recruitment from an IRB-approved trial registry, and local flyers or advertisements. Recruiting may begin with a brief telephone call between study staff and the potential participant. Information about the study will be presented to potential participants, and questions about their health and ability to comply with the study visit schedule will be asked of potential participants to presumptively determine eligibility. Information about the participant may be recorded from interviews or medical records. Appointments will be made at the research site for potential participants who are interested in the study for further screening procedures and additional protocol-specific information.

DMID/NIAID/NIH 

#### 5.6.2 Retention

Study retention strategies will include education and explanation of the study schedule and procedures during screening and enrollment visits and restriction of enrollment to persons who can attend all study visits. Study participants will be reminded of subsequent visits during each visit, and study staff may contact participants prior to appointments. Study staff will contact participants who miss appointments to encourage them to return for completion of evaluations.

#### **5.6.3** Compensation Plan for Participants

Participants may be compensated for their participation in this trial. Compensation will be in accordance with local institution requirements, and pursuant to IRB approval. Reimbursements will be disbursed at specific timepoints during the study with the amount contingent on completing study procedures.

#### 5.6.4 Costs

There is no cost to participants for the research tests, procedures, and study product while taking part in this trial. Procedures and treatment for clinical care may be billed to the participant, participant's insurance or third party.

## 6. STUDY PRODUCT

## 6.1 Study Product(s) and Administration

## **6.1.1** Study Product Description

JYNNEOS is FDA-approved for adults and licensed as a smallpox and monkeypox vaccine in the United States. The vaccine, when thawed, is a milky, light yellow to pale white colored suspension that is licensed for subcutaneous injection. JYNNEOS is a live vaccine produced from the strain Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN), an attenuated, non-replicating orthopoxvirus. MVA-BN is grown in primary Chicken Embryo Fibroblast (CEF) cells suspended in a serum-free medium containing no material of direct animal origin, harvested from the CEF cells, purified, and concentrated by several Tangential Flow Filtration (TFF) steps including benzonase digestion. Each 0.5 mL dose is formulated to contain 0.5 x  $10^8$  to 3.95 x  $10^8$  infectious units of MVA-BN live virus in 10 mM Tris (tromethamine), 140 mM sodium chloride at pH 7.7. Each 0.5 mL dose may contain residual amounts of host-cell DNA ( $\leq 20$  mcg), protein ( $\leq 500$  mcg), benzonase ( $\leq 0.0025$  mcg), gentamicin ( $\leq 0.163$  mcg), and ciprofloxacin ( $\leq 0.005$  mcg).

#### 6.1.2 Dosing and Administration

In this trial, a licensed vaccine is being evaluated (i.e., JYNNEOS) and there is no placebo arm. Use of the contralateral arm is an option if there is any residual local reaction at Day 29 or if participant requests that this be done.

DMID/NIAID/NIH 

## **Table 6 Study Arms**

| Arm | Dose of JYNNEOS (MVA-BN) | Route of Administration* | Vaccination Day | |
|---|---|---|---|---|
| | | | Day 1 | Day 29 |
| 1 | 2 x 10 <sup>7</sup> TCID <sub>50</sub> , (0.1 mL) | Intradermal | X | X |
| 2 | 1 x 10 <sup>7</sup> TCID <sub>50</sub> , (0.05 mL) | Intradermal | X | X |
| 3 | 1 x 10 <sup>8</sup> TCID <sub>50</sub> , (0.5 mL) | Subcutaneous | X | X |

<sup>\*</sup>Subcutaneous is administered in the deltoid region, intradermal is administered in the volar aspect (inner side) of the forearm.

#### **6.1.3 Dose Escalation**

Not Applicable.

#### **6.1.4 Dose Modifications**

Not Applicable.

## 6.1.5 Criteria for Redosing

If study product administration is unsuccessful, another administration will not be attempted.

## 6.2 Preparation/Handling/Storage/Accountability

## 6.2.1 Acquisition and Accountability

#### **Product: JYNNEOS (MVA-BN vaccine)**

The JYNNEOS (MVA-BN vaccine) will be stored and provided by DMID Repository. Study product will be shipped to the clinical research site upon request and approval from DMID.

#### **Accountability**

The participating site PI is responsible for study product distribution and disposition and has ultimate responsibility for study product accountability. The participating site PI may delegate to the participating site's research pharmacist responsibility for study product accountability. The participating site's research pharmacist will be responsible for maintaining complete records and documentation of study product receipt, accountability, dispensation, storage conditions, and final disposition of the study products.

Time of vaccine administration to the participant will be recorded on the appropriate data collection form (DCF). All study product(s), including the amount of JYNNEOS (MVA-BN vaccine), and whether administered or not, must be documented on the appropriate study product accountability record or dispensing log. The sponsor's monitoring staff will verify the participating site's study product accountability records and dispensing logs per the DMID- approved clinical monitoring plan (CMP).

Once all participant dosing is complete, the pharmacy staff should retain or dispose of used study products and complete study product accountability procedures in accordance with site-specific standard operating procedures (SOPs). This applies to:

DMID/NIAID/NIH 

- used and unused JYNNEOS (MVA-BN vaccine) vials
- JYNNEOS (MVA-BN vaccine) cartons

All used vials and cartons may either be sequestered from the unused supplies and retained until study conclusion or until study product accountability has occurred by the monitor and written notification stating retention is no longer required is received. Used syringes should be discarded per usual procedure.

#### **Destruction**

After the study treatment period has ended or as appropriate over the course of the study after study product accountability has been performed, disposition of unused and used JYNNEOS (MVA-BN vaccine) vials can be destroyed on-site following applicable site procedures. A certificate of destruction or documentation of destruction should be provided to the sponsor and retained in the Pharmacy Binder once completed.

# 6.2.2 Formulation, Appearance, Packaging, and Labeling Product: JYNNEOS (MVA-BN vaccine)

JYNNEOS is supplied in a single-dose vial with turquoise and white label for SC injection. Each 0.5 mL dose is formulated to contain 0.5 x  $10^8$  to 3.95 x  $10^8$  infectious units of MVA-BN live virus in 10 mM Tris (tromethamine), 140 mM sodium chloride at pH 7.7. Each 0.5 mL dose may contain residual amounts of host-cell DNA ( $\leq 20$  mcg), protein ( $\leq 500$  mcg), benzonase ( $\leq 0.0025$  mcg), gentamicin ( $\leq 0.163$  mcg), and ciprofloxacin ( $\leq 0.005$  mcg). JYNNEOS is a sterile vaccine formulated without preservatives. The vial stoppers are not made with natural rubber latex.

## 6.2.3 Product Storage and Stability Product: JYNNEOS (MVA-BN vaccine)

JYNNEOS should be kept frozen at -25°C to -15°C (-13°F to +5°F) and stored in the original package to protect from light. JYNNEOS should not be re-frozen once a vial has been thawed. Once thawed, the vaccine may be kept at +2°C to +8°C (+36°F to +46°F) for 12 hours. The package insert provides additional instructions for the handling and storage of JYNNEOS.

## 6.2.4 Preparation

Each dose (0.5 mL) is supplied in a single-dose vial. Sites should allow the vaccine to thaw and reach room temperature before use (about 15 to 30 minutes). After thawing, the total time stored at +2°C to +8°C (+36°F to +46°F) should not exceed 12 hours. Once the vial is punctured and a dose is withdrawn, if it is not used in its entirety, it should be stored at +2°C to +8°C (+36°F to +46°F) and discarded within 8 hours of the first puncture. If the unpunctured vial is initially shipped/stored at 2-8C then it is stable for up to 8 weeks. Sites should not refreeze the vaccine. JYNNEOS may be kept frozen until the expiration date.

JYNNEOS is a light yellow to pale white colored, milky suspension when thawed. Sites will visually inspect the product for particulate matter and discoloration prior to administration. If either condition is present, the vaccine will not be administered. Study product administrators will gently swirl the vial for at least 30 seconds.

• For the ID injection (Arm 1), 0.1 mL of vaccine will be withdrawn from the vial into a sterile syringe and injected intradermally into the volar aspect (inner side) of the forearm.

DMID/NIAID/NIH 

• For the ID injection (Arm 2), 0.05 mL of vaccine will be withdrawn from the vial into a sterile syringe and injected intradermally into the volar aspect of the forearm.

• For the SC injection (Arm 3), 0.5 mL of vaccine will be withdrawn from the vial into a sterile syringe and injected into the fatty tissue over the deltoid area.

See the protocol-specific MOP for detailed information on the preparation, labeling, storage, and administration for each arm.

## 6.3 Measures to Minimize Bias: Randomization and Blinding

### **6.3.1** Treatment Assignment Procedures

The randomization procedure will be described in the MOP.

#### 6.3.2 Randomization

There will be a 1:1:1 randomization allocation. Randomization will not be stratified. Randomized treatment assignments will be generated by a statistician at The Emmes Company, LLC, the Statistical and Data Coordinating Center (SDCC) for this study. Participants will be registered using a web-based application developed by The Emmes Company, LLC. Upon entry of demographic data and confirmation of eligibility for the trial, the participant will be enrolled and randomized. The randomization procedure will be described in more detail in the MOP.

#### **6.3.3** Blinding and Masking Procedures

This study will not utilize blinding or masking procedures as it is an open-label, non-placebocontrolled trial. Research laboratories will be blinded to participant study arm for the purposes of immunogenicity/efficacy evaluations.

# **6.4** Study Intervention Compliance

Each dose of JYNNEOS will be administered by a member of the clinical research team that is qualified and licensed to administer the study product. Administration and date, time, and location of injection will be recorded on the appropriate eCRF.

# **6.5** Concomitant Therapy

At screening (i.e., the screening visit or Day 1 visit if the screening visit is not conducted), participants will be asked about receipt of immunosuppressive therapy, experimental therapeutic agents and vaccines, other medications, and vaccines. At each subsequent study visit through Day 57, new concomitant medication(s) and changes to existing medications will be recorded as well as receipt of a vaccine. For this study, concomitant medications to be reported in the Case Report Form (CRF) are prescription drugs, over-the-counter medications, and supplements.

Concomitant medications taken and vaccines received in the 4 weeks prior to providing informed

DMID/NIAID/NIH 

consent will be recorded in the CRF. Any drug taken or vaccine received by the participant during the trial should be recorded on the appropriate CRF through Day 57. After Day 57, only concomitant medications that are associated with a related SAE or MAAE through Day 181 and clinically relevant to report will be recorded in the CRF. An exception to this schedule for recording concomitant therapy, is during sick visits for those who have laboratory-confirmed monkeypox (illness). During sick visits, concomitant medications and treatment will be collected.

Medications that might interfere with the evaluation of the immune response to MVA-BN should not be used by the participant during the study-reporting period unless clinically indicated as part of the participant's health care for a condition diagnosed after enrollment. This would include any systemic immunosuppressant medication that may impact the immunogenicity endpoints. In the event medical conditions dictate the use of these medications, participants are encouraged to obtain adequate care, comply with the course of therapy as prescribed by their physician and inform the study Investigator as soon as practical.

#### 6.5.1 Rescue Medicine

Not applicable.

# 7. STUDY INTERVENTION DISCONTINUATION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

# 7.1 Halting Criteria and Discontinuation of Study Intervention

## 7.1.1 Study Halting Criteria

The study will be paused for safety analysis if any of the following events occur:

- 1. One (1) participant experiences a SAE after the administration of the vaccine that is considered related to the vaccine.
- 2. One (1) participant experiences a Grade 4 solicited AE after the administration of the vaccine that is considered related to the vaccine.
- 3. Three (3) or more participants experience a Grade 3 or higher unsolicited AE coded to the same Preferred Term based on the medical dictionary for Regulatory Activities (MedDRA) that are deemed related to the vaccine.

In the event a halting rule is met, an unscheduled safety analysis by the DSMB will be required for approval of further enrollment. Further administration of the vaccine, including a second dose, is suspended for all participants until an assessment by the DSMB takes place.

#### 7.1.1.1 Sentinel Participant Halting Rules

Not Applicable.

#### 7.1.1.2 Cohort Halting Rules

Not Applicable.

DMID/NIAID/NIH 

## 7.1.2 Individual Halting Criteria

If a single participant meets an individual halting criterion, this will not halt the whole study but halts the participant's involvement in terms of the administration of the second dose of the vaccine. However, while the participant is discontinued from receipt of vaccine, they should be encouraged to remain in the study to monitor safety and evaluate immunogenicity until the end of the study.

- 4. Any participant experiences laryngospasm, bronchospasm or anaphylaxis within 24 hours after the administration of the vaccine that is considered related to the vaccine within the 24 hours after vaccination.
- 5. Any participant experiences generalized urticaria (defined as urticarial lesions occurring at more than two body parts) within 3 days after the administration of the vaccine.
- 6. Any participant experiences any Grade 4 solicited AE or an SAE after the administration of the vaccine that is deemed related to the vaccine.
- 7. Any participant that experiences ulceration, abscess or necrosis at the injection site that is considered related to the vaccine administration.

A participant may be removed from the study if the Investigator or the medical monitor deems it in the best interest of the participant. The participant could be withdrawn from the study at any time during the trial.

## 7.1.3 Follow up for participants that discontinued study intervention

Discontinuation from vaccination administration does not mean discontinuation from the study, and remaining study procedures should be completed as indicated by the study protocol. If a clinically significant finding is identified (including, but not limited to changes from baseline) after enrollment, the investigator or qualified designee will determine if any change in participant management is needed.

The second vaccination will not be given, but other follow up visits will continue, if the participant:

- Becomes pregnant.
- Develops monkeypox (symptomatic disease) after the first vaccination
- Meets an exclusion criterion for participation in the study (either newly developed or not previously recognized) that precludes further study participation.

If a participant meets an exclusion criterion after enrollment/randomization and first dose, it does not necessarily mean the participant cannot receive the second dose of JYNNEOS. The decision of what "precludes further study participation" depends on what exclusion criteria are met, with a focus on what is best for participant safety. The most likely exclusion criteria to be met are participants that receive a licensed vaccine after randomization (i.e., exclusion criteria 7 and 8). If a participant receives an off-study vaccine during the study-defined restricted time periods (i.e., as defined in exclusion criteria and Section 5.4), receipt of the off- study vaccine should be reported as a deviation. The participant can receive the second study vaccination if the investigator determines that the participant is otherwise eligible to receive the second MVA-BN in this trial.

There is no reactogenicity threshold for administration of the second dose of vaccine, that is the

DMID/NIAID/NIH 

second dose may be administered even if there is residual erythema, induration or other reactogenicity from the first vaccination. Participants may decline the second vaccination due to residual reactogenicity at the Day 29 visit and will be discontinued from the study intervention. However, the participant will remain in the study and followed for safety and immunogenicity through Day 365 unless they withdraw from the study.

The data to be collected at the time of study intervention discontinuation will include:

- Reason for discontinuation study vaccination including, but not limited to, unacceptable (intolerable) reactogenicity, new medical condition identified that places participant at risk, participant unwillingness to have second vaccination.
- Confirmation of willingness to remain in the study and understanding of study schedule. Participant Withdrawal from the Study and Replacement Participants are free to withdraw from participation in the study at any time upon request. An investigator may withdraw a participant from the study if the participant:
  - Has an AE or other medical condition that continued participation in the study would not be in the best interest of the participant.
  - Is lost to follow-up

The reason for participant discontinuation or withdrawal from the study, whether the decision was made by investigator or participant, and the extent of the withdrawal (i.e., whether participant withdrew from all components of research study or just the study intervention) will be recorded on the CRF. If the participant agrees, every attempt will be made to follow all AEs through resolution (return to baseline) or until defined as stable. The investigator will inform the participant that already collected data will be retained and analyzed for this study even if the participant withdraws from this study. Biospecimens collected will still be used to analyze the study endpoints.

Participants who withdraw, or are withdrawn from this study, or are lost to follow-up after signing the ICF and administration of the study product will not be replaced.

# 7.2 Lost to Follow-Up

A participant will be considered lost to follow-up if he or she fails to return for two scheduled visits and is unable to be contacted by the study site staff after three attempts. Extensive effort (i.e., generally three documented contact attempts via telephone calls, e-mail, etc., made on separate occasions) will be made to locate or recall the participant, or at least to determine the participant's health status. These efforts will be documented in the participant's study file.

## 8. STUDY ASSESSMENTS AND PROCEDURES

# **8.1** Screening Procedures

In this study, screening assessments can occur in an optional screening visit on Day -7 to -1, or at Visit 1 on Day 1 before the first vaccination. At the time of the screening assessment, the participant will be provided with detailed study information and written informed consent will be obtained. The following assessments are performed to determine eligibility requirements as specified in the inclusion and exclusion criteria:

DMID/NIAID/NIH 

- Obtain demographic data.
- Obtain monkeypox exposure history in the 3 weeks prior to signing ICF.
- Review vaccination history, including any experimental vaccines, and determine receipt of exclusionary vaccine(s):
  - o Live vaccine in the prior 4 weeks or an inactivated vaccine in the prior 2 weeks.
  - o Licensed or investigation smallpox or monkeypox vaccine.
- Obtain medical history. Ask specifically about worsening of any chronic medical condition or hospitalizations in the prior 4 weeks, and whether they have the following medical conditions:
  - HIV infection
  - o History of monkeypox, cowpox or vaccinia infection
  - o History of anaphylaxis or severe adverse reaction to a vaccine or vaccine product
  - o History of allergy to gentamicin, ciprofloxacin, chicken or egg protein
  - History of keloid scar formation
- Review medications and therapies up to 4 weeks prior to signing ICF and record on the appropriate CRF and determine receipt of exclusionary medication(s):
  - o Experimental therapeutic agent (or vaccine) in the 3 months prior to consent
  - o Use of immunosuppressing drugs prior to consent.
- Perform targeted physical examination and inspect arms for smallpox vaccination scar
- Measure vital signs (Heart rate (HR), Blood pressure (BP), and oral temperature).
- Review of birth control history with female participants.
  - Counsel participants to use adequate birth control methods required during the trial to avoid pregnancy.
  - o Do serum or urine pregnancy test (in participants of childbearing potential)
- Review inclusion and exclusion criteria.

The overall eligibility of the participant to participate in the study will be assessed once all screening values are available. The screening process can be suspended prior to complete assessment at any time if exclusions are identified by the study team.

Study participants who qualify for inclusion will be enrolled.

# 8.1.1 Procedures to be Followed in the Event of Abnormal Clinical Laboratory Test Values or Abnormal Clinical Findings During Screening

A participant may be re-screened once if a protocol eligibility criterion that is not met at the initial time of screening, will be met by rescreening at a later date. No participant may be screened more than twice due to a screening failure result.

Participants will be provided the results of pregnancy testing and abnormal clinical findings necessitating follow-up at the discretion of the participating site PI or appropriate sub-investigator.

#### 8.1.2 Sick Visit

Participants with signs and symptoms consistent with monkeypox (e.g., vesicular or pustular lesions, fever, chills, lymphadenopathy, malaise, myalgias, headache, or respiratory symptoms) during the study are asked to call the study site. Those who have laboratory-confirmed monkeypox will be evaluated at the clinical site; those who have not been tested will be asked to have a

DMID/NIAID/NIH 
diagnostic test done. During the visit, the participant will be asked about the current illness (e.g., onset date, treatment received) and for information about the diagnostic testing that was done. Participants will have a targeted physical examination done, and a blood sample will be taken. For more information about this visit, see the MOP and the CRF.

# 8.2 Immunogenicity Assessments

# 8.2.1 Immunogenicity/Efficacy Evaluations

Prior comparator studies used the Bavarian Nordic (BN) Vaccina virus Western Reserve strain (VV-WR) plaque reduction neutralizing antibody (PRNT) assay and enzyme-linked immunosorbent assay (ELISA) to evaluate immunogenicity. <sup>16,23,28</sup> In this study, we will use the PRNT as the primary assay to determine immunogenicity and will test a minimum of 4 timepoints (i.e., at least Days 1, 29, 43, 90 from Days 1, 15, 29, 43, 57, 90, 181 and 365).

This study will also measure a monkeypox virus specific PRNT and will test a minimum of 2 timepoints (Days 1 and 43). The monkeypox PRNT assay is not yet developed, and therefore this endpoint is as an exploratory endpoint. Additional timepoints for each will be evaluated as able (given lab throughput and cost).

# **8.2.2** Exploratory Assessments

Additional assessments of humoral immunity including ELISAs may be performed on samples from this trial.

# 8.3 Safety and Other Assessments

Study procedures are specified in the SOA and more detailed information as needed is provided in the MOP. A study clinician, licensed to make medical diagnoses and listed on the Form FDA 1572 as the participating site PI or appropriate sub-investigator, will be responsible for all study- related medical decisions.

- Medical history
  - o A complete medical history will be obtained by interview of participants at screening (i.e., the screening visit or on Day 1 if no screening visit is conducted).
  - o An interim medical history will be obtained by interview of participants at subsequent study visits or ad hoc telephone call with participant. Any changes since the previous clinic visit will be noted. The interim medical history should include an assessment for adverse events and new medical conditions.
- Physical examination
  - A symptom-directed (targeted) physical exam will be performed if indicated by medical history.
- Reactogenicity Assessments
  - Reactogenicity assessments of solicited systemic reactogenicity occurring from the time of each vaccination through 14 days post each vaccination will include fever, chills, nausea, headache, fatigue, change in appetite, myalgia, and arthralgia.
  - O Assessments of solicited local (injection site) reactogenicity occurring from the time of each vaccination through 14 days post each vaccination will include pain

DMID/NIAID/NIH 

Protocol 22-0020
Appendix A
Version 7.0
23 May 2024

- at injection site, erythema/redness, induration/swelling, and pruritis at site.
- Any ongoing events at Day 15 will be followed at subsequent visits in order to note a resolution date. See Memory Aid section below on measurement of ongoing erythema/redness and/or induration/swelling.

## Memory Aid

- All participants will complete a Memory Aid to document local and systemic reactogenicity from time of each vaccination through 14 days post each vaccination (Days 1-15 for the first vaccination and Days 29-43 for the second vaccination).
- Memory Aids will be reviewed with the participants for any solicited reactions, as well as unsolicited AEs and SAEs.
- The vaccination injection site will be examined at all visits until symptoms resolve.
- o For those with no residual systemic or local reactogenicity at the Day 15 or Day 43 visit, no more data is collected by the participant in the Memory Aid.
- For those with ongoing systemic and/or local reactogenicity at Day 15 or Day 43 visit, they will be asked to do the following:
  - Measure erythema/redness and/or induration/swelling and record in the Memory Aid until it has resolved, if applicable.
  - Record end date of all other signs and symptoms
- Nodules and hyperpigmentation are AEs, and not collected in the Memory Aid to avoid double counting these events which tend to develop at end of second week as a post-inflammatory reaction.

# Assessment of tolerability

On Day 15 and Day 43, the participants will be asked several global assessment questions to evaluate how well the vaccine is tolerated.

## Vital signs

o Vital sign measurements will include systolic and diastolic BP, HR, and oral temperature. Vital signs will be measured at timepoints specified in the SOA.

## • Clinical laboratory evaluations

- Serum or urine pregnancy test will be performed locally by the site laboratory at the screening and must be negative within 24 hours prior to each vaccination on Days 1 and 29. This means that if the screening visit is conducted more than 24 hours prior to vaccination, pregnancy test will need to be done on Day 1. Pregnancy tests may be done as needed at interim or unscheduled visits for all women of childbearing potential.
- O Results must be confirmed as negative prior to enrollment on Day 1 and administration of each vaccination.

# 8.3.1 Procedures to be Followed in the Event of Abnormal Clinical Laboratory Test Values or Abnormal Clinical Findings During Conduct of the Trial

In this study, there will be no clinical laboratory screening or safety tests done except for pregnancy testing. Participants will be notified of the results of the pregnancy test.

## 8.4 Adverse Events and Serious Adverse Events

# 8.4.1 Definition of Adverse Events (AE)

DMID/NIAID/NIH 

Adverse event means any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related (21 CFR 312.32 (a)). An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product.

Any medical condition that is present at the time the participant is screened will be considered as baseline and not reported as an AE. However, if the severity (i.e., grade) of any pre-existing medical condition increases, it should be recorded as an AE.

Adverse events can be further divided into solicited adverse events and unsolicited adverse events. Solicited adverse events are those for which the study team will specifically query the participant whether they occurred. Unsolicited adverse events are those events that the participant report occurring without being queried about the specific event.

#### **8.4.1.1** Solicited Adverse Events

Reactogenicity will be especially important to document because of prior studies demonstrating more local (measurement) reactogenicity among participants who received the ID MVA-BN vaccine injection. In this study, we will collect the following solicited adverse events based on prior studies. This includes local (pain at the site of the injection, erythema/redness, induration/swelling, pruritis) and systemic (fever, chills, nausea, headache, fatigue, change in appetite, myalgia [exclusive of the injection site], and arthralgia) reactogenicity. In addition, we expect that some participants will develop skin discoloration and nodules which will be reported as AEs and not collected on the memory aid and followed through to resolution. For this study, we will use the following toxicity grading scale:

"FDA Guidance for Industry, Toxicity Grading Scale for Healthy Adults and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" as a reference.

Of note, pruritis/itching, arthralgia, chills, and change in appetite are not included in the FDA toxicity table. However, the FDA Guidance allows for addition of other signs and symptoms as follows:

| Mild: | No interference with activity |
|-------------------------------|---------------------------------|
| Moderate: | Some interference with activity |
| Severe: | Prevents daily activity |
| Potentially Life Threatening: | ER visit or hospitalization |

## **8.4.1.2** Unsolicited Events

Unsolicited events are all AEs spontaneously reported by the participant and/or in response to an open question from study personnel or revealed by observation, physical examination or other diagnostic procedures.

# **8.4.2** Definition of Serious Adverse Events

An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the

DMID/NIAID/NIH 

investigator or sponsor, it results in any of the following outcomes (21 CFR 312.32 (a)):

- death
- a life-threatening adverse event\*
- inpatient hospitalization or prolongation of existing hospitalization
- a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or
- a congenital anomaly/birth defect.

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, convulsions that do not result in inpatient hospitalization, etc.

\* An adverse event is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient or participant at immediate risk of death. It does not include grade 4 severity unless the adverse event might have caused death.

## 8.4.2.1 Definition of Medically Attended Adverse Events (MAAE)

A medically attended adverse event (MAAE) is an unsolicited AE that results in unscheduled medical attention such as a hospitalization for less than 24 hours, an emergency room visit, or an otherwise unscheduled healthcare visit for any reason. All SAEs and MAAEs will be collected from Day 1 through Day 57, and all SAE/MAAEs related to the vaccine through Day 181.

# 8.4.2.2 Definition of Suspected Unexpected Serious Adverse Reactions (SUSAR)

A SUSAR is a SAE that is considered related to study product and unexpected.

Unexpectedness to study product will be determined by what is listed in the JYNNEOS package insert.

## 8.4.3 Classification of an Adverse Event

The determination of seriousness, severity, and causality will be made by an on-site investigator or other staff as listed on the delegation log.

Any potential grade 3 or 4 AE should be evaluated by someone qualified to provide a medical evaluation of AEs. This includes but is not limited to physicians, physician assistants, and nurse practitioners.

## **8.4.3.1** Severity of Event

All AEs or SAEs will be assessed for severity, according to the toxicity grading scale, FDA Guidance for Industry, Toxicity Grading Scale for Healthy Adults and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. For adverse events (AEs) not included in the

DMID/NIAID/NIH 

protocol-defined grading scale, the following guidelines will be used to describe severity.

<u>Mild (Grade 1)</u>: Events that are usually transient and may require only minimal or no treatment or therapeutic intervention and generally do not interfere with the participant's usual activities of daily living.

<u>Moderate (Grade 2)</u>: Events that are usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant.

<u>Severe (Grade 3)</u>: Events interrupt usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Severe events are usually incapacitating.

<u>Life-threatening (Grade 4)</u>: Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or care provided.

## **8.4.3.2** Relationship to Study Intervention

For each reported adverse event or reaction, the Principal Investigator or designee must assess the relationship of the event to the study product using the following guideline:

<u>Related</u> – The AE is known to occur with the study intervention, there is a reasonable possibility that the study intervention caused the AE, or there is a temporal relationship between the study intervention and event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study intervention and the AE.

<u>Not Related</u> – There is not a reasonable possibility that the administration of the study intervention caused the event, there is no temporal relationship between the study intervention and event onset, or an alternate etiology has been established.

# 8.4.4 Time Period and Frequency for Event Assessment and Follow-Up

For this study:

- Systemic and local solicited adverse events will be collected from Day 1 through Day 15, and Day 29 through Day 43. However, participants with ongoing systemic and/or local reactogenicity at Day 15 or Day 43 visit, will be asked to measure erythema/redness and/or induration/swelling until it has resolved, if applicable, and record end date of all other signs and symptoms.
- Unsolicited adverse events will be collected from Day 1 through Day 29, and Day 29 through Day 57.
- All Serious adverse events (SAEs) and MAAEs will be collected from Day 1 through Day 57, and all SAE/MAAEs related to the vaccine through Day 181.
- All SAEs will be followed through resolution or until the site investigator deems the event to be chronic or the participant is stable.
- AEs will be followed through resolution.

DMID/NIAID/NIH 

Protocol 22-0020
Appendix A
23 May 2024

## 8.4.5 Adverse Event Reporting

# 8.4.5.1 Investigators Reporting of AEs

All clearly related signs, symptoms, and results of diagnostic procedures performed because of an AE should be grouped together and recorded as a single diagnosis or AE term, if available. If the AE is a laboratory abnormality that is part of a clinical condition or syndrome, it should be recorded as the syndrome or diagnosis rather than the individual laboratory abnormality. Each AE will also be described in terms of duration (start and stop date), severity, association with the study product, action(s) taken, and outcome.

AEs characterized as intermittent require documentation of onset and duration of each episode. All AEs will be assessed for severity, relatedness to study vaccine (see Section 8.4.3), and seriousness (see section 8.4.2) by the study PI or sub-investigator.

All AEs will be captured on the appropriate data collection form. Information to be collected for AEs includes event term or description, date of onset, assessment of severity, relationship to study product, and alternate etiology (assessed only by those with the training and authority to make a diagnosis and listed on the Form FDA 1572 as an investigator), date of resolution, seriousness, and outcome. AEs occurring during the trial collection and reporting period will be documented appropriately regardless of relationship.

# 8.4.5.2 Special Reporting of Adverse Events

Not applicable.

## 8.4.6 Serious Adverse Event Reporting

# 8.4.6.1 Investigators Reporting of SAEs

Any AE that meets a protocol-defined serious criterion must be submitted immediately (within 24 hours of site awareness) on an SAE form to the DMID Pharmacovigilance Group, at the following address:

### **DMID Pharmacovigilance Group**

**Clinical Research Operations and Management Support (CROMS)** 

6500 Rock Spring Dr. Suite 650 Bethesda, MD

20817, USA

SAE Hot Line: 1-800-537-9979 (US) or 1-301-897-1709 (outside US)

SAE FAX Number: 1-800-275-7619 (US) or 1-301-897-1710 (outside US)

SAE Email Address: PVG@dmidcroms.com

In addition to the SAE form, select SAE data fields must also be entered into the SDCC system. See the protocol-specific MOP for details regarding this procedure.

Other supporting documentation of the event may be requested by the DMID Pharmacovigilance Group and should be provided as soon as possible. The DMID Medical Monitor will review and assess the SAE for regulatory reporting and potential impact on study participant safety and

DMID/NIAID/NIH 

protocol conduct.

At any time after completion of the study, if the site principal investigator or appropriate sub-investigator becomes aware of an SAE that is suspected to be related to study product, the site principal investigator or appropriate sub-investigator will report the event to the DMID Pharmacovigilance Group.

## 8.4.6.2 Regulatory Reporting of SAEs

Following notification from the site Principal Investigator or appropriate sub-investigator, DMID, as the IND sponsor, will report any SUSAR to the FDA as an IND safety report. DMID will report an AE as a suspected unexpected adverse event only if there is evidence to suggest a causal relationship between the study intervention and the AE.

The Sponsor must ensure the event meets all three of the definitions:

- Suspected adverse reaction.
- Serious.
- Unexpected.

Both serious and unexpectedness are important, but the event will be reported only if there is evidence to suggest a causal relationship between the drug and the adverse event, such as:

- A single occurrence of an event that is uncommon and known to be strongly associated with drug exposure.
- One or more occurrences of an event that is not commonly associated with drug exposure but is otherwise uncommon in the population exposed to the drug.
- On review as an aggregate analysis when the occurrence is higher than the historical control.

DMID will report to the FDA any unexpected fatal or life-threatening suspected adverse reaction as soon as possible, but in no case later than 7 calendar days after the sponsor's initial receipt of the information. If the event is not fatal or life-threatening the IND safety report will be submitted within 15 calendar days after the sponsor determines that the information qualifies for reporting as specified in 21 CFR Part 312.32. Relevant follow up information to an IND safety report will be submitted as soon as the information is available. Upon request from FDA, DMID will submit to the FDA any additional data or information that the agency deems necessary, as soon as possible, but in no case later than 15 calendar days after receiving the request.

DMID will submit an IND safety report to the FDA and will notify all participating site Principal Investigators (i.e., all Principal Investigators to whom the sponsor is providing drug under its IND(s) or under any Principal Investigator's IND(s) of potential serious risks from clinical studies or any other source, as soon as possible. SAEs that are not SUSARs will be reported to the FDA at least annually in a summary format which includes all SAEs.

# **8.4.7** Reporting Events to Participants

Participants have the right to be informed of any new findings of AEs or SAEs that may affect their safety or influence their choice to participate or continue participating in the study.

DMID/NIAID/NIH 

# 8.4.8 Adverse Events of Special Interest (AESI)

There are no pre-specified AESI for this trial.

## 8.4.9 Reporting of Pregnancy

Pregnancy is not an AE. However, any pregnancy that occurs during study participation (through Day 365) should be reported to the sponsor on the appropriate DCF. Pregnancy should be followed for safety and outcome. This follow-up will include pregnancy outcome (termination, pre-term birth, term birth) and newborn outcome (live birth, fetal demise, stillbirth; presence of any congenital anomalies). No in-person visits will be required for pregnancy outcome determination.

# 8.5 Unanticipated Problems

# 8.5.1 Definition of Unanticipated Problems (UP)

The Department of Health and Human Services Office for Human Research Protections (OHRP) considers unanticipated problems (UPs) involving risks to participants or others to include, in general, any incident, experience, or outcome that meets all of the following criteria:

- Unexpected in terms of nature, severity, or frequency given (a) the research procedures that are described in the protocol-related documents, such as the Institutional Review Board (IRB)-approved research protocol and informed consent document; and (b) the characteristics of the participant population being studied; and
- Related or possibly related to participation in the research ("possibly related" means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research); and
- Suggests that the research places participants or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

Incidents arising from noncompliance with study procedures should be reported as protocol deviations (see Section 10.1.10). An incident that qualifies as both a UP and a protocol deviation should be reported as both.

## 8.5.2 Unanticipated Problem Reporting

The investigator will report unanticipated problems (UPs) to the study sponsor, the reviewing IRB and to the SDCC.

The UP report will include the following information:

- Protocol identifying information: protocol title and number, PI's name, and the IRB project number;
- A detailed description of the event, incident, experience, or outcome;
- An explanation of the basis for determining that the event, incident, experience, or outcome represents an UP;
- A description of any changes to the protocol or other corrective actions that have been taken or are proposed in response to the UP.

DMID/NIAID/NIH 

To satisfy the requirement for prompt reporting, UPs will be reported using the following timeline:

- UPs that are serious adverse events (SAEs) will be reported to the IRB and to the SDCC/study sponsor within 24 hours of the investigator becoming aware of the event.
- Any other UP will be reported to the IRB and to the SDCC/study sponsor within a timeline defined according to the relevant policies.
- UPs will be collected through the end of the study.

# **8.5.3** Reporting Unanticipated Problems to Participants

Participants will be informed of any UPs that will potentially influence their participation in this trial.

# 9. STATISTICAL CONSIDERATIONS

# 9.1 Statistical Hypotheses

The primary hypothesis involves a two-step hierarchical process. The study will first test non-inferiority of the  $2 \times 10^7$  ID regimen relative to  $1 \times 10^8$  SC (standard dose regimen). If the  $2 \times 10^7$  ID regimen is non-inferior to the standard dose regimen, hypothesis testing will proceed to test non-inferiority of the  $1 \times 10^7$  ID regimen relative to the standard dose regimen.

## **Primary Hypothesis 1**

• At Day 43 the humoral immune response of the 2 x 10<sup>7</sup> MVA-BN ID regimen will be non-inferior to the standard 1 x 10<sup>8</sup> MVA-BN SC regimen, as assessed by PRNT GMT.

### **Primary Hypothesis 2**

• At Day 43 the humoral immune response of the  $1 \times 10^7$  MVA-BN ID regimen will be non-inferior to standard  $1 \times 10^8$  MVA-BN SC regimen, as assessed by PRNT GMT.

# **Secondary hypotheses**

- At Day 365 the humoral immune response of the 2 x 10<sup>7</sup> MVA-BN ID regimen will be non-inferior to the standard 1 x 10<sup>8</sup> MVA-BN SC regimen, as assessed by PRNT GMT.
- At Day 365 the humoral immune response of the 1 x 10<sup>7</sup> MVA-BN ID regimen will be non-inferior to the standard 1 x 10<sup>8</sup> MVA-BN SC regimen, as assessed by PRNT GMT.
- The humoral immune responses, as assessed by PRNT GMT, for each ID regimen will be similar to the SC regimen at all study days. [Note, this corresponds to two hypotheses, one for each ID study arm.]
- The humoral immune responses, as assessed by vaccinia specific PRNT half-life, for each ID regimen will be similar to the SC regimen. [Note, this corresponds to two hypotheses, one for each ID study arm.]
- The humoral immune responses, as assessed by monkeypox specific PRNT GMT, for each ID regimen will be similar to the SC regimen at Day 1 and 43. [Note, this corresponds to two hypotheses, one for each ID study arm.]

DMID/NIAID/NIH 

# 9.2 Sample Size Determination

Approximately 210 evaluable (mITT) participants (70 per study arm; 140 total for each test of non-inferiority) will provide ample power for both tests of non-inferiority with a type I error rate of 0.05 (Table 7), and assumes, conservatively, that both arms have a standard deviation of 0.6.

A sample size of 140 total for the test of non-inferiority will provide 84% power with the non-inferiority (NI) margin of 0.5 and two-sided type I error rate of 0.05. Power calculations conservatively assume a standard deviation of 0.6 in both arms (Table 8 and Table 9). Data from prior studies by Pittman and Frey suggest that the standard deviation will be lower than 0.6 at later expected peak times, in which case power should be higher for the non-inferiority tests. Note that the power is expected to be lower for the comparison of the 1 x  $10^7$  ID regimen and the standard dose regimen for two reasons: 1) the hypothesis test is conditional on rejecting the null hypothesis comparing the 2 x  $10^7$  ID arm to the standard regimen arm, and 2) the true GMT for the 1 x  $10^7$  ID may be less than the standard SC dose.

In a prior study that compared ID and SC routes of MVA-BN<sup>16</sup>, 10% of the randomized participants did not receive the second vaccination. Therefore, this trial will enroll up to 231 participants (210 x 1.1) to have 210 evaluable participants.

### **Table 7: Power calculations**

Power calculations for a non-inferiority test of means using unequal variances and two-sided type one error rate of 0.05. Non-inferiority margin of 0.5. Assumed standard deviation (on log10 scale) of 0.6.

| | Sample Size | | |
|---|---|---|---|
| NI margin | per arm | Total sample size for NI test | Power |
| $0.5 \\ \text{Log}_{10}(0.5) = -0.301$ | | | |
| $Log_{10}(0.5) = -0.301$ | 60 | 120 | 0.78 |
| 0.5 | 70 | 140 | 0.84 |
| 0.5 | 80 | 160 | 0.88 |
| 0.5 | 85 | 170 | 0.90 |
| 0.5 | 90 | 180 | 0.92 |

**Table 8: Standard deviation estimates** 

Standard deviation estimates computed from Table S4 of Pittman et al, 2019<sup>29</sup>

| | MVA-BN | | | ACAM2000 | | | Ratio of | 95% CI | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Week | N | GMT | 95% CI | SD<br>(for<br>log <sub>10</sub><br>GMT) | N | GMT | 95% CI | SD<br>(for<br>log <sub>10</sub><br>GMT) | GMTs | |
| 2 | 184 | 16.2 | [13.0, 20.1] | 0.65 | 184 | 16.2 | [13.1, 20.0] | 0.63 | 0.997 | [0.738, 1.348] |
| 4 | 185 | 16.9 | [13.7, 20.8] | 0.63 | 186 | 79.3 | [67.1, 93.8] | 0.51 | 0.213 | [0.163, 0.278] |
| 6 | 185 | 153.5 | [134.3, 175.6] | 0.41 | 181 | 64.7 | [54.9, 76.2] | 0.49 | 2.372 | [1.922, 2.928] |
| 8 | 179 | 118.2 | [102.9,135.8] | 0.41 | 183 | 67.1 | [56.9, 79.0] | 0.49 | 1.763 | [1.422, 2.185] |
| Peak | 185 | 153.5 | [134.3, 175.6] | 0.41 | 186 | 79.3 | [67.1, 93.8] | 0.51 | 1.935 | [1.562, 2.397] |

DMID/NIAID/NIH 

Protocol 22-0020
Appendix A
23 May 2024

**Table 9: Standard deviation estimates** 

Standard deviation estimates computed from Frey et al, 2015<sup>16</sup>

| Study Visit Day | Liquid SC 1x10 <sup>8</sup> N=149 | | Liquid ID 2x10 <sup>7</sup> N=146 | |
|---|---|---|---|---|
| | VV-WR GMT [95% CI] | SD | VV-WR GMT [95% CI] | SD |
| Day 14 | 10.0 [9.0, 11.1] | 0.28 | 10.3 [9.3, 11.3] | 0.27 |
| Day 28 | 9.6 [8.7, 10.6] | 0.27 | 10.8 [9.9, 11.9] | 0.23 |
| Day 42 | 45.2 [36.4, 56.2] | 0.59 | 54.4 [43.7, 67.8] | 0.59 |
| Peak post 2 <sup>nd</sup> vaccination | 49.5 [40.0, 61.3] | 0.58 | 59.6 [48.1, 74.0] | 0.59 |

# 9.3 Statistical Analyses

# 9.3.1 General Methodology

Hypothesis testing will be stepwise, starting with the non-inferiority test of the 2 x 10<sup>7</sup> ID regimen relative to standard regimen, with an unequal-variance, two-sample t-test statistic and 95% two-sided confidence intervals. The ID-dose regimen will be considered non-inferior if the lower bound of the confidence interval (original scale) is no less than half that of the standard dose, giving a non-inferiority (NI) margin of 0.5 (NI= -0.301 log10 scale). The selection of this NI margin was based on the pivotal Phase 3 trial by Pittman et al., in 2019 comparing one dose of ACAM2000 and the now licensed 2-dose standard MVA-BN regimen, which provided an estimated relative (peak) immune response of approximately 2-times higher for MVA-BN (Table 8). An NI margin of 0.5 will correspond an immune response of the lower-dose MVA-BN at least as high as what would be expected for ACAM2000.

If the null hypothesis from analysis 1 is rejected in favor of non-inferiority (i.e., the lower limit of the 95% CI of the difference in log of GMTs for 2 x 10<sup>7</sup> TCID<sub>50</sub> MVA-BN ID compared to 1 x 10<sup>8</sup> MVA-BN SC is greater than log(0.5) which is equal to -0.301), testing will proceed with a non- inferiority test of the 1 x 10<sup>7</sup> MVA-BN ID regimen relative to the standard dose regimen, using an unequal variance, two-sample t-test statistic with 95% confidence interval.

# 9.3.2 Timing of Analyses

# 9.3.2.1 Interim Safety Analyses

Given the need for rapid review and dissemination of study data for public health reasons, AEs and SAEs may be reviewed as necessary outside of DSMB reviews. The DSMB may not need to meet (unless halting rules are met), and materials will be provided electronically. Documentation of review and any concerns noted will be solicited electronically.

The DSMB will review separate cumulative AE data reports for all participants within each arm. Given the safety database known for authorized/approved vaccines, there is no routine mandatory review by the DSMB unless halting rules are triggered.

DMID/NIAID/NIH 

# 9.3.2.2 Interim Immunogenicity Analyses

Interim data review of immunogenicity may be performed after all participants have completed Day 181. Analyses will be performed as needed to inform public health decisions. It is recognized that the data may not be frozen, but the risk of introducing bias at that point in the trial is considered small. The analyses will be provided to the study team. There is no blinded data in this trial. However, research laboratories will be blinded to participant study arm for the purposes of immunogenicity/efficacy evaluations.

Data may be disseminated to public health officials and partners as needed and included in publications and presentations to inform the global scientific community.

## 9.3.2.3 Final Analyses

The final efficacy/immunological/safety outcome(s) may be analyzed after all data for the primary and secondary outcome(s) have been collected and locked.

# 9.3.3 Populations for Analyses

There will be three analysis populations in this study. The safety analysis population includes all enrolled participants who received at least one dose of study vaccine. Analyses for the safety population will include safety reported through the end of the study. The modified intent-to-treat (mITT) population includes all participants who received at least one dose of vaccine and contributed both pre- and at least one post-vaccination venous blood sample for immunogenicity testing for which valid results were reported.

In the final analysis, protocol deviations will be reviewed to determine which protocol deviations may affect the analysis. The per protocol (PP) population will then be defined – and this includes all participants in the mITT subset with the following exclusions:

- Data from all available visits for participants found to be ineligible at baseline.
- Data from all visits after the protocol deviations that are considered to affect the science (as determined by the sponsor at an ad hoc meeting).
- Data from any visit that occurs substantially out of window.

For the PP and mITT analyses, participants will be analyzed according to the study product that they received.

## 9.3.4 Baseline Characteristics and Participant Disposition

Summaries of demographic characteristics of the study population including age, sex, ethnicity, and race will be presented by vaccination arm and overall. In addition, this descriptive analysis will be done by reported HIV infection status.

# 9.3.5 Immunogenicity Analyses

Descriptive summaries of immunogenicity data will be presented for the mITT population. If there are protocol deviations which may affect the analysis, a per-protocol (PP) analysis may also be performed.

DMID/NIAID/NIH 

Geometric Mean Titers (GMT) and Geometric Mean Fold Rise (GMFR) from baseline of VV-WR PRNT will be calculated, along with 95% CIs, for all groups, at each timepoint. Summaries will also be displayed graphically. Geometric Mean Titer Ratio, defined as the ratio of each ID arm to the control SC arm, will also be reported at each timepoint, along with 95% CIs. There are no imputations planned for missing data.

A Statistical Analysis Plan (SAP) will be developed and will detail the full planned analysis.

# 9.3.6 Safety Analyses

The safety outcomes for the three study arms will be evaluated including systemic reactogenicity for 14 days after each vaccination, local reactogenicity for 14 days after each vaccination, and unsolicited adverse events for 28 days after each vaccination. All SAEs and MAAE will be evaluated from Day 1 through Day 57 of the trial as compared to licensed dose, and all related SAE/MAAEs will be evaluated through Day 181.

## 9.3.6.1 Reactogenicity

The number, percentage (observed rate) and exact two-sided 95% CI for participants reporting each solicited local (injection site) reaction and solicited systemic reaction following vaccination will be summarized by study arm after first and second vaccination, and overall (i.e., after any vaccination). In addition, the most severe local and systemic reactions recorded during the follow-up period (i.e., maximum severity) for each participant will be determined and summarized by study arm following each vaccination (as well as overall) and the resulting number and percentage of participants will be summarized by severity grade (none, mild,

moderate, severe, life-threatening). Last, the daily severity of local and systemic reactions will be determined for each participant and the proportion of participants having a sign/symptom each day will summarized by grade and presented by study arm following each vaccination. Rates for any severe (Grade 3 or 4) solicited local or systemic reaction following any vaccination will be compared between study arms.

### 9.3.6.2 Other Adverse Events

The number of associated unsolicited AEs, MAAEs and SAEs following vaccine administration is expected to be small. A complete listing of all events will therefore be provided, including the nature of the event, timing relative to vaccination, severity, duration, and the investigator's assessment of the likely relationship to vaccination. For each type of AE, the observed rate and exact two-sided confidence intervals will be computed for each study arm and listed by toxicity grade. AEs will be MedDRA® coded for preferred term and system organ class. Event rates and exact 95% confidence intervals for each study arm and the entire study cohort will be presented, in aggregate and by MedDRA® categories. Related unsolicited AEs, MAAE and SAEs rates will be compared between the study arms.

The number, percentage (observed rate) for participants that withdrew or discontinued their vaccination series due to safety or reactogenicity events will be tabulated. Rates of withdrawal/discontinuation will be compared between study arms using Fisher's exact test.

DMID/NIAID/NIH 

Protocol 22-0020
Appendix A
23 May 2024

Refer to the SAP for additional information.

# 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

# 10.1 Regulatory, Ethical, and Study Oversight Considerations

This study will be conducted in conformity with the principles set forth in The Belmont Report: Ethical Principles and Guidelines for the Protection of Human Participants of Research (US National Commission for the Protection of Human Participants of Biomedical and Behavioral Research; April 18, 1979), and the federal policy for the Protection of Human Participants codified in 45 CFR Part 46, 21 CFR Part 50 (Protection of Human Participants), and the ICH E6(R2).

An OHRP-registered IRB will review and approve this protocol, associated informed consent documents, recruitment materials, and handouts or surveys intended for the participants, prior to the recruitment, screening and enrollment of participants. The IRB review shall be in accordance with 45 CFR 46 and 21 CFR 50, 21 CFR 56 (IRBs), and other federal, state, and local regulations and policies, as applicable.

Each institution engaged in this research will hold a current Federalwide Assurance (FWA) issued by the Office for Human Research Protections (OHRP) for federally funded research. and provide the FWA number to DMID. Each site principal investigator will obtain IRB approval for this protocol and any amendments to be conducted at his/her research site(s).

Any amendments to the protocol or informed consent documents will be approved by the IRB before they are implemented. IRB review and approval will occur at least annually throughout enrollment and follow-up of participants, in accordance with applicable regulations and the requirements of the IRB/IEC. The participating site PI will notify the IRB of deviations from the protocol and reportable SAEs, as applicable to the IRB policy.

DMID must receive the documentation that verifies IRB/IEC approval for this protocol, informed consent documents and associated documents, prior to the recruitment, screening and enrollment of participants, and any IRB approvals for continuing review or amendments as required by DMID.

## 10.1.1 Informed Consent Process

Informed consent is a process that is initiated prior to an individual agreeing to participate in a trial and continuing throughout the individual's trial participation. Before any study procedures are performed, informed consent will be obtained and documented. Participants will receive a concise and focused presentation of key information about the clinical trial, verbally and with a written consent form. The key information about the purpose of the study, the procedures and experimental aspects of the study, study interventions/products, probability for random assignment to treatment groups, risks and discomforts, the expected duration of the participant's participation in the trial, any expected benefits to the participant, and alternative treatments and procedures that may be available to the participant. The explanation will be organized and presented in lay terminology and language that facilitates understanding why one might or might not want to participate.

DMID/NIAID/NIH 

Participants will receive an explanation as to whether any compensation and any medical treatments are available if injury occurs, and, if so, what they consist of, or where further information may be obtained. Participants will be informed of the anticipated financial expenses, if any, to the participant for participating in the trial, as well as any anticipated prorated payments, if any, to the participant for participating in the trial. They will be informed of whom to contact (e.g., the investigator) for answers to any questions relating to the research project.

Information will also include the foreseeable circumstances and/or reasons under which the participant's participation in the trial may be terminated. The participants will be informed that participation is voluntary and that they are free to withdraw from the study for any reason at any time without penalty or loss of benefits to which the participant is otherwise entitled.

Participants will be informed that records identifying the participant will be kept confidential, and, to the extent permitted by the applicable laws and/or regulations, will not be made publicly available and, if the results of the trial are published, the participant's identity will remain confidential. Participants will be informed whether private information collected from this research and/or specimens will be used for additional research, even if identifiers are removed. Participants will be informed that the monitor(s), auditors(s), IRB, NIAID, and regulatory authority(ies) will be granted direct access to the participant's original medical records for verification of clinical trial procedures and/or data without violating the confidentiality of the participant, to the extent permitted by the applicable laws and regulations, and that, by signing a written informed consent form, the participant is authorizing such access.

Participants will be allowed sufficient time to consider participation in this research trial and can discuss this trial with their family, friends or legally authorized representative, or think about it prior to agreeing to participate.

Informed consent forms will be IRB-approved, and participants will be asked to read and review the consent form. Participants must sign the informed consent form prior to starting any study procedures being done specifically for this trial. Once signed, a copy of the informed consent form will be given to the participant(s) for their records.

New information will be communicated by the site principal investigator to participants who consent to participate in this trial in accordance with IRB requirements. The informed consent document will be updated, and participants will be re-consented per IRB requirements, if necessary.

# 10.1.1.1 Requirements for Permission by Parents/Guardians and Assent by Children (in case of a minor)

Not applicable.

### **10.1.1.2** Other Informed Consent Procedures

Participants will be asked for consent to collect blood for the use of residual specimens and samples for secondary research. This extra/residual blood and corresponding serum will be used as back-up specimens for PP defined assays or designated for secondary research use and stored indefinitely at a designated storage facility. Collection of extra/residual samples during the study will help

DMID/NIAID/NIH 

facilitate rapid follow-on analyses, if warranted, to provide more comprehensive scientific insights into the impact (safety and immunological) of the vaccine on the host response to vaccination. To maintain statistical power in follow-on analyses it is important that extra blood collection and secondary research use be included in as many participants as possible, due to the limited sample size per treatment arm. For this reason, if participants choose not to provide permission for extra blood and secondary research use, they will not be eligible for enrollment into the study.

The stored samples will be labeled with barcodes to maintain confidentiality. Research with identifiable samples and data may occur as needed, however, participant confidentiality will be maintained as described for this protocol and with IRB approval. Samples designated for secondary research use may be used for additional immunological assessments that may include but are not limited to antibody epitope mapping, B and T cell repertoire determination, non-traditional immune assay development, determination of innate immune factors and the ability of vaccine-induced antibodies to cross-react to different proteins and virus strains. These blood samples might be used in new or different immunological laboratory tests, to provide information for the development of new vaccines or therapeutics, or for the studies of monkeypox virus or other related viruses. Samples will not be sold for commercial profit.

Although the results of any future research may be patentable or have commercial profit, participants will have no legal or financial interest in any commercial development resulting from any future research. There are no direct benefits to the participant for extra specimens collected or from the secondary research. No results from secondary research will be entered into the participant's medical record. Incidental findings will not be shared with the participant, including medically actionable incidental findings, unless required by law.

Risks are associated with the additional volume of blood collected, such as anemia. Risks for loss of privacy and confidentiality are described below. Participants may withdraw permission to use samples for secondary use at any time. They will need to contact the participating site and the samples will be removed from the study repository after this study is completed and documentation will be completed that outlines the reason for withdrawal of permission for secondary use of samples. Participants who withdraw consent before the last visit will not have the extra blood drawn for secondary use.

Participants will be asked to consent specifically on primary and secondary research samples. The consent process will include an explanation of the potential risks to the individual participants associated with data submitted to an NIH data repository and subsequent sharing. Data that may potentially identify human participants will not be released in unrestricted databases. Participants will be informed that analytical methods are associated with the risk of re-identification, even when specimens are de-identified. The consent will include whether individual participant data will be shared through a NIH controlled access data repository.

# **10.1.2** Study Termination and Closure

Section 7, Study Intervention Discontinuation and Participant Discontinuation/Withdrawal, describes the temporary halting of the study.

This study may be prematurely terminated if there is sufficient reasonable cause, including but not limited to:

• Determination of unexpected, significant, or unacceptable risk to participants

DMID/NIAID/NIH 

- Results of interim efficacy or futility analysis
- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable
- Regulatory authorities' determination
- Sponsor's determination

If the study is prematurely terminated, the Principal Investigator (PI) will promptly inform study participants and the Institutional Review Board (IRB) and regulatory authorities as applicable.

Study participants will be contacted, as applicable, and be informed of changes to study visit schedule. The PI will assure appropriate follow-up for the participants, as necessary. The sponsor will notify regulatory authorities as applicable.

# 10.1.3 Confidentiality and Privacy

Participant confidentiality is strictly held in trust by the participating investigators, their staff, and the sponsor(s) and their agents. This confidentiality is extended to cover clinical information relating to participants, test results of biological samples and genetic tests, and all other information generated during participation in the study. No identifiable information concerning participants in the study will be released to any unauthorized third party. Participant confidentiality will be maintained when study results are published or discussed in conferences.

The study monitor, other authorized representatives of the sponsor, representatives of the Institutional Review Board (IRB), and/or regulatory agencies may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical study site will permit access to such records.

All source records including electronic data will be stored in secured systems in accordance with institutional policies and federal regulations. All study data and research specimens that leave the site (including any electronic transmission of data) will be identified only by a coded number that cannot be linked to a participant.

As this research is funded by the NIH, it is covered by NIH policy which effectively issues the research a Certificate of Confidentiality. By this policy, researchers cannot be forced to disclose or provide, in any Federal, State, or local civil, criminal, administrative, legislative, or other proceeding, the name of such individual or any such information, document, or biospecimen that contains identifiable, sensitive information about the individual and that was created or compiled for purposes of the research, unless such disclosure or use is made with the consent of the individual to whom the information, document, or biospecimen pertains.

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects, like this study, or for information that must be released in order to meet the requirements of the Federal Food and Drug Administration (FDA).

DMID/NIAID/NIH 

Protocol 22-0020
Appendix A
23 May 2024

A Certificate of Confidentiality does not prevent the participant from voluntarily releasing information about themselves or their involvement in this research. If any person or agency obtains a written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

The Certificate of Confidentiality does not prevent the researchers from reporting without the participant's consent, information that would identify the participant as a participant in the research project regarding matters that must be legally reported including child and elder abuse, sexual abuse, or wanting to harm themselves or others.

The release of individual private information or specimens for other research will only occur if consent was obtained from the individual to whom the information, document, or biospecimen pertains, *or* for the purposes of other research that the release is in compliance with applicable Federal regulations governing the protection of human participants in research.

# 10.1.4 Secondary Use of Stored Specimens and Data

## 10.1.4.1 Samples for Secondary Research

Repository Research Sample

To participate in this study, participants will be asked for consent for storage of samples for secondary use. Samples will be stored indefinitely at a DMID-designated storage facility. Each sample will be encoded (labeled) only with a barcode and a unique tracking number to protect participant confidentiality. Secondary research with coded samples and data may occur, however, participant confidentiality will be maintained as described for this protocol. An IRB review of the secondary research using coded specimens is required.

Repository Research Samples, upon written request and approval from DMID and any approvals required by the site, may be shared for secondary research with investigators at the participating site, with researchers at other sites or other institutions, or company-designated research laboratories. The samples will not be sold or used directly for production of any commercial product. DMID will authorize shipment from the repository.

Reports from secondary research will not be kept in the participants' health records or shared with participants, unless required by law. Reports will not be sent to the specimen repository. The participant's decision for secondary research can be changed at any time by notifying the study doctors or nurses in writing. If the participant changes his/her decision, the samples will be destroyed if the samples have not been used for research or released for a specific research project.

## 10.1.4.2 Data Sharing for Secondary Research

Data from this study may be used for secondary research. Individual participant data collected during the trial that are sufficient to reanalyzed primary and secondary endpoints will be made available after deidentification. The Statistical Analysis Plan and Analytic Code will also be made available. This data will be available following publication, with no end date. The data will be made available to researchers who provide a methodologically sound proposal. The data will be available for any purpose outlined in the approved proposal. Proposals should be directed to DMID. To gain

DMID/NIAID/NIH 

access, data requestors will need to sign a data access agreement.

The investigator may request removal of data on individual study participants from NIH data repositories in the event that a research participant withdraws or changes his or her consent. However, data that have been distributed for approved research use cannot be retrieved.

# **10.1.5** Key Roles and Study Governance

This is a multi-site clinical trial and as such, all study team members and roles are listed in the Manual of Procedures (MOP).

# 10.1.6 Safety Oversight

Safety oversight will be conducted by a DSMB that is an independent group of experts that monitors participant safety and advises DMID. The DSMB members will be separate and independent of study personnel participating in this trial and should not have scientific, financial or other conflict of interest related to this trial. The DSMB will consist of members with appropriate expertise to contribute to the interpretation of the data from this trial. The DSMB will operate under the rules of a DMID-approved charter that will be written at the organizational meeting of the DSMB. Procedures for DSMB reviews/meetings will be defined in the charter.

Reports may include enrollment and demographic information and solicited and unsolicited AE/SAEs. The DSMB will review SAEs on a regular basis and ad hoc during this trial. The DMID Medical Monitor will be responsible for reviewing SAEs in real time.

The DSMB will conduct the following reviews:

- Approximately Day 22-29 after study start. Given the planned short enrollment period (3-4 weeks) and second dose of vaccine given on day 29, there is a narrow window for review. As such the review will focus on AEs utilizing real time reports where able.
- Ad hoc meeting:
  - o When trial-level halting criteria are met
  - o At the request of DMID to review a potential safety concern identified in the trial.
- Interim and final data will be shared with the DSMB, but the DSMB does not need to meet to review the final data.

Additional data may be requested by the DSMB. The DSMB may receive data in aggregate and presented by treatment arm. The DSMB may also be provided with expected and observed rates of the expected AEs in an unblinded fashion and may request the treatment assignment be unblinded for an individual participant if required for safety assessment. The DSMB will review grouped and unblinded data in the closed session only. As an outcome of each review/meeting, the DSMB will make a recommendation as to the advisability of proceeding with study interventions (as applicable), and to continue, modify, or terminate this trial.

The DSMB will operate under the rules of a DMID-approved charter that will be written at the organizational meeting of the DSMB. At this time, each data element that the DSMB needs to assess will be clearly defined. Procedures for DSMB reviews/meetings will be defined in the charter. The

DMID/NIAID/NIH 

Protocol 22-0020
Appendix A

23 May 2024

DSMB will review applicable data to include, but not limited to, study progress and participant, clinical, safety and safety related data. Reports may include enrollment and demographic information, medical history, concomitant medications, physical assessments, clinical laboratory values, dosing compliance, and solicited and unsolicited AE/SAEs.

DMID or the DSMB chair may convene the DSMB on an ad hoc basis according to protocol criteria or if there are immediate concerns regarding observations during the course of this trial. The DMID Medical Monitor is empowered to stop enrollment and study product administration if AEs that meet the halting criteria are reported. The DMID Medical Monitor will be responsible for reviewing SAEs in real time. The DSMB will review SAEs on a regular basis and ad hoc during this trial.

# 10.1.7 Clinical Monitoring

Clinical site monitoring is conducted to ensure that the rights and well-being of trial participants are protected, that the reported trial data are accurate, complete, and verifiable. Clinical Monitoring ensures that the conduct of the trial is in compliance with the currently approved protocol/amendment(s), International Council for Harmonisation (ICH), Good Clinical Practice, and with applicable regulatory requirement(s) and sponsor requirements.

Monitoring for this study will be overseen by NIAID/DMID and conducted by NIAID/DMID contractors. Details of clinical site monitoring are documented in a Clinical Monitoring Plan (CMP). The CMP describes in detail who will conduct the monitoring, at what frequency monitoring will be done, at what level of detail monitoring will be performed, and the distribution of monitoring reports. Monitoring visits will include, but are not limited to, review of regulatory files, investigational product administration and accountability records, eCRFs, informed consent forms, medical and laboratory reports, site study storage records, training records, and protocol and GCP compliance. Site monitors will have access to each participating site, study personnel, and all study documentation according to the NIAID or DMID-approved site monitoring plan. Study monitors will meet with site principal investigators (or designee) to discuss any problems and outstanding issues and will document site visit findings and discussions.

## **10.1.8 Quality Assurance and Quality Control**

Quality control (QC) and quality assurance (QA) activities are essential to the safety of participants, and the reliability of study data. Each site participating in the study is responsible for integrating quality control checks throughout the study and implementing a QA Checklist or Clinical Quality Management Plan (CQMP). The site will conduct the following:

- 8. Routine internal QC and QA activities for the purposes of measuring, documenting and reporting study conduct, protocol adherence, human participants' protections, and reliability of the protocol-driven data collected.
- 9. Processes for addressing data quality issues (i.e., collecting, recording), and reporting findings in a timely manner.
- 10. Identify systemic issues (e.g., protocol or human participant protections non-compliance), and implementation and evaluation of Corrective and Preventative Action Plan (CAPA) procedures, if applicable.

DMID/NIAID/NIH 

# 10.1.9 Data Handling and Record Keeping

## 10.1.9.1 Data Collection and Management Responsibilities

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site investigator. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported. All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data.

## 10.1.9.2 Data Coordinating Center / Biostatistician Responsibilities

The data coordinating center for this study will be responsible for data management, quality review, analysis, and reporting of the study data. Adverse events and medical history will be coded according to the MedDRA dictionary. Concomitant medications will be coded according to the WHO Drug dictionary. At the end of the study, a copy of all datasets including annotated case report forms and data dictionary will be provided to DMID.

A separate Study Data Standardization Plan (SDSP) will be developed which describes the technical recommendations for the submission of human study data and related information in a standardized electronic format throughout product development.

# 10.1.9.3 Data Capture Methods

Clinical research data, including, but not limited to, AE/SAEs, concomitant medications, medical history, physical assessments will be abstracted from the source documentation and/or collected on source document worksheet by study personnel then entered into an eCRFs via a 21 CFR Part 11-compliant internet data entry system provided by the study data coordinating center. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate.

The IND Sponsor is responsible for review of data collection tools and processes, and review of data and reports.

Study data will be collected on paper CRFs and then entered into the eCRF or data will be entered directly into the eCRF.

## **10.1.9.4** Study Record Retention

Study related records, including the regulatory file, study product accountability records, consent forms, participant source documents and electronic records should be maintained for a period of 2 years following the date a marketing application is approved for the investigational product for the indication for which it is being investigated; or, if no application is to be filed or if the application is not approved for such indication, until 3 years after the investigation is discontinued and FDA is notified. These documents should be retained for a longer period, however, if required by local policies or regulations. No records will be destroyed without the written consent of DMID. Consent forms with specimen retention linked to identifiable specimens will be maintained for as long as

DMID/NIAID/NIH 

the specimens remain in identifiable format, and a minimum of three years after use of the identifiable specimens in nonexempt human participant research.

## 10.1.9.5 Source Records

Source data are all information, original records of clinical findings, observations, or other activities documented in a clinical trial necessary for the reconstruction and evaluation of the trial. Each participating site will maintain appropriate medical and research records for this trial, in compliance with ICH GCP, regulatory, and institutional requirements. Data recorded in the electronic case report form (eCRF) derived from source documents should be consistent with the data recorded on the source documents. Data entered directly into the eCRFs will be considered the source document. All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data.

Interview of participants is sufficient for obtaining medical history. Solicitation of medical records from the participant's primary care provider is not required.

#### 10.1.10 Protocol Deviations

A protocol deviation is any noncompliance with the clinical trial protocol, any process that is noted in the protocol and refers to details in the MOP, or GCP requirements.

The noncompliance may be either on the part of the participant, the investigator, or the study site staff. Following a deviation(s), corrective actions should be developed by the site and implemented promptly. All individual protocol deviations will be addressed in participant study records.

It is the responsibility of the site principal investigator and personnel to use continuous vigilance to identify and report deviations within five working days of identification of the protocol deviation, or within five working days of the scheduled protocol-required activity. All deviations must be promptly reported to DMID per the protocol deviation reporting procedures. Protocol deviations must be sent to the local IRB/IEC per their guidelines. The site principal investigator and personnel are responsible for knowing and adhering to their IRB requirements.

## 10.1.11 Publication and Data Sharing Policy

# 10.1.11.1 Human Data Sharing Plan

All NIH protocols are required to have a Data Sharing Plan describe provisions for protecting the participants' privacy and the confidentiality of the data. This study will be conducted in accordance with the following publication and data sharing policies and regulations:

National Institutes of Health (NIH) Public Access Policy, which ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive <u>PubMed Central</u> upon acceptance for publication.

As of January 2018, all clinical trials supported by the NIH must be registered on Clinical Trials.gov,

DMID/NIAID/NIH 

no later than 21 days after the enrollment of the first participant. Results of all clinical trials supported by the NIH, generally, need to be submitted no later than 12 months following the primary completion date. As part of the result posting, a copy of this protocol and a copy of the Statistical Analysis Plan will be posted on ClinicalTrials.gov.

## 10.1.11.2 Genomic Data Sharing Plan

Not Applicable.

### **10.1.11.3** Publication

This study will comply with the NIH Public Access Policy, which ensures that the public has access to the published results of NIH funded research. As such, the final peer-reviewed journal manuscripts will be accessible to the public on PubMed Central no later than 12 months after publication.

## 10.1.12 Conflict of Interest Policy

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct of this trial. DMID has established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

## 10.2 Additional Considerations

## 10.2.1 Research Related Injuries

For any potential research related injury, the site principal investigator or designee will assess the participant. The site principal investigator should then determine if an injury occurred as a direct result of the tests or treatments that are done for this trial. As needed, referrals to appropriate health care facilities will be provided to the participant. No financial compensation will be provided by the NIAID, NIH, or the federal government to the participant, for any injury suffered due to participation in this trial.

## **10.2.2 PREP Act**

The study vaccine and the efforts for this clinical trial are covered under the Public Readiness and Emergency Preparedness Act (PREP Act). The PREP Act applies under the terms of the PREP Act declaration in place for smallpox/orthopoxvirus countermeasures for activities conducted pursuant to federal agreements or federal programs (ref: www.federalregister.gov/documents/2015/12/09/2015-31092/smallpox-medical-countermeasures-amendment). JYNNEOS is used under an IND for monkeypox pursuant to a federal agreement/program and is therefore covered under the PREP Act. The PREP Act covers persons

DMID/NIAID/NIH 

(such as manufacturers, distributers, program planners, and other qualified persons who prescribe, administer or dispense study product) are immune from liability from the administration, or use of a covered countermeasure, such as JYNNEOS. The PREP Act provides immunity for covered persons from liability, unless the injury was caused by willful misconduct.

The PREP Act also established the Countermeasures Injury Compensation Program (CICP) to provide compensation for serious injuries or death that occur as the direct result of the administration or use of certain countermeasures. Any requests for compensation must be filed within one year of the administration or use of the covered countermeasure. Requests for Benefits must be made to the Health Resources and Services Administration's (HRSA) Countermeasures Injury Compensation Program (http://www.hrsa.gov/cicp/) by filing a Request for Benefits Form and all required medical records and supporting documentation. Additional information on filing a Request for Benefits is available on the CICP's website at http://www.hrsa.gov/cicp/. Compensation may then be available for reasonable and necessary medical benefits, lost wages and/or death benefits to eligible individuals for certain injuries in accordance with regulations published by the Secretary of HHS (found at 42 CFR part 110).

If an individual suffers a serious physical injury or death from the administration or use of a covered countermeasure in this study, the individual, the individual's legal or personal representative, the administrator/executor of a deceased individual's estate, or certain survivors may request benefits from the CICP. A serious physical injury means an injury that warranted hospitalization (whether or not the person was actually hospitalized) or that led to a significant loss of function or disability. The CICP is the payer of last resort. This means that it only covers expenses or provides benefits that other third-party payers (such as health insurance, the Department of Veterans Affairs, or Workers' Compensation programs) do not have an obligation to pay.

If the Secretary of HHS does not make a final determination on the individual's request within 240 days, or if the individual decides not to accept the compensation, the injured individual or his representative may pursue a tort claim in the US District Court for the District of Columbia, but only if the claim involves willful misconduct and meets the other requirements for suit under the PREP Act. Any award is reduced by any public or private insurance or worker's compensation available to the injured individual. Awards for non-economic damages, such as pain, suffering, physical impairment, mental anguish, and loss of consortium are also limited. If the individual accepts compensation, or if there is no willful misconduct, then the individual does not have a tort claim that can be filed in a US Federal or a State court.

DMID/NIAID/NIH 

# 11. REFERENCES

1. McCollum AM, Damon IK. Human monkeypox. Clin Infect Dis 2014;58(2):260-7. DOI: 10.1093/cid/cit703.

- 2. Grant R, Nguyen LL, Breban R. Modelling human-to-human transmission of monkeypox. Bull World Health Organ 2020;98(9):638-640. DOI: 10.2471/BLT.19.242347.
- 3. Gong Q, Wang C, Chuai X, Chiu S. Monkeypox virus: a re-emergent threat to humans. Virol Sin 2022. DOI: 10.1016/j.virs.2022.07.006.
- 4. Rimoin AW, Mulembakani PM, Johnston SC, et al. Major increase in human monkeypox incidence 30 years after smallpox vaccination campaigns cease in the Democratic Republic of Congo. Proceedings of the National Academy of Sciences of the United States of America 2010;107(37):16262-7. DOI: 10.1073/pnas.1005769107.
- 5. Emergence of monkeypox in West Africa and Central Africa, 1970-2017. Wkly Epidemiol Rec 2018;93(11):125-32. (https://www.ncbi.nlm.nih.gov/pubmed/29546750).
- 6. Centers for Disease C, Prevention. Multistate outbreak of monkeypox--Illinois, Indiana, and Wisconsin, 2003. MMWR Morb Mortal Wkly Rep 2003;52(23):537-40. (https://www.ncbi.nlm.nih.gov/pubmed/12803191).
- 7. Erez N, Achdout H, Milrot E, et al. Diagnosis of Imported Monkeypox, Israel, 2018. Emerging infectious diseases 2019;25(5):980-983. DOI: 10.3201/eid2505.190076.
- 8. Yong SEF, Ng OT, Ho ZJM, et al. Imported Monkeypox, Singapore. Emerging infectious diseases 2020;26(8):1826-1830. DOI: 10.3201/eid2608.191387.
- 9. Rao AK, Schulte J, Chen TH, et al. Monkeypox in a Traveler Returning from Nigeria Dallas, Texas, July 2021. MMWR Morb Mortal Wkly Rep 2022;71(14):509-516. DOI: 10.15585/mmwr.mm7114a1.
- 10. Vaughan A, Aarons E, Astbury J, et al. Human-to-Human Transmission of Monkeypox Virus, United Kingdom, October 2018. Emerging infectious diseases 2020;26(4):782-785. DOI: 10.3201/eid2604.191164.
- 11. Hobson G, Adamson J, Adler H, et al. Family cluster of three cases of monkeypox imported from Nigeria to the United Kingdom, May 2021. Euro Surveill 2021;26(32). DOI: 10.2807/1560-7917.ES.2021.26.32.2100745.
- 12. Mauldin MR, McCollum AM, Nakazawa YJ, et al. Exportation of Monkeypox Virus From the African Continent. The Journal of infectious diseases 2022;225(8):1367-1376. DOI: 10.1093/infdis/jiaa559.
- 13. Yinka-Ogunleye A, Aruna O, Dalhat M, et al. Outbreak of human monkeypox in Nigeria in 2017-18: a clinical and epidemiological report. The Lancet Infectious diseases 2019;19(8):872-879. DOI: 10.1016/S1473-3099(19)30294-4.
- 14. Durski KN, McCollum AM, Nakazawa Y, et al. Emergence of Monkeypox West and Central Africa, 1970-2017. MMWR Morb Mortal Wkly Rep 2018;67(10):306-310. DOI: 10.15585/mmwr.mm6710a5.
- 15. Vollmar J, Arndtz N, Eckl KM, et al. Safety and immunogenicity of IMVAMUNE, a promising candidate as a third generation smallpox vaccine. Vaccine 2006;24(12):2065-70. DOI: 10.1016/j.vaccine.2005.11.022.
- 16. Frey SE, Wald A, Edupuganti S, et al. Comparison of lyophilized versus liquid modified vaccinia Ankara (MVA) formulations and subcutaneous versus intradermal routes of administration in healthy vaccinia-naive subjects. Vaccine 2015;33(39):5225-34. DOI: 10.1016/j.vaccine.2015.06.075.

DMID/NIAID/NIH 

17. Wilck MB, Seaman MS, Baden LR, et al. Safety and immunogenicity of modified vaccinia Ankara (ACAM3000): effect of dose and route of administration. The Journal of infectious diseases 2010;201(9):1361-70. DOI: 10.1086/651561.

- 18. Food and Drug Administration. Summary Basis for Regulatory Action https://www.fda.gov/media/131802/download. (https://www.fda.gov/media/131802/download).
- 19. Overton ET, Lawrence SJ, Wagner E, et al. Immunogenicity and safety of three consecutive production lots of the non replicating smallpox vaccine MVA: A randomised, double blind, placebo controlled phase III trial. PLoS One 2018;13(4):e0195897. DOI: 10.1371/journal.pone.0195897.
- 20. Suter M, Meisinger-Henschel C, Tzatzaris M, et al. Modified vaccinia Ankara strains with identical coding sequences actually represent complex mixtures of viruses that determine the biological properties of each strain. Vaccine 2009;27(52):7442-50. DOI: 10.1016/j.vaccine.2009.05.095.
- 21. Stittelaar KJ, Kuiken T, de Swart RL, et al. Safety of modified vaccinia virus Ankara (MVA) in immune-suppressed macaques. Vaccine 2001;19(27):3700-9. DOI: 10.1016/s0264-410x(01)00075-5.
- 22. Overton ET, Stapleton J, Frank I, et al. Safety and Immunogenicity of Modified Vaccinia Ankara-Bavarian Nordic Smallpox Vaccine in Vaccinia-Naive and Experienced Human Immunodeficiency Virus-Infected Individuals: An Open-Label, Controlled Clinical Phase II Trial. Open Forum Infect Dis 2015;2(2). DOI: 10.1093/ofid/ofv040.
- 23. Greenberg RN, Overton ET, Haas DW, et al. Safety, immunogenicity, and surrogate markers of clinical efficacy for modified vaccinia Ankara as a smallpox vaccine in HIV-infected subjects. The Journal of infectious diseases 2013;207(5):749-58. DOI: 10.1093/infdis/jis753.
- 24. Overton ET, Lawrence SJ, Stapleton JT, et al. A randomized phase II trial to compare safety and immunogenicity of the MVA-BN smallpox vaccine at various doses in adults with a history of AIDS. Vaccine 2020;38(11):2600-2607. DOI: 10.1016/j.vaccine.2020.01.058.
- 25. von Sonnenburg F, Perona P, Darsow U, et al. Safety and immunogenicity of modified vaccinia Ankara as a smallpox vaccine in people with atopic dermatitis. Vaccine 2014;32(43):5696-702. DOI: 10.1016/j.vaccine.2014.08.022.
- Greenberg RN, Hurley MY, Dinh DV, et al. A Multicenter, Open-Label, Controlled Phase II Study to Evaluate Safety and Immunogenicity of MVA Smallpox Vaccine (IMVAMUNE) in 18-40 Year Old Subjects with Diagnosed Atopic Dermatitis. PLoS One 2015;10(10):e0138348. DOI: 10.1371/journal.pone.0138348.
- 27. Cassimatis DC, Atwood JE, Engler RM, Linz PE, Grabenstein JD, Vernalis MN. Smallpox vaccination and myopericarditis: a clinical review. J Am Coll Cardiol 2004;43(9):1503-10. DOI: 10.1016/j.jacc.2003.11.053.
- 28. von Krempelhuber A, Vollmar J, Pokorny R, et al. A randomized, double-blind, dose-finding Phase II study to evaluate immunogenicity and safety of the third generation smallpox vaccine candidate IMVAMUNE. Vaccine 2010;28(5):1209-16. DOI: 10.1016/j.vaccine.2009.11.030.
- 29. Pittman PR, Hahn M, Lee HS, et al. Phase 3 Efficacy Trial of Modified Vaccinia Ankara as a Vaccine against Smallpox. The New England journal of medicine 2019;381(20):1897-1908. DOI: 10.1056/NEJMoa1817307.

DMID/NIAID/NIH 

Protocol 22-0020
Appendix B
23 May 2024

# APPENDIX B – STAGE 2: ADOLESCENT AND ADULT NONINFERIORITY STUDY

# TABLE OF CONTENTS

| APPENDI | X B – Stage 2: Adolescent and Adult Noninferiority Study | 99 |
|-----------|----------------------------------------------------------|-----|
| 1. Introd | duction | 103 |
| 1.1 | Study Rationale | 103 |
| | Background | |
| | Risk/Benefit Assessment | |
| 1.3.1 | | |
| 1.3.2 | | |
| 1.3.3 | | |
| 2. OBJE | ECTIVES AND ENDPOINTS | 108 |
| 3. STUI | DY DESIGN | 109 |
| 3.1 | Overall Design | 109 |
| | Scientific Rationale for Study Design | |
| | Justification for Dose | |
| 4. STUI | DY POPULATION | 111 |
| 4.1 | Inclusion Criteria | 112 |
| | Exclusion Criteria | |
| 4.2.1 | | |
| 4.3 | Inclusion of Vulnerable Participants | |
| 4.4 | Lifestyle Considerations | 114 |
| 4.5 | Screen Failures | 115 |
| 4.6 | Strategies for Recruitment and Retention | 115 |
| 4.6.1 | Recruitment | 115 |
| 4.6.2 | Retention | 115 |
| 4.6.3 | Compensation Plan for Participants | 115 |
| 4.6.4 | Costs | 116 |
| 5. STUI | DY PRODUCT | 116 |
| 5.1 | Study Product(s) and Administration | 116 |
| 5.1.1 | Study Product Description | 116 |
| 5.1.2 | Dosing and Administration | 116 |
| 5.1.3 | | |
| 5.1.4 | $oldsymbol{arepsilon}$ | |
| | Preparation/Handling/Storage/Accountability | |
| 5.2.1 | Acquisition and Accountability | |
| 5.2.2 | | |
| 5.2.3 | | |
| 5.2.4 | 1 | |
| | Measures to Minimize Bias: Randomization and Blinding | |
| 5.3.1 | Treatment Assignment Procedures | 118 |

| 5.3 | .2 Randomization | 118 |
|---|---|---|
| 5.3 | .3 Blinding and Masking Procedures | 118 |
| 5.4 | Study Intervention Compliance | 118 |
| 5.5 | Concomitant Therapy | 118 |
| 6. ST | UDY INTERVENTION DISCONTINUATION AND PARTICIPANT | |
| | VTINUATION/WITHDRAWAL | 119 |
| 6.1 | Holting Criteria and Discontinuation of Study Intervention | 110 |
| 6.1 | Halting Criteria and Discontinuation of Study Intervention | |
| 6.1 | | |
| 6.1 | - Carlotte and the second of t | |
| 6.2 | Participant Withdrawal from the Study and Replacement | |
| 6.3 | Lost to Follow-Up | |
| 7. ST | UDY ASSESSMENTS AND PROCEDURES | |
| 7.1 | Screening Procedures | |
| | .1 Procedures to be Followed in the Event of Abnormal Clinical Laborato lues or Abnormal Clinical Findings During Screening | • |
| 7.2 | Sick Visit | |
| 7.3 | Additional Study Procedures in Stage 2 | |
| 7.3 | | |
| 7.3 | | |
| 7.4 | Immunogenicity Assessments | |
| 7.4 | | |
| 7.4 | | |
| 7.5 | Safety and Other Assessments | 124 |
| 7.5 | | |
| 7.5 | | • |
| | lues or Abnormal Clinical Findings During the Trial | |
| 7.6 | | |
| 7.6 | | |
| | e main section of the protocol for a description of the classification of an AE in | |
| 7.6 | rerity and causality | |
| 7.6 | · | |
| 7.7 | Unanticipated Problems | |
| | • | |
| | ATISTICAL CONSIDERATIONS | |
| 8.1 | Statistical Hypotheses | |
| 8.2 | Sample Size Determination | |
| 8.3 | Statistical Analyses | |
| 8.3 | $\mathcal{E}_{j}$ | |
| 8.3<br>8.3 | | |
| 8.3<br>8.3 | 1 | |
| 8.3 | | |
| 8.3 | | |
| 0.5 | · | |

| 9. | SUPPOF | RTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | 133 |
|---|---|---|---|
| g | 0.1 Res | gulatory, Ethical, and Study Oversight Considerations | 133 |
| | 9.1.1 | Informed Consent Process | |
| | 9.1.2 | Study Termination and Closure | |
| | 9.1.3 | Confidentiality and Privacy | |
| | 9.1.4 | Secondary Use of Stored Specimens and Data | |
| | 9.1.5 | Key Roles and Study Governance | |
| | 9.1.6 | Safety Oversight | |
| | 9.1.7 | Clinical Monitoring. | |
| | 9.1.8 | Quality Assurance and Quality Control | |
| | 9.1.9 | Data Handling and Record Keeping | |
| | 9.1.10 | Protocol Deviations | |
| | 9.1.11 | Publication and Data Sharing Policy | |
| | 9.1.12 | Conflict of Interest Policy | |
| 9 | ).2 Ad | ditional Considerations | |
| | 9.2.1 | Research Related Injuries | |
| | 9.2.2 | PREP Act | |
| 10. | Reference | es | 145 |

# 1. Introduction

# 1.1 Study Rationale

On July 23, 2022, the WHO Director-General declared that the multi-country outbreak of mpox constitutes a Public Health Emergency of International Concern (PHEIC). Since the first case of mpox was detected in the United Kingdom in a returning traveler from Nigeria on May 6, 2022, the outbreak has rapidly spread to 110 countries or locations worldwide, including 103 that are non-endemic, marking the first time mpox has spread widely outside Central and West Africa. By August of 2022, the number of confirmed mpox cases in the U.S. surpassed that of any other country<sup>2,3</sup>. To mitigate the consequences of this outbreak in the U.S., JYNNEOS vaccine is being offered to individuals considered to be at high risk for acquiring the disease. In Stage 1 of this platform study, we evaluated dose sparing strategies in adults because JYNNEOS, the only licensed vaccine for mpox, was in short supply. In Stage 2 of this study, we will evaluate vaccine safety and immunogenicity among adolescents ages 12 to 17 years to extend eligibility to adolescent population, a population that may be at risk if the outbreak persists in 2023.

# 1.2 Background

Mpox is a reemerging infectious disease caused by Monkeypox virus (MPXV), a large double-stranded DNA virus belonging to the genus, *Orthopoxvirus*.<sup>4</sup> MPXV is a zoonotic orthopoxvirus, primarily transmitted to humans via contact with infected animals, and causing disease similar to smallpox, although with substantially lower mortality.<sup>4-6</sup> MPXV is endemic to West and Central Africa, where the incidence of human mpox cases has increased as much as 20-fold since the end of the smallpox vaccination campaign in 1980.<sup>7,8</sup> Outbreaks in non-endemic countries have been related to the exotic pet trade<sup>9</sup> and international travel.<sup>10-12</sup> Prior to the current global mpox outbreak, secondary human-to-human transmission in non-endemic countries was rare, and documented only twice since 2018, both cases involving travelers returning from Nigeria. The first case involved transmission between the index patient and a healthcare provider<sup>13</sup> and second case involved transmission to another adult and an infant within the household of the index case.<sup>14,15</sup> Mpox reemerged in Nigeria in 2017 after more than 40 years with no reported cases.<sup>16,17</sup>

On May 18, 2022, the first U.S. case of mpox was detected as part of the larger global outbreak.<sup>18</sup> The U.S. was the fourth non-endemic country to detect a case in a returning traveler. On August 4, the U.S. Department of Health and Human Services declared the U.S. mpox outbreak to be a public health emergency with 7,510 confirmed cases of mpox detected in all U.S. states, D.C, and Puerto Rico.<sup>19</sup> As of January 11, 2023, there have been 84,648 confirmed mpox cases worldwide including 29,980 confirmed cases and 21 deaths in the United States.<sup>2</sup>

Vaccination is being used as a mitigation strategy in the current mpox outbreak for those exposed to and those deemed to be at higher risk of being exposed to mpox. There is one FDA-approved vaccine for mpox: JYNNEOS Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN). A second vaccine, ACAM2000, is likely effective but is not FDA-approved for mpox and associated with moderate risk of myocarditis and pericarditis (5.7 cases per 1,000 vaccinated) as well as encephalomyelitis, progressive vaccinia, generalized vaccinia, and ocular complications.

DMID/NIAID/NIH 

Protocol 22-0020 Appendix B

23 May 2024

ACAM2000 should not be given to people with a weakened immune system, eczema, cardiac disease, infants <12 months, or pregnant women. Given these attributes, JYNNEOS is the preferred vaccine during the current outbreak however it is only FDA approved for individuals age 18 and older. On August 9, 2022, the U.S. Food and Drug Administration (FDA) issued an Emergency Use Authorization (EUA) for the emergency use of the licensed SC dose for individuals less than 18 years of age determined to be at high risk for mpox for the emergency use of a lower (2 x 10<sup>7</sup> TCID<sub>50</sub>) ID dose of JYNNEOS for individuals 18 years of age and older determined to be at high risk for MPXV infection. In addition, because of limited vaccine supply, the EUA allowed for the use of a lower (2 x 10<sup>7</sup> TCID<sub>50</sub>) ID dose of JYNNEOS for individuals 18 years of age and older determined to be at high risk for mpox.

While JYNNEOS is available under EUA for individuals younger than 18 years of age, an FDA approved mpox vaccine for adolescents is lacking yet remains a public health need. Most reported cases in the global 2022 mpox outbreak have involved men who have sex with men, with a median age of 34 years. Among global cases with age data available, 1.2% are individuals ages 0-17 years;<sup>23</sup> in the United States, from May 17 through September 24, 2022, MPXV infections in persons under 18 years of age accounted for 0.3% of reported cases.<sup>24</sup> Among 55 adolescents ages 13-17 years, 89% were male, and the most common route of exposure was through male-to-male sexual contact (66%). Prior to the global 2022 outbreak, mpox occurred primarily in children and adolescents in endemic countries.<sup>25,26</sup> Increased MPXV transmission within adolescent populations could occur if the outbreak continues, or in future outbreaks, given the mode of transmission through skin and mucosal contact during sexual activity or other activities involving close contact with an infected individual.

## 1.3 Risk/Benefit Assessment

### 1.3.1 Known Potential Risks

The potential risks to the participants in the study are those related to venipuncture and local reactogenicity as well as possible systemic adverse reactions to the vaccine and vaccination procedure.

## Venipuncture

Venipuncture may cause transient mild discomfort and/or fainting. Bruising at the site of the venipuncture may occur but can be prevented or lessened by applying pressure for several minutes after the injection. Infection at the site is possible but highly unlikely with the use of aseptic technique.

#### **Adverse Reactions**

MVA-BN administered SC was approved by the FDA as the vaccine JYNNEOS for smallpox and mpox on September 24, 2019.<sup>27</sup> At the time of licensure, the clinical development program for JYNNEOS included 22 studies involving 7,093 smallpox vaccine-naïve and 766 smallpox vaccine-experienced participants who received at least 1 dose of JYNNEOS and were monitored for safety for at least 6 months following the first vaccination. There were mostly local and systemic reactogenicity and rare cases of allergy/hypersensitivity observed. Within 8 days of administration of a first or second dose of JYNNEOS, the most common solicited local (injection site) reactions among 2,943 smallpox vaccine-naïve healthy adult participants included pain (84.9%), redness

DMID/NIAID/NIH 

(60.8%), swelling (51.6%), induration (45.4%), and itching (43.1%). The most common solicited systemic adverse reactions were muscle pain (42.8%), headache (34.8%), fatigue (30.4%), nausea (17.3%), and chills (10.4%). The majority of these solicited AEs were mild and moderate severity. However, there were severe (Grade3) solicited AEs the most common being pain in 7.4% of participants. In a large clinical trial involving 3,003 participants who received at least one dose of MVA-BN, the majority of solicited local and systemic adverse reactions had a median duration of 1 to 6 days, and there was a similar frequency of reported adverse reactions after the first and second dose of JYNNEOS except for site pain which was more common after the first dose (79.3% versus 69.9%).<sup>28</sup>

An analysis of serious adverse events (SAEs) among 7,093 smallpox vaccine-naïve and 766 smallpox vaccine-experienced participants who received at least 1 dose of JYNNEOS identified only four SAEs (0.05%) in which a causal relationship could not be ruled out. All were non-fatal SAEs and included Crohn's disease, sarcoidosis, extraocular muscle paresis, and throat tightness (angioedema). The trial that had the related angioedema had three other post-vaccination hypersensitivity reactions which were non-serious and judged to be related to the vaccine.

As with all injectable vaccines, there is a risk of an allergic reaction or an anaphylactic event. To mitigate the risk, individuals with known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products will not be eligible to participate in the study. In addition, sites must observe participants for 30 minutes after each vaccination and will have appropriate medical treatment available to manage possible anaphylactic reactions. Participants who have an allergic reaction that is temporally associated with vaccination and that the PI believes to be related, will not receive any more study product. However, the participant will be encouraged not to withdraw from the study so that they may be followed for safety and immunogenicity until the end of the study.

## **Risk During Pregnancy**

There were four developmental toxicity studies that evaluated the effect of JYNNEOS on fetal and postnatal development and found no vaccine-related fetal malformations or adverse effects on postnatal development. JYNNEOS has not been evaluated in preclinical studies for carcinogenicity or mutagenicity.

No safety signals were observed in 29 pregnancies that occurred during the clinical development program of MVA-BN and the rate of spontaneous abortions observed was similar to the published background incidence. However, there is insufficient data to assess the vaccine risk to the pregnant woman and her fetus and because of this, participants who are pregnant will not be eligible to participate in this study and female of reproductive potential who are having sexual intercourse with male partners will be asked to use effective birth control through Day 57.

## **Risk to Breast Feeding Infant**

It is not known whether JYNNEOS is excreted in human milk. Data are not available to assess the effects of JYNNEOS in the breastfed infant or on milk production/excretion. For this reason, woman who are breastfeeding will not be eligible to participate in this study.

DMID/NIAID/NIH 

## Risk to Children and Adolescents

Safety and immunogenicity of JYNNEOS have not been established in individuals less than 18 years of age. In stage 2 of this study, adolescents ages 12 to 17 years will be enrolled. This data will be used to inform a label change for JYNNEOS in the United States to include full licensure for adolescents of the  $1 \times 10^8$  TCID<sub>50</sub> MVA-BN given subcutaneously 4 weeks apart.

An EUA was issued on August 9, 2022, for the use of a 2-dose 1 x 10<sup>8</sup> regimen of JYNNEOS administered subcutaneously for prevention of mpox disease in individuals younger than 18 years of age who were at high risk for MPXV infection.<sup>29</sup> The EUA was based on "safety and effectiveness data from clinical trials in adults and efficacy data from animal challenge studies and historical data with use of live vaccinia virus (smallpox vaccine) in pediatric populations". Per the EUA, the vaccination provider was responsible for mandatory reporting to the Vaccine Adverse Event Reporting System (VAERS) of all serious adverse events (irrespective of attribution to vaccination); cases of cardiac events, including myocarditis and pericarditis; and cases of thromboembolic events and neurovascular events following vaccination with JYNNEOS. The FDA initially required cardiac screening and prospective monitoring for cardiac events in all early clinical trials of MVA-BN vaccine. A review of six Phase 1 trials conducted between 2004 and 2012 found no myo/pericarditis cases that met the CDC case definition and were judged to be related to vaccine in 382 subjects receiving at least one dose of MVA-BN.<sup>30</sup> Moreover, the MVA vector has been studied in multiple adolescent and pediatric populations in other vaccine trials with no serious safety concerns identified.<sup>31-33</sup>

## Risk to Individuals with Chronic Diseases

JYNNEOS does not replicate in human cell lines and therefore the vaccine can be safely administered to immunocompromised individuals. Safety has been demonstrated in clinical trials and studies involving severely immunocompromised animals<sup>34,35</sup> and humans with HIV infection. The safety of JYNNEOS in HIV-infected individuals was evaluated in an open label trial that included 351 HIV-infected smallpox vaccine-naïve participants, 131 HIV-infected participants who previously received smallpox vaccine, 88 non-HIV-infected smallpox vaccine-naïve participants, and 9 non-HIV-infected participants who had previously received a smallpox vaccine. HIV-infected participants had CD4 counts ≥ 200 and ≤ 750 cells/μL at study entry. Among smallpox vaccine-naïve participants, solicited local and systemic adverse reactions were reported at similar or lower frequencies in HIV-infected participants than in non-HIV-infected participants. Frequencies of other solicited local and systemic adverse reactions were similar to those reported in other trials. His study, individuals infected with HIV can participate in the study unless they had an AIDS defining illness within the last year or their viral load is not well-controlled with antiretroviral therapy (ART) (see Section 5.1).

Individuals with atopic dermatitis (AD) are not able to receive replicating smallpox vaccines including ACAM2000. However, two clinical trials have shown that they can safely be given JYNNEOS.<sup>39,40</sup> The larger of the two studies was a multicenter, open-label clinical trial that evaluated the safety of JYNNEOS in 350 smallpox vaccine-naïve participants either with active or a history of AD and in 282 participants without AD.<sup>40</sup> The proportion of participants reporting solicited local and systemic adverse reactions was similar between the arms, except for redness (61.2% with AD vs. 49.3% without AD), swelling (52.2% with AD vs. 40.8% without AD), chills (15.9% with AD vs. 7.8% without AD) and headache (47.2% with AD vs. 34.8% without AD).

DMID/NIAID/NIH 

However, most adverse events were mild to moderate in severity. In this study, individuals with AD are eligible to participate.

# **Cardiac Adverse Events of Special Interest (AESI)**

During the 2002-2004 smallpox vaccination campaign initiated by the US Department of Defense (DoD) and Department of Health and Human Services (DHHS) to protect military personnel and civilian first-responders, there were high rates of pericarditis and myocarditis reported among those vaccinated with Dryvax. Similarly, high rates were detected after receipt of ACAM2000. Because of this, during the clinical development of MVA-BN, participants were monitored for cardiac-related signs or symptoms through at least 6 months after the last vaccination. In 22 studies, cardiac AESIs were reported to occur in 1.3% (95/7,093) of JYNNEOS recipients and in 0.2% (3/1,206) of placebo recipients who were smallpox vaccine naïve. The higher proportion of JYNNEOS recipients who experienced cardiac AESIs was driven by cases of asymptomatic post-vaccination elevation of troponin I, the clinical significance of which is unknown.

Among the cardiac AESIs reported, there were six, non-serious cases (0.08%) deemed causally related to JYNNEOS vaccination including tachycardia, electrocardiogram (ECG) T wave inversion, unspecified ECG abnormality, ECG ST segment elevation, ECG T wave abnormality, and palpitations. These data are consistent with findings from a randomized, double-blind, placebo-controlled Phase 3 trial that evaluated the immunogenicity and safety of three consecutive production lots of MVA-BN. In that trial, eight out of 3,003 (0.3%) participants who received at least one dose of MVA-BN had a cardiac AESI. Of these events, two of the eight were considered possibly related to MVA-BN vaccination; one participant had a right bundle branch block on ECG, and the other participant had clinical symptoms consistent with acute pericarditis but had a negative cardiac work-up. This same participant had positive serology to Coxsackie B virus suggesting that an acute viral infection may have been the cause of their symptoms. Given these data, we are not monitoring for cardiac AESI during Stage 1 of this study which involves adults ages 18 to 50 years, inclusive. However, in Stage 2, which involves adolescent participants, monitoring for protocol specified AESI (see Section 8.6.3.2) will be part of the study as less is known about the product's safety profile in this population. In addition, an exclusion criterion for adolescents and adults with relevant cardiac history that could place them at risk was added in Stage 2. In Stage 1 and Stage 2, the occurrence of AE, MAAE, and SAE will be monitored allowing detection of symptomatic cardiac events as well as cases of thromboembolic events and neurovascular events following vaccination with JYNNEOS.

#### 1.3.2 Known Potential Benefits

JYNNEOS was licensed in 2019 based on pre-clinical studies and clinical trial data showing that the vaccinia virus-specific (VV-WR) geometric mean titer (GMT) elicited by two doses of JYNNEOS was non-inferior to that elicited by ACAM2000; ACAM2000 was licensed based on non-inferiority to Dryvax. Participation in this study may result in protection against mpox during this current outbreak. However, participation may also provide no direct benefit to the participant and/or if they develop an immune response to vaccinia virus the immune response may not be fully protective against mpox. Data from Stage 2 may benefit society by expanding the population for whom JYNNEOS is FDA approved.

DMID/NIAID/NIH 

Protocol 22-0020 Appendix B

23 May 2024

## 1.3.3 Assessment of Potential Risks and Benefits

JYNNEOS is a licensed product with a good safety profile for the adult population. Stage 2 compares the standard 2-dose SC dosing regimen which is licensed for adults and under EUA for adolescents. Because the safety profile of JYNNEOS is largely unknown among adolescents, research in Stage 2 is categorized as greater than minimal risk but presenting the prospect of benefit for individual subjects (45 CFR 46.405). Risk to participants will be minimized by excluding groups of individuals identified to be at greatest risk for serious adverse reactions following vaccination with JYNNEOS.

# 2. OBJECTIVES AND ENDPOINTS

**Table 1 Stage 2 Objectives and Endpoints** 

| ODJECTIVEC | ENDROINTE |
|---|---|
| OBJECTIVES | ENDPOINTS |
| Duimour | (OUTCOME MEASURES) |
| Primary | |
| To determine if peak (Day 43) humoral immune responses in adolescents ages 12 to 17 years are non-inferior to adults after receipt of a 2-dose SC regimen of 1 x 10 <sup>8</sup> TCID <sub>50</sub> MVA-BN. | Vaccinia virus specific PRNT GMT at Day 43 |
| To describe safety of a 2-dose 1 x 10 <sup>8</sup> TCID <sub>50</sub> | Frequency and severity of solicited systemic and |
| MVA-BN regimen administered SC in adolescents ages 12 to 17 years. | local AE for 7 days after each vaccination. Frequency severity, and relatedness of unsolicited AEs for 28 days after each vaccination. Frequency and description of protocol specified AESIs from Day 1 through 210. Frequency and description of related MAAEs from Day 1 through 210. Frequency and relatedness of SAEs for duration of the study. Frequency and description of withdrawals and discontinuations of vaccination. |
| Secondary | |
| To evaluate humoral immune responses at baseline, prior to the second vaccination, and following receipt of the 2-dose SC regimen of 1 x 10 <sup>8</sup> TCID <sub>50</sub> MVA-BN in adolescents compared to adults on each study day. | Vaccinia virus specific PRNT GMT at Study Day 1, 29, 43, 210, and 394 |
| To evaluate the kinetics of the humoral immune responses to the 2-dose SC regimen of 1 x 10 <sup>8</sup> TCID <sub>50</sub> MVA-BN in adolescents and adults through Day 365 after the second dose is administered. | Vaccinia virus specific PRNT half-life (t ½) |

DMID/NIAID/NIH 
| To compare relative safety and reactogenicity between adolescent and adult study arms. | Frequency and severity of solicited systemic and local AE for 7 days after each vaccination. Frequency severity, and relatedness of unsolicited AEs for 28 days after each vaccination. Frequency and description of protocol specified AESIs from Day 1 through 210. Frequency and description of related MAAEs from Day 1 through 210. Frequency and relatedness of SAEs for duration of the study. Frequency of withdrawals or discontinuation of vaccination in each study arm. |
|---|---|
| To evaluate seroconversion between adolescent and adult study arms. | Vaccinia virus specific PRNT GMT at Study Day 29, 43, 210, and 394 |
| Exploratory | |
| To evaluate other measures of the humoral immune responses for each regimen | Results from additional immunologic assays for vaccinia and other related viruses. |
| To evaluate humoral immune responses of the 2-dose SC regimen of 1 x 10 <sup>8</sup> TCID <sub>50</sub> MVA-BN to monkeypox virus in adolescents compared to adults. | Monkeypox virus specific PRNT GMT at Day 1 and 43. |

## 3. STUDY DESIGN

# 3.1 Overall Design

This study is a Phase 2 open-label, non-placebo controlled, multi-site clinical trial that will evaluate the standard SC regimen in adolescents ages 12 through 17 years, inclusive, and compared to the standard SC regimen in adults ages 18 to 50, inclusive. Approximately 135 healthy, vaccinia-naïve adults will be enrolled in a comparator arm (Arm 4) and will be given the standard, licensed regimen of 1x10<sup>8</sup> TCID<sub>50</sub> MVA-BN administered SC on Day 1 and 29. These adults (Arm 4) will be combined with the 76 healthy, vaccinia-naïve adults that received the standard SC regimen in Stage 1 (Arm 3). Together, this will be the comparator group for non-inferiority testing for the primary endpoint. Approximately 315 healthy, vaccinia-naïve adolescents will be enrolled and given 1x10<sup>8</sup> TCID<sub>50</sub> MVA-BN administered SC on Days 1 and 29 (Arm 5). The study will have a set target enrollment of at least 25% adolescents ages 12 to 14 years, inclusive, to ensure that adequate numbers of younger adolescents are enrolled. Participants will be followed as outlined in the Schedule of Activities (Table 2):

DMID/NIAID/NIH 

Protocol 22-0020
Appendix B
23 May 2024

Table 2 Stage 2 Schedule of Activities (SOA)

| Procedures | Optional<br>Screening<br>Visit<br>Day -7 to<br>-1 | Visit 1<br>Enroll<br>Baseline<br>Day 1 | Visit<br>2<br>Day<br>8 +/-<br>1<br>day | Visit<br>3<br>Day<br>29 +/-<br>3<br>days | Visit 4<br>Day<br>36 +/-<br>1 day | Visit 5<br>Day 43<br>+/- 3<br>days | Visit 6<br>Day 57<br>+/- 3<br>days <sup>6</sup> | Visit 7<br>Day 90<br>+/- 5<br>days <sup>6</sup> | Visit 8<br>Day 210<br>+/- 7<br>days | Visit 9<br>Day 394<br>+/- 14<br>days | Sick or<br>Unscheduled<br>Visit <sup>7</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Days post | | | | | 7 +/-1 | 14 +/-3 | 28 +/-3 | 61 +/-5 | 181 +/- | 365 +/- | |
| second<br>vaccination | | | | | days | days | days | days | 7 days | 14 days | |
| Informed consent and assent where appropriate | X | $X^1$ | | | | | | | | | |
| Demographics | X | $\mathbf{X}^1$ | | | | | | | | | |
| Medical history | X | $X^1$ | X | X | X | X | X | X | X | X | X |
| Vaccine administration | | X | | X | | | | | | | |
| Targeted physical exam | X | $\mathbf{X}^{1}$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | X <sup>6</sup> | $X^2$ | $X^2$ | $X^2$ |
| Vital signs | X | $\mathbf{X}^{1}$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | X <sup>6</sup> | $X^2$ | $X^2$ | $X^2$ |
| Concomitant medicine review <sup>3</sup> | X | X | X | X | X | X | X | X | X | X | X |
| SAE <sup>4</sup> | | | | | All SAE, | Day 1 thro | ugh 394 | | | | $X^4$ |
| Protocol<br>specified AESI<br>and related<br>MAAE <sup>4</sup> | | F | Protocol | specified | AESI and | d related MA | AAEs, Day | 1 through 2 | 210 | | X <sup>4</sup> |
| Unsolicited<br>AEs <sup>4</sup> | | | Unsolic | ited AEs | s, Day 1 th | nrough Day | 57 | | | | $X^4$ |
| Solicited (Local<br>and Systemic)<br>AEs | | Day 1 th<br>Day | | | through<br>y 36 | | | | | | X |
| Pregnancy<br>test <sup>5</sup> | X | $\mathbf{X}^1$ | | X | | | | | | | |
| Maximum<br>blood volume<br>per visit (ml) <sup>8</sup> | | 15 | | 15 | | 15 | | | 15 | 15 | |
| Maximum<br>blood volume<br>total (ml) <sup>8</sup> | | 15 | | 30 | | 45 | | | 60 | 75 | |
| Blood<br>collection visits | | X | | X | | X | | | X | X | |

<sup>&</sup>lt;sup>1</sup> If there is no screening visit, these activities should be conducted at the Day 1 visit prior to enrollment.

DMID/NIAID/NIH 

<sup>&</sup>lt;sup>2</sup> A targeted (symptom-driven) physical exam will be done at screening (i.e., screening visit or Day 1), on Days 8, 29, 36, and 43 (at least assessment of vaccination site and presence of skin reactogenicity will be done), and as needed in all other visits if interim change in medical status reported by participant. Vital signs (temperature, blood

pressure and heart rate) will be done on Day 1 and 29 prior to vaccination. However, if there was a separate screening visit and vital signs (temperature, BP, and HR) were done at that visit, only a temperature is needed on Day 1. Vital signs can be done at other visits on an as needed basis.

- <sup>3</sup> For Stage 2, after Day 57, only concomitant medications that are associated with a protocol specified AESI or related MAAE through Day 210, and all SAE through Day 394 and clinically relevant to report, will be recorded in the CRF. In addition, during sick visits concomitant medications will be collected.
- <sup>4</sup> If SAE/MAAE/AESI or unsolicited AE are reported during a sick visit or unscheduled visit and within the reporting window, it will be reported. See more information about collection of AEs in the safety section of the protocol. See section 8.6.3.2 for additional details on AESIs.
- <sup>5</sup> A pregnancy test will be done at the screening visit (if conducted) and on Day 1 prior to enrollment. If there is no screening visit, then pregnancy test done will be done on Day 1 only. Females of reproductive potential must have negative serum or urine pregnancy test in the 24 hours prior to Day 1 and 29 study vaccinations and results confirmed prior to enrollment. Pregnancy testing is required only for adolescents who have reached menarche based on medical history.
- <sup>6</sup> The Day 57 visit may occur via phone call visit if the participant has no skin changes at either injection site documented at the Day 43 visit. All Day 90 visits in Stage 2 will occur via phone call by a delegated study staff member. For both Day 57 and Day 90 visits, the site may opt to have the participant come in for an in-person visit if deemed necessary. In addition, those who qualify for a phone visit at Day 57 and all Day 90 visits may be conducted virtually via video teleconference (e.g., Zoom, FaceTime) if deemed necessary. If an in-person visit is deemed necessary, site may do vital signs and a physical examination on an as needed basis.
- <sup>7</sup> Participants reporting mpox-like illness who have a positive diagnostic test result will be seen at a sick visit. An unscheduled visit may also occur for reasons including, but not limited to AE follow up, blood draw, or early termination final visit.
- <sup>8</sup> Stage 2 participants will have blood drawn on Days 1, 29, 43, 210 and 394. For Stage 2, a minimally acceptable blood volume on Day 1 and on Day 43 is set at 5-mL of whole blood (SST for serum), regardless of age. Should the site not be able to collect that blood before the first vaccination, the participant will not be permitted to continue. Maximum blood draw at the pre-specified visits in Stage 2 is 15 mL

# 3.2 Scientific Rationale for Study Design

The rationale for each of the study arms in Stage 2 are as follows:

1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN SC on Days 1, 29 (Study Arms 4, and 5) – This regimen is the licensed dose and route for adults ages 18 and above. Arms 4 (adult) and 5 (adolescent) will be used to evaluate noninferiority of this regimen among adolescents compared to adults.

#### 3.3 **Justification for Dose**

This study will use the FDA-approved, licensed dose 1 x 10<sup>8</sup> administered SC on Day 1 and 29 in Stage 2 of the study. It is anticipated that the licensed, 2-dose SC regimen will be safe and immunogenic in adolescents.

## 4. STUDY POPULATION

Stage 2 will enroll healthy, non-pregnant, non-breastfeeding, vaccinia-naïve adolescents ages 12 to 17 years, inclusive and a comparator arm of healthy, non-pregnant, non-breastfeeding, vaccinia-naïve adults ages 18 to 50 years, inclusive. Participants with stable medical conditions and well-controlled HIV infection can participate. Stage 2 will aim to enroll a population that is representative of the U.S. population based on the 2020 U.S. Census data to ensure broad applicability of the study findings given the aim of obtaining full licensure of JYNNEOS in adolescents. In addition, the goal is to enroll at least 25% adolescent participants ages 12 to 14 years.

DMID/NIAID/NIH 

Participant Eligibility Criteria must be confirmed by an investigator named on the delegation log. If there is any uncertainty, the PI should make the decision on whether a potential participant is eligible for study enrollment. They may also contact DMID Medical Officers to discuss. No exemptions are granted on Inclusion/Exclusion Criteria.

#### 4.1 Inclusion Criteria

Study inclusion criteria are similar between stages. To be eligible to participate in Stage 2, an individual must meet the following inclusion criteria:

- Adult ages 18 to 50 years inclusive at the time of consent; OR Adolescent ages 12 to 17 years inclusive at the time of consent.
- Adult participant is able to read the written informed consent, states willingness to comply with all study procedures and is anticipated to be available for all study visits; OR

Parent(s)/Legal Authorized Representative (LAR)(s) of the participating adolescent is able to read and provides written informed permission and participating adolescent provides assent as appropriate for age or development and approved by IRB. Adolescent states willingness to comply with all study procedures and is anticipated to be available for all study visits.

Adult participant is able to understand and agrees to adhere to Lifestyle Considerations (section 5.4) during the study; OR

Parent(s)/LAR(s) of the participating adolescent is able to understand and states willingness to comply with Lifestyle Considerations (section 5.4).

4 Females of reproductive potential who have sexual intercourse with male partners must be using highly effective contraception for at least 1 month prior to signing ICF and agrees to use acceptable method of contraception through Day 57.

Note: See MOP for definitions and list of acceptable method of contraception

In good general health as evidenced by medical history, physical examination, and clinical judgement of the investigator to be in stable state of health.

Note: Participants with pre-existing stable chronic medical conditions defined as conditions not requiring significant change in therapy or hospitalization for worsening disease in the 4 weeks prior to enrollment can be included at the discretion of the investigator. This includes stable, well-controlled HIV positive individuals.

6 Individuals with HIV must be on suppressive ART for at least 6 months, report a CD4 count of greater than 350 cells/μL and no AIDS-defining illness in the last year.

#### 4.2 Exclusion Criteria

DMID/NIAID/NIH 

For Stage 2 of the study, an individual who meets any of the following criteria will be excluded from participation in this study. Of note, the only differences between exclusion criteria in Stage 1 and Stage 2 is criterion 8 and the addition of criterion 13:

1. Ever received a licensed or an investigational smallpox or mpox vaccine.

Note: this includes Dryvax, Acam2000, LC 16 m8, MVA-based vaccine candidate or licensed vaccines, and Jynneos, Imvamune or Imvanex)

- 2. Any history of mpox, cowpox, or vaccinia infection.
- 3. Close contact of anyone known to have mpox in the 3 weeks prior to signing ICF
- 4. Immunocompromised as determined by the investigator
- 5. Recent or current use of any immunosuppressing medications in the 4 weeks prior to signing ICF.

Note: topical, ophthalmic, inhaled, intranasal and intraarticular corticosteroids are acceptable, but receipt of  $\geq 20$  mg/day of prednisone or equivalent for  $\geq 14$  consecutive days in the 4 weeks prior to signing ICF is exclusionary.

- 6. Pregnant or breast feeding.
- 7. Received or plans to receive a live vaccine or any COVID-19 vaccine in the 4 weeks before or after each study vaccination.
- 8. Received or plans to receive any other vaccine in the one week before or after each study vaccination.
- 9. Received experimental therapeutic agent or vaccine in the 3 months prior to signing ICF.
- 10. Has known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products.

Note: this includes individuals with history of severe allergic reaction to gentamicin, ciprofloxacin, chicken or egg protein.

- 11. Has tattoos, scars, or other marks which would, in the opinion of the investigator, interfere with assessment of the vaccination site.
- 12. Has any medical disease or condition that, in the opinion of the participating site PI or appropriate sub-investigator, precludes study participation.

Note: this includes acute, subacute, intermittent, or chronic medical disease or condition that would place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the participant's successful completion of this trial.

- 13. Adolescent or adult participant has a history of myocarditis/pericarditis or a history of structural congenital heart defect/cardiac dysrhythmia that, in the opinion of the investigator, poses increased risk to the participant.
- 14. Adolescent or adult participant has a history of COVID-19 (with positive test for SARS-CoV-2) in the 4 weeks prior to receipt of the first study vaccination.

Note: This includes positive rapid antigen test, polymerase chain reaction (PCR) assay, or other nucleic acid amplification (NAAT) test including those performed by the participant at home.

DMID/NIAID/NIH 

## **4.2.1** Exclusion of Specific Populations

As in Stage 1, Stage 2 of this study will enroll healthy non-pregnant, non-breastfeeding adults ages 18 to 50 years, inclusive. Adults with a history of receiving smallpox vaccine as a child and those born before 1971 will be excluded as they are likely to have received smallpox vaccination during the smallpox eradication campaign. Because the effects on the fetus are not known, pregnant individuals will not be eligible for the trial (see Risk/Benefit Assessment Section). In addition, individuals who are breastfeeding will not be eligible because it is not known if JYNNEOS is excreted in the breastmilk. Stage 2 of the study will also enroll healthy non-pregnant, non-breastfeeding adolescents ages 12 to 17 years, inclusive. Should the outcome of this trial be deemed acceptable, additional trials may be initiated, including those in other populations.

Given that safety of MVA-BN among adolescents ages 12 to 17 years is largely unknown and myocarditis and pericarditis were found to be associated with vaccination with ACAM2000 and Dryvax, replicating smallpox vaccines, adolescents with a history of myocarditis/pericarditis or a history of structural congenital heart defect/cardiac dysrhythmia that, in the opinion of the investigator, poses increased risk to the participant will not be eligible to participate.

# 4.3 Inclusion of Vulnerable Participants

This study will enroll vulnerable participants in Stage 2, including adolescents ages 12 to 17 years. This research can be categorized as greater than minimal risk but presenting the prospect of direct benefit to the participant (45 CFR 46.405) given that MPXV continues to cause disease in the U.S., and may spread into additional populations, including sexually active adolescents. Adolescents will be recruited from communities that represent the general population that attend the clinics associated with the institution for research sites, or individuals who respond to advertisements posted publicly.

# 4.4 Lifestyle Considerations

During Stage 2 of this study, participants are asked to:

- Follow public health guidance on preventing mpox infection and notify the clinical site if exposed to an individual with mpox.
- Contact the clinical site immediately if they develop signs and symptoms consistent with mpox and a positive MPXV diagnostic test to schedule a study sick visit. See Section 8.2 and the MOP.
- Contact the clinical site if they develop COVID-19 illness (with positive test for SARS-CoV-2 including those performed at home by the participant) during the study.
- Refrain from receiving a live vaccine or COVID-19 vaccine in the 4 weeks before or after each study vaccination.
- Refrain from receiving any other vaccine in the one week before or after each study vaccination.
- Decline participation in another study evaluating investigational vaccines through Day 210 in Stage 2.

DMID/NIAID/NIH 

• Decline participation in another study evaluating an investigational mpox vaccine, smallpox vaccine, or MVA-based vaccine through end of trial.

Of note, participants may enroll in non-interventional, observational studies (e.g., natural history study of mpox). However, concurrent participation in this trial and observational studies can only occur if the recommended blood collection volumes as specified by site Institutional Review Board guidance are not exceeded.<sup>42</sup>

#### 4.5 Screen Failures

After the screening evaluations have been completed, the investigator or designee is to review the inclusion/exclusion criteria and determine the participant's eligibility for the study. The following information will be collected on screen failures: demographics (age, screen number, sex, ethnicity, and race) and reason(s) for ineligibility. Participants who are found to be ineligible will be told the reason for ineligibility.

A participant may be re-screened once if a protocol eligibility criterion that is not met at the initial time of screening, will be met by rescreening at a later date (e.g., a vaccine was received within exclusionary window at first screening that would not be in the exclusionary window at a later rescreen).

# 4.6 Strategies for Recruitment and Retention

#### 4.6.1 Recruitment

Potential participants will learn about the study via IRB-approved recruitment strategies, which may include direct mailing, recruitment from an IRB-approved trial registry, and local flyers or advertisements. Recruiting may begin with a brief telephone call between study staff and the potential participant. Information about the study will be presented to potential participants, and questions about their health and ability to comply with the study visit schedule will be asked of potential participants to presumptively determine eligibility. Information about the participant may be recorded from interviews or medical records. Appointments will be made at the research site for potential participants who are interested in the study for further screening procedures and additional protocol-specific information.

#### 4.6.2 Retention

Study retention strategies will include education and explanation of the study schedule and procedures during screening and enrollment visits and restriction of enrollment to persons who can attend all study visits. Study participants will be reminded of subsequent visits during each visit, and study staff may contact participants prior to appointments. Study staff will contact participants who miss appointments to encourage them to return for completion of evaluations.

#### 4.6.3 Compensation Plan for Participants

Participants may be compensated for their participation in this trial. Compensation will be in accordance with local institution requirements, and pursuant to IRB approval. Reimbursements

DMID/NIAID/NIH 

will be disbursed at specific timepoints during the study with the amount contingent on completing study procedures.

#### 4.6.4 Costs

There is no cost to participants for the research tests, procedures, and study product while taking part in this trial. Procedures and treatment for clinical care may be billed to the participant, participant's insurance or third party.

# 5. STUDY PRODUCT

# 5.1 Study Product(s) and Administration

## 5.1.1 Study Product Description

JYNNEOS is FDA-approved and licensed for adults as a smallpox and mpox vaccine in the United States. The vaccine, when thawed, is a milky, light yellow to pale white colored suspension that is licensed for subcutaneous injection. JYNNEOS is a live vaccine produced from the strain Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN), an attenuated, non-replicating orthopoxvirus. MVA-BN is grown in primary Chicken Embryo Fibroblast (CEF) cells suspended in a serum-free medium containing no material of direct animal origin, harvested from the CEF cells, purified, and concentrated by several Tangential Flow Filtration (TFF) steps including benzonase digestion. Each 0.5 mL dose is formulated to contain 0.5 x  $10^8$  to  $3.95 \times 10^8$  infectious units of MVA-BN live virus in 10 mM Tris (tromethamine), 140 mM sodium chloride at pH 7.7. Each 0.5 mL dose may contain residual amounts of host-cell DNA ( $\leq 20$  mcg), protein ( $\leq 500$  mcg), benzonase ( $\leq 0.0025$  mcg), gentamicin ( $\leq 0.163$  mcg), and ciprofloxacin ( $\leq 0.005$  mcg).

#### 5.1.2 Dosing and Administration

In this platform trial, only JYNNEOS (MVA-BN vaccine) is being evaluated and there is no placebo group. Vaccine will be administered by subcutaneous injection in the fatty subcutaneous tissue of the upper arm. See the MOP for additional details.

In Stage 2, the second vaccination will be given in the contralateral arm unless the site deems that using the same arm is in the best interest of the participant in terms of safety or using the same arm (for the second injection) will enable the site to better evaluate reactogenicity (e.g., tattoo on opposite upper arm). If the second vaccination is given in the same arm as the first vaccination, the second injection should be given approximately 5 cm away from the first injection site if physically possible.

Table 3 Study Arms Stage 2 (Adult and Adolescent)

| Arm | Dose of JYNNEOS (MVA-BN) | Route of Administration* | Vaccination | Day |
|---|---|---|---|---|
| | | | Day 1 | Day 29 |
| 4 (Adult) | 1 x 10 <sup>8</sup> TCID <sub>50</sub> (0.5 mL) | Subcutaneous | X | X |

| 5 (Adolescent) | 1 x 10 <sup>8</sup> TCID <sub>50</sub> (0.5 mL) | Subcutaneous | X | X |
|---|---|---|---|---|

<sup>\*</sup>Subcutaneous is administered in the fatty subcutaneous tissue of the upper arm.

#### **5.1.3 Dose Escalation**

Not Applicable.

#### **5.1.4 Dose Modifications**

Not Applicable.

#### 5.1.5 Criteria for Redosing

If study product administration is unsuccessful, another administration will not be attempted.

# 5.2 Preparation/Handling/Storage/Accountability

#### 5.2.1 Acquisition and Accountability

See main section of this document for information about accountability and disposition of the study product, JYNNEOS (MVA-BN vaccine).

### 5.2.2 Formulation, Appearance, Packaging, and Labeling

See main section of this document for information about JYNNEOS.

#### **5.2.3** Product Storage and Stability

See main section of this document for information about storage and stability of JYNNEOS.

#### 5.2.4 Preparation

Each dose (0.5 mL) is supplied in a single-dose vial. Sites should allow the vaccine to thaw and reach room temperature before use (about 15 to 30 minutes). After thawing, the total time stored at +2°C to +8°C (+36°F to +46°F) should not exceed 4 weeks. Once the vial is punctured and a dose is withdrawn, if it is not used in its entirety, it should be stored at +2°C to +8°C (+36°F to +46°F) and discarded within 8 hours of the first puncture. If the unpunctured vial is initially shipped/stored at 2-8C then it is stable for up to 8 weeks. Sites should not refreeze the vaccine. JYNNEOS may be kept frozen until the expiration date.

JYNNEOS is a light yellow to pale white colored, milky suspension when thawed. Sites will visually inspect the product for particulate matter and discoloration prior to administration. If either condition is present, the vaccine will not be administered. Study product administrators will gently swirl the vial for at least 30 seconds.

For the SC injection (Arms 4 and 5), 0.5 mL of vaccine will be withdrawn from the vial into a sterile syringe and injected into the fatty subcutaneous tissue of the upper arm.

DMID/NIAID/NIH 

See the protocol-specific MOP for detailed information on the preparation, labeling, storage, and administration for each study arm.

# 5.3 Measures to Minimize Bias: Randomization and Blinding

### **5.3.1** Treatment Assignment Procedures

All participants in Stage 2 will receive the 2-dose SC regimen of 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN.

#### 5.3.2 Randomization

Stage 2 is not randomized. All Stage 2 participants will receive the 2-dose SC regimen of  $1 \times 10^8$  TCID<sub>50</sub> MVA-BN. For Stage 2, the aim is to enroll at least 25% adolescents ages 12 to 14 years.

## **5.3.3** Blinding and Masking Procedures

This study will not utilize blinding or masking procedures as it is an open-label, non-placebo-controlled trial. Research laboratories will be blinded to participant study arm for the purposes of immunogenicity/efficacy evaluations.

# 5.4 Study Intervention Compliance

Each dose of JYNNEOS will be administered by a member of the clinical research team that is qualified per state and institution policies to administer the study product. Administration and date, time, and location of injection will be recorded on the appropriate eCRF.

# 5.5 Concomitant Therapy

At screening (i.e., the screening visit or Day 1 visit if the screening visit is not conducted), participants will be asked about receipt of immunosuppressive therapy, experimental therapeutic agents and vaccines, other medications, and vaccines. At each subsequent study visit through Day 57, new concomitant medication(s) and changes to existing medications will be recorded as well as receipt of a vaccine. For this study, concomitant medications to be reported in the Case Report Form (CRF) are prescription drugs, over-the-counter medications, and supplements. Concomitant medications taken and vaccines received in the 4 weeks prior to providing informed consent will be recorded in the CRF. Any drug taken or vaccine received by the participant during the trial should be recorded on the appropriate CRF through Day 57. In Stage 2, after Day 57, concomitant medication associated with a protocol specified AESI or related MAAE occurring through Day 210 and clinically relevant to report will be recorded in the CRF. After Day 57, concomitant medication associated with a related SAE occurring through the end of study and clinically relevant to report will be recorded in the CRF. Clinically relevant is defined as a medication that is prescribed or dose of an existing medication changed because of a SAE, AESI or MAAE. Medications taken that are unrelated to the adverse event do not need to be recorded (e.g., topical medication for acne). An exception to this schedule for recording concomitant therapy is during sick visits for those who have laboratory-confirmed mpox (illness). During sick visits, concomitant medications and treatment will be collected.

Medications that might interfere with the evaluation of the immune response to MVA-BN should not be used by the participant during the study-reporting period unless clinically indicated as part

DMID/NIAID/NIH 

of the participant's health care for a condition diagnosed after enrollment. This would include any systemic immunosuppressant medication that may impact the immunogenicity endpoints. In the event medical conditions dictate the use of these medications, participants are encouraged to obtain adequate care, comply with the course of therapy as prescribed by their physician and inform the study Investigator as soon as practical.

# 6. STUDY INTERVENTION DISCONTINUATION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

# 6.1 Halting Criteria and Discontinuation of Study Intervention

## 6.1.1 Study Halting Criteria

Stage 2 will be paused if any of the following four events occur:

- 1. One (1) participant experiences a SAE after the administration of the vaccine that is considered related to the vaccine.
- 2. One (1) participant experiences a Grade 4 solicited AE after the administration of the vaccine that is considered related to the vaccine.
- 3. Three (3) or more participants experience a Grade 3 or higher unsolicited AE coded to the same High-Level Term based on the medical dictionary for Regulatory Activities (MedDRA) that are deemed related to the vaccine.
- 4. Two or more participants experience a protocol specified AESI regardless of relatedness or severity.

In the event a halting rule is met, an unscheduled safety analysis by the DSMB will be required for approval of further enrollment. Further administration of the vaccine, including a second dose, is suspended for all participants until an assessment by the DSMB takes place.

#### **6.1.1.1** Sentinel Participant Halting Rules

Not Applicable.

#### **6.1.1.2** Cohort Halting Rules

Not Applicable.

#### 6.1.2 Individual Halting Criteria

If a single participant meets an individual halting criterion, this will not halt the whole study but halts the participant's involvement in terms of the administration of the second dose of the vaccine. However, while the participant is discontinued from receipt of vaccine, they should be encouraged to remain in the study to monitor safety and evaluate immunogenicity until the end of the study.

For Stage 2, all five criteria listed below apply:

DMID/NIAID/NIH 

1. Any participant experiences laryngospasm, bronchospasm, or anaphylaxis within 24 hours after the administration of the vaccine that is considered related to the vaccine within the 24 hours after vaccination.

- 2. Any participant experiences generalized urticaria (defined as urticarial lesions occurring at more than two body parts) within 3 days after the administration of the vaccine.
- 3. Any participant experiences any Grade 4 solicited AE or an SAE after the administration of the vaccine that is deemed related to the vaccine.
- 4. Any participant that experiences ulceration, abscess or necrosis at the injection site that is considered related to the vaccine administration.
- 5. Any participant experiences signs and symptoms consistent with myocarditis or pericarditis after the first vaccination and before the second vaccination is given.

A participant may be removed from the study if the Investigator or the medical monitor deems it in the best interest of the participant. The participant could be withdrawn from the study at any time during the trial.

#### 6.1.3 Follow up for participants that discontinued study intervention

Discontinuation from vaccination administration does not mean discontinuation from the study, and remaining study procedures should be completed as indicated by the study protocol. If a clinically significant finding is identified (including, but not limited to changes from baseline) after enrollment, the investigator or qualified designee will determine if any change in participant management is needed.

The second vaccination will not be given, but other follow up visits will continue, if the participant:

- Becomes pregnant.
- Develops mpox (symptomatic, laboratory-confirmed disease) after the first vaccination
- Meets an exclusion criterion for participation in the study (either newly developed or not previously recognized) that precludes further study participation.

If a participant meets an exclusion criterion after enrollment and first dose, it does not necessarily mean the participant cannot receive the second dose of JYNNEOS. The decision of what "precludes further study participation" depends on what exclusion criteria are met, with a focus on what is best for participant safety. The most likely exclusion criteria to be met are participants that receive a licensed vaccine after enrollment (i.e., exclusion criteria 7 and 8). If a participant receives an off-study vaccine during the study-defined restricted time periods (i.e., as defined in exclusion criteria and Section 5.4), receipt of the off-study vaccine should be reported as a deviation. The participant can receive the second study vaccination if the investigator determines that the participant is otherwise eligible to receive the second MVA-BN in this trial.

There is no reactogenicity threshold for administration of the second dose of vaccine, that is the second dose may be administered even if there is residual erythema, induration or other reactogenicity from the first vaccination. Participants and if applicable parent(s)/legal authorized representative (LAR) may decline the second vaccination for any reason at the Day 29 visit and will be discontinued from the study intervention. Parental/LAR permission is ongoing throughout the study and will be confirmed prior to the second vaccination. See MOP for operational details.

DMID/NIAID/NIH 

However, if second vaccination is declined, the participant should remain in the study and followed for safety and immunogenicity through Day 394 visit unless they withdraw from the study.

The data to be collected at the time of study intervention discontinuation will include:

- Reason for discontinuation study vaccination including, but not limited to, unacceptable (intolerable) reactogenicity, new medical condition identified that places participant at risk, participant or parent(s)/LAR(s) unwillingness to have second vaccination.
- Confirmation of willingness to remain in the study and understanding of study schedule.

# 6.2 Participant Withdrawal from the Study and Replacement

Participants and if applicable parent(s)/LAR(s) are free to withdraw from participation in the study at any time upon request. An investigator may withdraw a participant from the study if the participant:

- Has an AE or other medical condition that continued participation in the study would not be in the best interest of the participant.
- Is lost to follow-up

The reason for participant discontinuation or withdrawal from the study, whether the decision was made by investigator, participant, or parent(s)/LAR(s), and the extent of the withdrawal (i.e., whether participant withdrew from all components of research study or just the study intervention) will be recorded on the CRF. If the participant agrees, every attempt will be made to follow all AEs through resolution (return to baseline) or until defined as stable. The investigator will inform the participant and if applicable parent(s)/LAR(s) that already collected data will be retained and analyzed for this study even if the participant withdraws from this study. Biospecimens collected will still be used to analyze the study endpoints.

Participants who withdraw, or are withdrawn from this study, or are lost to follow-up after signing the ICF and administration of the study product will not be replaced.

# 6.3 Lost to Follow-Up

A participant will be considered lost to follow-up if he or she fails to return for two scheduled visits and is unable to be contacted by the study site staff after three attempts. Extensive effort (i.e., generally three documented contact attempts via telephone calls, e-mail, etc., made on separate occasions) will be made to locate or recall the participant, or at least to determine the participant's health status. These efforts will be documented in the participant's study file.

# 7. STUDY ASSESSMENTS AND PROCEDURES

# 7.1 Screening Procedures

In this study, screening assessments can occur in an optional screening visit on Day -7 to -1, or at Visit 1 on Day 1 before the first vaccination. At the time of the screening assessment, the participant and if applicable parent(s)/LAR(s) will be provided with detailed study information and written informed consent or parental/LAR permission and informed assent, where appropriate,

DMID/NIAID/NIH 

will be obtained. The following assessments are performed to determine eligibility requirements as specified in the inclusion and exclusion criteria:

- Obtain demographic data.
- Obtain mpox exposure history in the 3 weeks prior to signing ICF.
- Review vaccination history, including any experimental vaccines, and determine receipt of exclusionary vaccine(s):
  - Live vaccine or a COVID-19 vaccine in the prior 4 weeks or an inactivated non-COVID-19 vaccine in the prior 1 weeks.
  - o Licensed or investigation smallpox or mpox vaccine.
- Obtain medical history. Ask specifically about worsening of any chronic medical condition, hospitalizations, or history of COVID-19 (with positive test for SARS-CoV-2, including those performed at home) in the prior 4 weeks, and whether they have the following medical conditions:
  - o HIV infection
  - o History of mpox, cowpox or vaccinia infection
  - o History of anaphylaxis or severe adverse reaction to a vaccine or vaccine product
  - o History of allergy to gentamicin, ciprofloxacin, chicken or egg protein
  - o History of myocarditis or pericarditis, congenital heart defect or cardiac dysrhythmia (Stage 2 only, adolescents and adults)
- Review medications and therapies up to 4 weeks prior to signing ICF and record on the appropriate CRF and determine receipt of exclusionary medication(s):
  - o Experimental therapeutic agent (or vaccine) in the 3 months prior to consent.
  - Use of immunosuppressing drugs prior to consent.
- Perform targeted physical examination and inspect arms for smallpox vaccination scar
- Measure vital signs (HR, BP, and temperature).
- Review of birth control history with female of reproductive potential who are having sexual intercourse with male partners.
  - Counsel participants to use adequate birth control methods required during the trial to avoid pregnancy.
  - o Do serum or urine pregnancy test (in female participants of reproductive potential).
- Review inclusion and exclusion criteria.

The overall eligibility of the participant to participate in the study will be assessed once all screening values are available. The screening process can be suspended prior to complete assessment at any time if exclusions are identified by the study team.

Study participants who qualify for inclusion will be enrolled.

# 7.1.1 Procedures to be Followed in the Event of Abnormal Clinical Laboratory Test Values or Abnormal Clinical Findings During Screening

A participant may be re-screened once if a protocol eligibility criterion that is not met at the initial time of screening, will be met by rescreening at a later date. No participant may be screened more than twice due to a screening failure result.

DMID/NIAID/NIH 

Participants will be provided the results of pregnancy testing and abnormal clinical findings necessitating follow-up at the discretion of the participating site PI or appropriate sub-investigator.

#### 7.2 Sick Visit

Participants with signs and symptoms consistent with mpox (e.g., vesicular or pustular lesions, fever, chills, lymphadenopathy, malaise, myalgias, headache, or respiratory symptoms) during the study are asked to call the study site. Those who have laboratory-confirmed mpox will be evaluated at the clinical site; those who have not been tested will be asked to have a diagnostic test done. During the visit, the participant will be asked about the current illness (e.g., onset date, treatment received) and for information about the diagnostic testing that was done. Participants will have a targeted physical examination done. For more information about this visit, see the MOP and the CRF.

# 7.3 Additional Study Procedures in Stage 2

## 7.3.1 Phone Visits

In Stage 2, the Day 57 visit may occur via phone call visit if the participant has no skin changes found on physical examination at either injection site documented at the Day 43 visit. However, the site may opt to have the participant come in for an in-person visit if deemed necessary. In addition, those who qualify for a phone visit at Day 57 may have the visit conducted virtually via video teleconference (e.g., Zoom, FaceTime) if deemed necessary. If an in-person visit is thought to be necessary, the clinical site may do a physical examination on an as needed basis.

In Stage 2, Visit 7 (Day 90) is conducted by phone (teleconference call) by a delegated study staff member. However, the site may choose to conduct the visit by virtual method (e.g., Zoom, FaceTime) or in-person.

#### 7.3.2 Photography

In Stage 2, study staff may ask participants for permission to photograph the vaccination site for purposes of clinical documentation and follow-up. Photographs will contain no participant identifying information. Participants may grant or decline permission for photography without any effect on their participation in the study. Photographs will not be entered into the study database or used for determination of study objectives.

#### 7.3.3 Missed Study Visits

Participants should complete all study visits as specified in the SOA. Phone or virtual video teleconferences may be considered for subjects who cannot return for protocol specified in-clinic visits but are willing to be contacted by alternate means. See MOP for additional details.

# 7.4 Immunogenicity Assessments

# 7.4.1 Immunogenicity/Efficacy Evaluations

DMID/NIAID/NIH 

Prior comparator studies used the Bavarian Nordic (BN) Vaccina virus Western Reserve strain (VV-WR) plaque reduction neutralizing antibody (PRNT) assay and enzyme-linked immunosorbent assay (ELISA) to evaluate immunogenicity. For Stage 2, VV-WR PRNT will be used as the primary assay and plan to test timepoints of Days 1, 29, 43, 210, and 394.

This study will also measure a MPXV specific PRNT and will test a minimum of 2 timepoints (Days 1 and 43). The MPXV PRNT assay is not yet developed, and therefore this endpoint is as an exploratory endpoint. Additional timepoints for each will be evaluated as able (given lab throughput and cost).

# 7.4.2 Exploratory Assessments

Additional assessments of humoral immunity including ELISAs may be performed on samples from this trial.

# 7.5 Safety and Other Assessments

Study procedures are specified in the SOA and more detailed information as needed is provided in the MOP. A study clinician, licensed to make medical diagnoses and listed on the Form FDA 1572 as the participating site PI or appropriate sub-investigator, will be responsible for all study-related medical decisions.

- Medical history
  - o A complete medical history will be obtained by interview of participants at screening (i.e., the screening visit or on Day 1 if no screening visit is conducted).
  - O An interim medical history will be obtained by interview of participants at subsequent study visits or ad hoc telephone call with participant. Any changes since the previous clinic visit will be noted. The interim medical history should include an assessment for adverse events and new medical conditions.
- Physical examination
  - Stage 2: A targeted (symptom-driven) physical exam will be done at screening (i.e., screening visit or Day 1), on Days 8, 29, 36, and 43 (at least assessment of vaccination site and presence of skin discoloration and nodules will be done), and as needed in all other visits if interim change in medical status reported by participant.
- Reactogenicity Assessments
  - Reactogenicity assessments of solicited systemic reactogenicity occurring from the time of each vaccination through 7 days post each vaccination (Days 8 and 36 respectively) in Stage 2 will include fever, chills, nausea, headache, fatigue, change in appetite, myalgia, and arthralgia.
  - O Assessments of solicited local (injection site) reactogenicity occurring from the time of each vaccination 7 days post each vaccination in Stage 2 will include pain at injection site, erythema/redness, induration/swelling, and pruritis at site.
  - o In Stage 2, any ongoing events at Day 8, Day 36, or Day 43 will be followed at subsequent visits in order to note a resolution date. See Memory Aid section below on measurement of ongoing erythema/redness and/or induration/swelling.
- Memory Aid

DMID/NIAID/NIH 

> For Stage 2, the participant will document local and systemic reactogenicity from the time of each vaccination through 7 days post vaccination (Days 1 through 8 and Days 29 through 36).

- Memory Aids will be reviewed with the participants for any solicited reactions, as well as unsolicited AEs and SAEs.
- o The vaccination injection site will be examined at all visits until symptoms resolve.
- o In Stage 2, for those with no residual systemic or local reactogenicity at the Day 8 or Day 36 visit, no more data is collected by the participant in the Memory Aid.
- o For those with ongoing systemic and/or local reactogenicity at Day 8 and 36 in Stage 2, they will be asked to do the following:
  - Measure erythema/redness and/or induration/swelling and record in the Memory Aid until it has resolved, if applicable.
  - Record end date of all other signs and symptoms.
- O Nodules and hyperpigmentation are unsolicited AEs, and not collected in the Memory Aid to avoid double counting these events which tend to develop at end of second week as a post-inflammatory reaction. Occurrence will be documented on the physical examination eCRF and the unsolicited AE eCRF, and severity assessed per Section 8.6.3.1.
  - Nodules and hyperpigmentation will be followed through resolution.
- O Site research teams will review and align the subject responses on the memory aid with clinical assessments.

#### Vital signs

- o Vital sign measurements will include systolic and diastolic BP, HR, and oral temperature. Vital signs will be measured at timepoints specified in the SOA.
- Clinical laboratory evaluations
  - Serum or urine pregnancy test will be performed locally by the site laboratory at the screening and must be negative within 24 hours prior to each vaccination on Days 1 and 29. This means that if the screening visit is conducted more than 24 hours prior to vaccination, pregnancy test will need to be done on Day 1. Pregnancy tests may be done as needed at interim or unscheduled visits for all females of reproductive potential.
  - o Results must be confirmed as negative prior to enrollment on Day 1 and administration of each vaccination.

#### 7.5.1 Alternative Schedules

Given that peak humoral response after the second JYNNEOS vaccination is the primary endpoint and is likely to occur approximately two weeks (Day 43) to four weeks (Day 57) after the second dose is administered, it is important that subsequent visits occur within the protocol-specified window after the second dose is given. If a participant is unable to receive the second dose within the pre-specified window, the site should contact DMID to discuss an alternate schedule. If a participant receives the second dose on any day other than Day 29, the target date of the remaining scheduled visits will be shifted, as appropriate so that immunogenicity timepoints post-second vaccination are consistent among participants.

Participants may not receive Dose 1 or Dose 2 of JYNNEOS within 4 weeks of COVID-19 illness (with positive test for SARS-CoV-2 including those performed at home by the participant) or

DMID/NIAID/NIH 

receipt of a COVID-19 vaccine. This may require the second JYNNEOS dose to be delayed if a participant develops COVID-19 or receives a COVID-19 vaccine while enrolled in the study but after receiving Dose 1. See MOP for additional information.

# 7.5.2 Procedures to be Followed in the Event of Abnormal Clinical Laboratory Test Values or Abnormal Clinical Findings During the Trial

In this study, there will be no clinical laboratory screening or safety tests done except for pregnancy testing. Participants will be notified of the results of the pregnancy test.

## 7.6 Adverse Events and Serious Adverse Events

See the main document for standard definitions of adverse events (AE), solicited AEs, unsolicited AEs, and serious adverse events (SAE).

### 7.6.1.1 Definition of Medically Attended Adverse Events (MAAE)

A medically attended adverse event (MAAE) is defined as AEs with medically attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Adverse events (e.g., abnormal vitals) identified at a routine study visit will not be considered MAAEs. In Stage 2, MAAEs that are deemed related to the vaccine or vaccination procedure will be collected from Day 1 through 210 and all SAEs will be collected from Day 1 through the end of the study.

## 7.6.1.2 Definition of Suspected Unexpected Serious Adverse Reactions (SUSAR)

A SUSAR is a SAE that is considered related to study product and unexpected. Unexpectedness to study product will be determined by what is listed in the JYNNEOS package insert.

### 7.6.1.3 Definition of Adverse Event of Special Interest (AESI)

In Stage 2, protocol specified Adverse Events of Special Interest (AESIs) will be collected. AESIs are any adverse events for which additional data (in addition to standard AE data) are desired. The Sponsor (DMID), regulatory agency, or industry partner may request AESI reporting; the decision to collect AESI may be driven by a regulatory requirement or a known/potential risk from the study product or class. Non-structured data similar to SAEs will be collected for AESIs. AESIs encompass the following terms:

#### **Protocol Specified AESIs**

For Stage 2 of this trial, a protocol specified AESI is defined as a case of myocarditis or pericarditis. All participants with signs and symptoms of myocarditis/pericarditis (e.g., chest pain, shortness of breath, palpitations, etc.) in whom myocarditis/pericarditis is excluded, or for whom an alternative diagnosis is made, will not be considered a suspect case and as such, not reported as an AESI. All other suspected cases of myocarditis or pericarditis should be reported as an AESI and the case adjudicated using the Brighton Collaboration case definitions for myocarditis and pericarditis. The Brighton Collaboration case definitions will be used to classify into possible, probable, or definite myocarditis or pericarditis cases.<sup>43</sup> In Stage 2, protocol specified AESIs will be collected from Day 1 through 210.

DMID/NIAID/NIH 

#### 7.6.2 Classification of an Adverse Event

See main section of the protocol for a description of the classification of an AE in terms of severity and causality.

### 7.6.3 Time Period and Frequency for Event Assessment and Follow-Up

For Stage 2, adverse events will be collected during the following time periods:

- Systemic and local solicited adverse events will be collected from Day 1 through Day 8, and Day 29 through Day 36. However, participants with ongoing systemic and/or local reactogenicity at Day 8 or Day 36 visit, will be asked to measure erythema/redness and/or induration/swelling until it has resolved, if applicable, and record end date of all other signs and symptoms.
- Unsolicited adverse events will be collected from Day 1 through Day 57.
- For Stage 2, all SAEs will be collected from Day 1 through Day 394 (i.e., the end of study). Protocol specified AESIs, and related MAAEs will be collected from Day 1 through 210.

All AEs, related MAAEs, protocol specified AESIs, and SAEs will be followed through resolution or until the site investigator deems the event to be chronic or the participant is stable.

# 7.6.4 Adverse Event Reporting

See the main section of the protocol for a description of AE reporting.

# 7.7 Unanticipated Problems

See the main section of the protocol for a definition of Unanticipated Problems (UP) and information regarding UP reporting.

# 8. STATISTICAL CONSIDERATIONS

# 8.1 Statistical Hypotheses

Stage 2 will test non-inferiority of the 1 x  $10^8$  TCID<sub>50</sub> MVA-BN SC regimen (standard dose regimen) in adolescents compared to adults.

### **Primary Hypothesis**

• At Day 43 the humoral immune response of the 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN SC (standard dose regimen) in adolescents will be non-inferior to the standard 1 x 10<sup>8</sup> MVA-BN SC regimen in adults, as assessed by PRNT GMT.

#### **Secondary Hypotheses**

DMID/NIAID/NIH 

• At Day 394 the humoral immune response of the 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN SC regimen in adolescents will be non-inferior to the standard 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN SC regimen in adults, as assessed by PRNT GMT.

- The humoral immune response of the 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN SC regimen in adolescents, as assessed by PRNT GMT, will be similar to the 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN SC regimen in adults at all study days.
- The humoral immune response of the 1 x  $10^8$  TCID<sub>50</sub> MVA-BN SC regimen in adolescents as assessed by vaccinia specific PRNT half-life, will be similar to the 1 x  $10^8$  TCID<sub>50</sub> MVA-BN SC regimen in adults.
- The humoral immune response of the 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN SC regimen in adolescents, as assessed by monkeypox specific PRNT GMT, will be similar to the 1 x 10<sup>8</sup> TCID<sub>50</sub> MVA-BN SC regimen in adults at Day 1 and 43.

# 8.2 Sample Size Determination

As a primary endpoint in Stage 2, 500 participants (130 adults in Arm 4; 70 adults in Arm 3 (Stage 1); 300 adolescents in Arm 5) will provide approximately 92% power for a test of non-inferiority of geometric mean titers using unequal variances and two-sided, type I error of 0.05 (Table 4). This assumes that the adult arm will have a standard deviation of 0.6 and adolescent arm will have a standard deviation of 0.5. The standard deviation on Day 42 in prior large studies using the SC route was 0.41 (Pittman, NEJM 2019) and 0.59 (Frey, Vaccine 2015), so the estimates used in calculations are justifiable (Table 5 and Table 6). Stage 2 will enroll approximately 450 participants (135 adults in Arm 4; 315 adolescents in Arm 5) assuming a 5% drop-out rate. Participant enrollment into the adolescent cohort will be stratified into two 3-year age groups, at least 78, adolescents ages 12 to 14 years and a maximum of 237, adolescents ages 15 to 17 years, in order to ensure that adequate numbers of younger adolescents are enrolled (i.e., about 25% of all adolescents enrolled). Arms 3 and 4 will be combined as a comparator group in the primary analysis. It is not anticipated that there will be significant differences in immunogenicity outcomes between these two groups, however, a sensitivity analysis excluding Arm 3 participants will be performed, and will be described in the statistical analysis plan (SAP).

#### **Table 4: Power Calculation**

Power calculations for a non-inferiority test of means using unequal variances and two-sided type one error rate of 0.05. Non-inferiority margin of 0.67.

| NI Margin | Sample Size<br>Arm 5<br>(Standard<br>Deviation<br>0.5) | Sample Size<br>Arm 3+4<br>(Standard<br>Deviation 0.6) | Total sample size for NI test | Power |
|---|---|---|---|---|
| $0.67 \\ \text{Log}_{10}(0.67) = -0.174$ | 300 | 200 | 500 | 0.92 |

#### **Table 5: Standard Deviation Estimates**

Standard deviation estimates computed from Table S4 of Pittman et al, 2019<sup>44</sup>

| | MVA-BN | | | | | A( | CAM2000 | Ratio of | 95% CI |
|------|--------|-----|--------|----|---|-----|---------|----------|--------|
| Week | N | GMT | 95% CI | SD | N | GMT | 95% CI | SD | GMTs |

Protocol 22-0020 Appendix B Version 7.0 23 May 2024

| | | | | (for<br>log <sub>10</sub><br>GMT) | | | | (for<br>log <sub>10</sub><br>GMT) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| 2 | 184 | 16.2 | [13.0, 20.1] | 0.65 | 184 | 16.2 | [13.1, 20.0] | 0.63 | 0.997 | [0.738, 1.348] |
| 4 | 185 | 16.9 | [13.7, 20.8] | 0.63 | 186 | 79.3 | [67.1, 93.8] | 0.51 | 0.213 | [0.163, 0.278] |
| 6 | 185 | 153.5 | [134.3, 175.6] | 0.41 | 181 | 64.7 | [54.9, 76.2] | 0.49 | 2.372 | [1.922, 2.928] |
| 8 | 179 | 118.2 | [102.9,135.8] | 0.41 | 183 | 67.1 | [56.9, 79.0] | 0.49 | 1.763 | [1.422, 2.185] |
| Peak | 185 | 153.5 | [134.3, 175.6] | 0.41 | 186 | 79.3 | [67.1, 93.8] | 0.51 | 1.935 | [1.562, 2.397] |

**Table 6: Standard Deviation Estimates** 

Standard deviation estimates computed from Frey et al, 2015<sup>21</sup>

| Study visit day | Liquid SC 1x10 <sup>8</sup><br>N=149 | Liquid ID 2x10 <sup>7</sup><br>N=146 | | |
|---|---|---|---|---|
| | VV-WR GMT [95% CI] | SD | VV-WR GMT [95% CI] | SD |
| Day 14 | 10.0 [9.0, 11.1] | 0.28 | 10.3 [9.3, 11.3] | 0.27 |
| Day 28 | 9.6 [8.7, 10.6] | 0.27 | 10.8 [9.9, 11.9] | 0.23 |
| Day 42 | 45.2 [36.4, 56.2] | 0.59 | 54.4 [43.7, 67.8] | 0.59 |
| Peak post 2 <sup>nd</sup> vaccination | 49.5 [40.0, 61.3] | 0.58 | 59.6 [48.1, 74.0] | 0.59 |

# 8.3 Statistical Analyses

## 8.3.1 General Methodology

For Stage 2, the non-inferiority of adolescent immune response relative to adult immune response will be determined using a non-inferiority (NI) margin of 0.67 (NI=-0.174 log10 scale). No stepwise testing will be done in Stage 2. The primary safety endpoint is descriptive with no hypothesis testing planned.

## 8.3.2 Timing of Analyses

## 8.3.2.1 Interim Safety Analyses

AEs and SAEs may be reviewed as necessary outside of DSMB reviews. The DSMB may not need to meet (unless halting rules are met) and materials will be provided electronically. Documentation of review and any concerns noted will be solicited electronically.

The DSMB will review separate cumulative AE data reports for all participants within each arm. Given the safety database known for authorized/approved vaccines, there is no routine mandatory review by the DSMB unless halting rules are triggered.

## 8.3.2.2 Interim Immunogenicity Analyses

For Stage 2, interim immunogenicity analyses may be conducted and will include at least an analysis of Vaccinia virus specific PRNT GMT at Day 1 and 43 and Monkeypox virus specific PRNT GMT at Day 1 and 43.

Data may be disseminated to public health officials and partners as needed and included in publications and presentations to inform the global scientific community.

## 8.3.2.3 Final Analyses

Due to the 2023-2024 outbreak of mpox in the Democratic Republic of the Congo<sup>45</sup> an interim

DMID/NIAID/NIH 

Clinical Study Report (CSR), including an analysis of immunogenicity through Day 43 and safety through Day 210, will be produced to inform public health needs. The interim CSR will be prepared once all participants have completed the Day 210 visit and all of the relevant data have been cleaned and the database has been locked. The results in the interim CSR will be considered final for all immunogenicity endpoints through Day 43 and the clinical and safety endpoints followed up to Day 210. Any SAEs or study withdrawals occurring after Day 210, along with results from the analysis of outstanding immunogenicity data, will be detailed in an addendum to the CSR after the study is complete.

Results from the interim CSR and the subsequent CSR addendum will be disseminated to public health officials and partners as needed and included in publications and presentations to inform the global scientific community.

## **8.3.3** Populations for Analyses

There will be three analysis populations in this study. The safety analysis population includes all enrolled participants who received at least one dose of study vaccine. Analyses for the safety population will include safety reported through the end of the study. The modified intent-to-treat (mITT) population includes all participants who received at least one dose of vaccine and contributed both pre- and at least one post-vaccination venous blood sample for immunogenicity testing for which valid results were reported.

In the final analysis, protocol deviations will be reviewed to determine which protocol deviations may affect the analysis. The per protocol (PP) population will then be defined – and this includes all participants in the mITT subset with the following exclusions:

- Data from all available visits for participants found to be ineligible at baseline.
- Data from all visits after the protocol deviations that are considered to affect the science (as determined by the sponsor at an ad hoc meeting).
- Data from any visit that occurs substantially out of window.

For the PP and mITT analyses, participants will be analyzed according to the study product that they received.

#### 8.3.4 Baseline Characteristics and Participant Disposition

Summaries of demographic characteristics of the study population including age, sex, ethnicity, and race will be presented by vaccination arm and overall. In addition, this descriptive analysis will be done by reported HIV infection status.

#### 8.3.5 Immunogenicity Analyses

Descriptive summaries of immunogenicity data will be presented for the mITT population. If there are protocol deviations which may affect the analysis, a PP analysis may also be performed.

Geometric Mean Titers (GMT) and Geometric Mean Fold Rise (GMFR) from baseline of VV-WR PRNT will be calculated, along with 95% CIs, for all groups, at each timepoint. Summaries will

DMID/NIAID/NIH 

also be displayed graphically. Geometric Mean Titer Ratio, defined as the ratio of each ID arm to the control SC arm, will also be reported at each timepoint, along with 95% CIs. There are no imputations planned for missing data.

A SAP for Stage 2 will be developed and will detail the full planned analysis.

#### 8.3.6 Safety Analyses

In Stage 2 of this study, the safety outcomes for the two study arms will be evaluated including systemic reactogenicity for 7 days after each vaccination, local reactogenicity for 7 days after each vaccination, and unsolicited adverse events for 28 days after each vaccination. In Stage 2, protocol specified AESIs, and related MAAEs will be evaluated from Day 1 through Day 210. All SAEs will be evaluated from Day 1 through Day 394 or the end of the study (see SOA).

## 8.3.6.1 Reactogenicity

The number, percentage (observed rate) and exact two-sided 95% CI for participants reporting each solicited local (injection site) reaction and solicited systemic reaction following vaccination will be summarized by study arm after first and second vaccination, and overall (i.e., after any vaccination). In addition, the most severe local and systemic reactions recorded during the follow-up period (i.e., maximum severity) for each participant will be determined and summarized by study arm following each vaccination (as well as overall) and the resulting number and percentage of participants will be summarized by severity grade (none, mild, moderate, severe, life-threatening). Last, the daily severity of local and systemic reactions will be determined for each participant and the proportion of participants having a sign/symptom each day will summarized by grade and presented by study arm following each vaccination. Rates for any severe (Grade 3 or 4) solicited local or systemic reaction following any vaccination will be compared between study arms.

#### 8.3.6.2 Other Adverse Events

The number of associated unsolicited AEs, protocol specified AESIs (Stage 2 only), MAAEs and SAEs following vaccine administration is expected to be small. A complete listing of all events will therefore be provided, including the nature of the event, timing relative to vaccination, severity, duration, and the investigator's assessment of the likely relationship to vaccination. For each type of AE, the observed rate and exact two-sided confidence intervals will be computed for each study arm and listed by toxicity grade. AEs will be MedDRA® coded for preferred term and system organ class. Event rates and exact 95% confidence intervals for each study arm and the entire study cohort will be presented, in aggregate and by MedDRA® categories. Related unsolicited AE, protocol specified AESI (Stage 2 only), MAAE and SAE rates will be compared between the study arms.

The number, percentage (observed rate) for participants that withdrew or discontinued their vaccination series due to safety or reactogenicity events will be tabulated. Rates of withdrawal/discontinuation will be compared between study arms using Fisher's exact test.

Refer to the SAP for additional information.

DMID/NIAID/NIH 

Protocol 22-0020 Appendix B

23 May 2024

# 9. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

# 9.1 Regulatory, Ethical, and Study Oversight Considerations

This study will be conducted in conformity with the principles set forth in The Belmont Report: Ethical Principles and Guidelines for the Protection of Human Participants of Research (US National Commission for the Protection of Human Participants of Biomedical and Behavioral Research; April 18, 1979), and the federal policy for the Protection of Human Participants codified in 45 CFR Part 46, 21 CFR Part 50 (Protection of Human Participants), and the ICH E6(R2).

An OHRP-registered IRB will review and approve this protocol, associated informed consent, parental permission and assent documents, recruitment materials, and handouts or surveys intended for the participants, prior to the recruitment, screening and enrollment of participants. The IRB review shall be in accordance with 45 CFR 46 and 21 CFR 50, 21 CFR 56 (IRBs), and other federal, state, and local regulations and policies, as applicable.

Each institution engaged in this research will hold a current Federalwide Assurance (FWA) issued by the Office for Human Research Protections (OHRP) for federally funded research. and provide the FWA number to DMID. Each site principal investigator will obtain IRB approval for this protocol and any amendments to be conducted at his/her research site(s).

Any amendments to the protocol or informed consent, parental permission and assent documents will be approved by the IRB before they are implemented. IRB review and approval will occur at least annually throughout enrollment and follow-up of participants, in accordance with applicable regulations and the requirements of the IRB/IEC. The participating site PI will notify the IRB of deviations from the protocol and reportable SAEs, as applicable to the IRB policy.

DMID must receive the documentation that verifies IRB/IEC approval for this protocol, informed consent, parental permission and assent documents and associated documents, prior to the recruitment, screening and enrollment of participants, and any IRB approvals for continuing review or amendments as required by DMID.

#### 9.1.1 Informed Consent Process

Informed consent is a process that is initiated prior to an individual agreeing to participate in a trial and continuing throughout the individual's trial participation. Before any study procedures are performed, informed consent or parental permission and assent, where appropriate, will be obtained and documented. This research can be categorized as greater than minimal risk but presenting the prospect of direct benefit to the participant (45 CFR 46.405) given that MPXV may continue to cause disease in the U.S. in 2023. Given this, permission of one parent is sufficient for the adolescent participant.

Participants and the adolescent participant's parent or LAR will receive a concise and focused presentation of key information about the clinical trial, that includes both a verbal discussion as

DMID/NIAID/NIH 

well as written documentation. The key information about the purpose of the study, the procedures and experimental aspects of the study, study interventions/products, risks and discomforts, the expected duration of the participant's participation in the trial, any expected benefits to the participant, and alternative treatments and procedures that may be available to the participant. The explanation will be organized and presented in lay terminology and language that facilitates understanding why one might or might not want to participate, why one might or might not want to allow one's adolescent to participate or, in the case of assenting minors, why they themselves might or might not want to participate.

Participants and the adolescent participant's parent or LAR will receive an explanation as to whether any compensation and any medical treatments are available if injury occurs, and, if so, what they consist of, or where further information may be obtained. Participants and the adolescent participant's parent or LAR will be informed of the anticipated financial expenses, if any, to the participant for participating in the trial, as well as any anticipated prorated payments, if any, to the participant for participating in the trial. They will be informed of whom to contact (e.g., the investigator) for answers to any questions relating to the research project. Information will also include the foreseeable circumstances and/or reasons under which the participant's parent or LAR will be informed that participation is voluntary and that they are free to withdraw from the study for any reason at any time without penalty or loss of benefits to which the participant is otherwise entitled.

Participants and the adolescent participant's parent or LAR will be informed that records identifying the participant will be kept confidential, and, to the extent permitted by the applicable laws and/or regulations, will not be made publicly available and, if the results of the trial are published, the participant's identity will remain confidential. Participants and the adolescent participant's parent or LAR will be informed whether private information collected from this research and/or specimens will be used for additional research, even if identifiers are removed. They will be informed that the monitor(s), auditors(s), IRB, NIAID, and regulatory authority(ies) will be granted direct access to the participant's original medical records for verification of clinical trial procedures and/or data without violating the confidentiality of the participant, to the extent permitted by the applicable laws and regulations, and that, by signing a written informed consent or assent form, the participant is authorizing such access. Participants and the adolescent participant's parent or LAR will be allowed sufficient time to consider participation in this research trial and can discuss this trial with their family, friends or legally authorized representative, or think about it prior to agreeing to participate.

Informed consent, parental permission and assent forms will be IRB-approved, and participants will be asked to read and review the consent or assent form. Participants must sign the informed consent or assent form, where appropriate, prior to starting any study procedures being done specifically for this trial. Once signed, a copy of the informed consent or assent form will be given to the participant and the adolescent participant's parent or LAR for their records.

New information will be communicated by the site principal investigator to participants who consent to participate in this trial in accordance with IRB requirements. The informed consent and

DMID/NIAID/NIH 

Protocol 22-0020 Appendix B

23 May 2024

parental permission and assent documents will be updated, and participants will be re-consented per IRB requirements, if necessary.

# 9.1.1.1 Requirements for Permission by Parents/LARs and Assent by Children (in case of a minor)

Stage 2 of this study will enroll participants ages 12 to 17 years. Investigators or their designee will conduct the consent process with the parent or LAR, who will be given an IRB-approved permission form, which may be referred to as a consent form, to read, review, and sign prior to any study procedures. In addition, assent will be obtained in accordance with the approval by the site or central IRB.

The participant who reaches the age of majority or becomes emancipated during the study will be consented at the next visit prior to study procedures being performed. When no further visits are planned but the participant's participation is ongoing, the consent will be obtained via IRB-approved processes.

#### 9.1.1.2 Other Informed Consent Procedures

Participants and the adolescent participant's parent or LAR will be asked for consent and assent, where appropriate, to collect blood for the use of residual specimens and samples for secondary research. This extra/residual blood and corresponding serum will be used as back-up specimens for PP defined assays or designated for secondary research use and stored indefinitely at a designated storage facility. Collection of extra/residual samples during the study will help facilitate rapid follow-on analyses, if warranted, to provide more comprehensive scientific insights into the impact (safety and immunological) of the vaccine on the host response to vaccination. To maintain statistical power in follow-on analyses it is important that extra blood collection and secondary research use be included in as many participants as possible, due to the limited sample size per treatment arm. For this reason, if participants choose not to provide permission for extra blood and secondary research use, they will not be eligible for enrollment into the study.

The stored samples will be labeled with barcodes to maintain confidentiality. Research with identifiable samples and data may occur as needed, however, participant confidentiality will be maintained as described for this protocol and with IRB approval. Samples designated for secondary research use may be used for additional immunological assessments that may include but are not limited to antibody epitope mapping, B and T cell repertoire determination, nontraditional immune assay development, determination of innate immune factors and the ability of vaccine-induced antibodies to cross-react to different proteins and virus strains. These blood samples might be used in new or different immunological laboratory tests, to provide information for the development of new vaccines or therapeutics, or for the studies of monkeypox virus or other related viruses. Samples will not be sold for commercial profit. Although the results of any future research may be patentable or have commercial profit, participants will have no legal or financial interest in any commercial development resulting from any future research. There are no direct benefits to the participant for extra specimens collected or from the secondary research. No results from secondary research will be entered into the participant's medical record. Incidental findings will not be shared with the participant, including medically actionable incidental findings, unless required by law.

DMID/NIAID/NIH 

Risks are associated with the additional volume of blood collected, such as anemia. Risks for loss of privacy and confidentiality are described below. Participants may withdraw permission to use samples for secondary use at any time. They will need to contact the participating site and the samples will be removed from the study repository after this study is completed and documentation will be completed that outlines the reason for withdrawal of permission for secondary use of samples. Participants who withdraw consent before the last visit will not have the extra blood drawn for secondary use.

Participants will be asked to consent specifically on primary and secondary research samples. The consent process will include an explanation of the potential risks to the individual participants associated with data submitted to an NIH data repository and subsequent sharing. Data that may potentially identify human participants will not be released in unrestricted databases. Participants will be informed that analytical methods are associated with the risk of re-identification, even when specimens are de-identified. The consent will include whether individual participant data will be shared through a NIH controlled access data repository.

#### 9.1.2 Study Termination and Closure

Section 7, Study Intervention Discontinuation and Participant Discontinuation/Withdrawal, describes the temporary halting of the study. This study may be prematurely terminated if there is sufficient reasonable cause, including but not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants
- Results of interim efficacy or futility analysis
- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable
- Regulatory authorities' determination
- Sponsor's determination

If the study is prematurely terminated, the Principal Investigator (PI) will promptly inform study participants and the IRB and regulatory authorities as applicable. Study participants will be contacted, as applicable, and be informed of changes to study visit schedule. The PI will assure appropriate follow-up for the participants, as necessary. The sponsor will notify regulatory authorities as applicable.

#### 9.1.3 Confidentiality and Privacy

Participant confidentiality is strictly held in trust by the participating investigators, their staff, and the sponsor(s) and their agents. This confidentiality is extended to cover clinical information relating to participants, test results of biological samples and genetic tests, and all other information generated during participation in the study. No identifiable information concerning participants in the study will be released to any unauthorized third party. Participant confidentiality will be maintained when study results are published or discussed in conferences.

The study monitor, other authorized representatives of the sponsor, representatives of the Institutional Review Board (IRB), and/or regulatory agencies may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records

DMID/NIAID/NIH 

(office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical study site will permit access to such records.

All source records including electronic data will be stored in secured systems in accordance with institutional policies and federal regulations. All study data and research specimens that leave the site (including any electronic transmission of data) will be identified only by a coded number that cannot be linked to a participant.

As this research is funded by the NIH, it is covered by NIH policy which effectively issues the research a Certificate of Confidentiality. By this policy, researchers cannot be forced to disclose or provide, in any Federal, State, or local civil, criminal, administrative, legislative, or other proceeding, the name of such individual or any such information, document, or biospecimen that contains identifiable, sensitive information about the individual and that was created or compiled for purposes of the research, unless such disclosure or use is made with the consent of the individual to whom the information, document, or biospecimen pertains.

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects, like this study, or for information that must be released in order to meet the requirements of the FDA.

A Certificate of Confidentiality does not prevent the participant from voluntarily releasing information about themselves or their involvement in this research. If any person or agency obtains a written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

The Certificate of Confidentiality does not prevent the researchers from reporting without the participant's consent, information that would identify the participant as a participant in the research project regarding matters that must be legally reported including child and elder abuse, sexual abuse, or wanting to harm themselves or others.

The release of individual private information or specimens for other research will only occur if consent was obtained from the individual or the parent(s) or LAR of the adolescent participants to whom the information, document, or biospecimen pertains, *or* for the purposes of other research that the release is in compliance with applicable Federal regulations governing the protection of human participants in research.

### 9.1.4 Secondary Use of Stored Specimens and Data

### 9.1.4.1 Samples for Secondary Research

## **Repository Research Sample**

To participate in this study, participants and the parent or LAR of adolescent participants will be asked for consent for storage of samples for secondary use. Samples will be stored indefinitely at a DMID-designated storage facility. Each sample will be encoded (labeled) only with a barcode and a unique tracking number to protect participant confidentiality. Secondary research with coded

DMID/NIAID/NIH 

samples and data may occur, however, participant confidentiality will be maintained as described for this protocol. An IRB review of the secondary research using coded specimens is required.

Repository Research Samples, upon written request and approval from DMID and any approvals required by the site, may be shared for secondary research with investigators at the participating site, with researchers at other sites or other institutions, or company-designated research laboratories. The samples will not be sold or used directly for production of any commercial product. DMID will authorize shipment from the repository.

Reports from secondary research will not be kept in the participants' health records or shared with participants, unless required by law. Reports will not be sent to the specimen repository. The participant's decision for secondary research can be changed at any time by notifying the study doctors or nurses in writing. If the participant changes his/her decision, the samples will be destroyed if the samples have not been used for research or released for a specific research project.

## 9.1.4.2 Data Sharing for Secondary Research

Data from this study may be used for secondary research. Individual participant data collected during the trial that are sufficient to reanalyzed primary and secondary endpoints will be made available after deidentification. The SAP and Analytic Code will also be made available. This data will be available following publication, with no end date. The data will be made available to researchers who provide a methodologically sound proposal. The data will be available for any purpose outlined in the approved proposal. Proposals should be directed to DMID. To gain access, data requestors will need to sign a data access agreement. The investigator may request removal of data on individual study participants from NIH data repositories in the event that a research participant withdraws or changes his or her consent. However, data that have been distributed for approved research use cannot be retrieved.

#### 9.1.5 Key Roles and Study Governance

This is a multi-site clinical trial and as such, all study team members and roles are listed in the Manual of Procedures (MOP).

## 9.1.6 Safety Oversight

Safety oversight will be conducted by a DSMB that is an independent group of experts that monitors participant safety and advises DMID. The DSMB members will be separate and independent of study personnel participating in this trial and should not have scientific, financial or other conflict of interest related to this trial. The DSMB will consist of members with appropriate expertise to contribute to the interpretation of the data from this trial. The DSMB will operate under the rules of a DMID-approved charter that will be written at the organizational meeting of the DSMB. Procedures for DSMB reviews/meetings will be defined in the charter. Reports may include enrollment and demographic information and solicited and unsolicited AE/SAEs. The DSMB will review SAEs on a regular basis and ad hoc during this trial. The DMID Medical Monitor will be responsible for reviewing SAEs in real time.

For Stage 2 of the study, the DSMB will conduct the following reviews:

• Approximately 115 to 130 days after the study start. Given the planned 8 to 10-week enrollment period, and second dose of vaccine given on day 29, the window for review in

DMID/NIAID/NIH 

Stage 2 was extended. As such, the review will focus on AEs utilizing real time reports where able.

- Ad hoc meeting:
  - When trial-level halting criteria are met
  - o At the request of DMID to review a potential safety concern identified in the trial.
- Interim and final data will be shared with the DSMB, but the DSMB does not need to meet to review the final data.

Additional data may be requested by the DSMB. The DSMB may receive data in aggregate and presented by treatment arm. The DSMB may also be provided with expected and observed rates of the expected AEs in an unblinded fashion. As an outcome of each review/meeting, the DSMB will make a recommendation as to the advisability of proceeding with study interventions (as applicable), and to continue, modify, or terminate this trial.

The DSMB will operate under the rules of a DMID-approved charter that will be written at the organizational meeting of the DSMB. At this time, each data element that the DSMB needs to assess will be clearly defined. Procedures for DSMB reviews/meetings will be defined in the charter. The DSMB will review applicable data to include, but not limited to, study progress and participant, clinical, safety and safety related data. Reports may include enrollment and demographic information, medical history, concomitant medications, physical assessments, clinical laboratory values, dosing compliance, and solicited and unsolicited AE/SAEs.

DMID or the DSMB chair may convene the DSMB on an ad hoc basis according to protocol criteria or if there are immediate concerns regarding observations during the course of this trial. The DMID Medical Monitor is empowered to stop enrollment and study product administration if AEs that meet the halting criteria are reported. The DMID Medical Monitor will be responsible for reviewing SAEs in real time. The DSMB will review SAEs on a regular basis and ad hoc during this trial.

#### 9.1.7 Clinical Monitoring

Clinical site monitoring is conducted to ensure that the rights and well-being of trial participants are protected, that the reported trial data are accurate, complete, and verifiable. Clinical Monitoring ensures that the conduct of the trial is in compliance with the currently approved protocol/amendment(s), International Council for Harmonisation (ICH), Good Clinical Practice, and with applicable regulatory requirement(s) and sponsor requirements.

Monitoring for this study will be overseen by NIAID/DMID and conducted by NIAID/DMID contractors. Details of clinical site monitoring are documented in a Clinical Monitoring Plan (CMP). The CMP describes in detail who will conduct the monitoring, at what frequency monitoring will be done, at what level of detail monitoring will be performed, and the distribution of monitoring reports. Monitoring visits will include, but are not limited to, review of regulatory files, investigational product administration and accountability records, eCRFs, informed consent, parental permission and assent forms, medical and laboratory reports, site study storage records, training records, and protocol and GCP compliance. Site monitors will have access to each participating site, study personnel, and all study documentation according to the NIAID or DMID-approved site monitoring plan. Study monitors will meet with site principal investigators (or

DMID/NIAID/NIH 

designee) to discuss any problems and outstanding issues and will document site visit findings and discussions.

# 9.1.8 Quality Assurance and Quality Control

Quality control (QC) and quality assurance (QA) activities are essential to the safety of participants, and the reliability of study data. Each site participating in the study is responsible for integrating quality control checks throughout the study and implementing a QA Checklist or Clinical Quality Management Plan (CQMP). The site will conduct the following:

- 4. Routine internal QC and QA activities for the purposes of measuring, documenting and reporting study conduct, protocol adherence, human participants' protections, and reliability of the protocol-driven data collected.
- 5. Processes for addressing data quality issues (i.e., collecting, recording), and reporting findings in a timely manner.
- 6. Identify systemic issues (e.g., protocol or human participant protections non-compliance), and implementation and evaluation of Corrective and Preventative Action Plan (CAPA) procedures, if applicable.

#### 9.1.9 Data Handling and Record Keeping

#### 9.1.9.1 Data Collection and Management Responsibilities

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site investigator. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported. All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data.

#### 9.1.9.2 Data Coordinating Center / Biostatistician Responsibilities

The data coordinating center for this study will be responsible for data management, quality review, analysis, and reporting of the study data. Adverse events and medical history will be coded according to the MedDRA dictionary. Concomitant medications will be coded according to the WHO Drug dictionary. At the end of the study, a copy of all datasets including annotated case report forms and data dictionary will be provided to DMID.

A separate Study Data Standardization Plan (SDSP) will be developed which describes the technical recommendations for the submission of human study data and related information in a standardized electronic format throughout product development.

## 9.1.9.3 Data Capture Methods

Clinical research data, including, but not limited to, AE/SAEs, concomitant medications, medical history, physical assessments will be abstracted from the source documentation and/or collected on source document worksheet by study personnel then entered into an eCRFs via a 21 CFR Part 11-compliant internet data entry system provided by the study data coordinating center. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate.

DMID/NIAID/NIH 

The IND Sponsor is responsible for review of data collection tools and processes, and review of data and reports.

Study data will be collected on paper CRFs and then entered into the eCRF or data will be entered directly into the eCRF.

### 9.1.9.4 Study Record Retention

Study related records, including the regulatory file, study product accountability records, consent, parental permission and assent forms, participant source documents and electronic records should be maintained for a minimum period of 2 years following the date a marketing application is approved for the investigational product for the indication for which it is being investigated; or, if no application is to be filed or if the application is not approved for such indication, until 3 years after the investigation is discontinued and FDA is notified. These documents should be retained in compliance with all federal and local regulations and institutional policies; which may be longer. No records will be destroyed without the written consent of DMID. Consent and assent forms with specimen retention linked to identifiable specimens will be maintained for as long as the specimens remain in identifiable format, and a minimum of three years after use of the identifiable specimens in nonexempt human participant research.

#### 9.1.9.5 Source Records

Source data are all information, original records of clinical findings, observations, or other activities documented in a clinical trial necessary for the reconstruction and evaluation of the trial. Each participating site will maintain appropriate medical and research records for this trial, in compliance with ICH GCP, regulatory, and institutional requirements. Data recorded in the electronic case report form (eCRF) derived from source documents should be consistent with the data recorded on the source documents. Data entered directly into the eCRFs will be considered the source document. All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data.

Interview of participants is sufficient for obtaining medical history. Solicitation of medical records from the participant's primary care provider is not required.

#### 9.1.10 Protocol Deviations

A protocol deviation is any noncompliance with the clinical trial protocol, any process that is noted in the protocol and refers to details in the MOP, or GCP requirements.

The noncompliance may be either on the part of the participant, the investigator, or the study site staff. Following a deviation(s), corrective actions should be developed by the site and implemented promptly. All individual protocol deviations will be addressed in participant study records.

It is the responsibility of the site principal investigator and personnel to use continuous vigilance to identify and report deviations within five working days of identification of the protocol deviation, or within five working days of the scheduled protocol-required activity. All deviations

DMID/NIAID/NIH 

must be promptly reported to DMID per the protocol deviation reporting procedures. Protocol deviations must be sent to the local IRB/IEC per their guidelines. The site principal investigator and personnel are responsible for knowing and adhering to their IRB requirements.

#### 9.1.11 Publication and Data Sharing Policy

#### 9.1.11.1 Human Data Sharing Plan

All NIH protocols are required to have a Data Sharing Plan describe provisions for protecting the participants' privacy and the confidentiality of the data. This study will be conducted in accordance with the following publication and data sharing policies and regulations:

National Institutes of Health (NIH) Public Access Policy, which ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive <u>PubMed Central</u> upon acceptance for publication.

As of January 2018, all clinical trials supported by the NIH must be registered on ClinicalTrials.gov, no later than 21 days after the enrollment of the first participant. Results of all clinical trials supported by the NIH, generally, need to be submitted no later than 12 months following the primary completion date. As part of the result posting, a copy of this protocol and a copy of the Statistical Analysis Plan will be posted on ClinicalTrials.gov.

## 9.1.11.2 Genomic Data Sharing Plan

Not Applicable.

#### 9.1.11.3 Publication

This study will comply with the NIH Public Access Policy, which ensures that the public has access to the published results of NIH funded research. As such, the final peer-reviewed journal manuscripts will be accessible to the public on PubMed Central no later than 12 months after publication.

#### 9.1.12 Conflict of Interest Policy

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct of this trial. DMID has established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

#### 9.2 Additional Considerations

#### 9.2.1 Research Related Injuries

DMID/NIAID/NIH 

For any potential research related injury, the site principal investigator or designee will assess the participant. The site principal investigator should then determine if an injury occurred as a direct result of the tests or treatments that are done for this trial. As needed, referrals to appropriate health care facilities will be provided to the participant. No financial compensation will be provided by the NIAID, NIH, or the federal government to the participant, for any injury suffered due to participation in this trial.

#### **9.2.2 PREP Act**

The study vaccine and the efforts for this clinical trial are covered under the Public Readiness and Emergency Preparedness Act (PREP Act). The PREP Act applies under the terms of the PREP Act declaration in place for smallpox/orthopoxvirus countermeasures for activities conducted pursuant federal agreements (ref: federal programs www.federalregister.gov/documents/2015/12/09/2015-31092/smallpox-medicalcountermeasures-amendment). JYNNEOS is used under an IND for mpox pursuant to a federal agreement/program and is therefore covered under the PREP Act. The PREP Act covers persons (such as manufacturers, distributers, program planners, and other qualified persons who prescribe, administer or dispense study product) are immune from liability from the administration, or use of a covered countermeasure, such as JYNNEOS. The PREP Act provides immunity for covered persons from liability, unless the injury was caused by willful misconduct.

The PREP Act also established the Countermeasures Injury Compensation Program (CICP) to provide compensation for serious injuries or death that occur as the direct result of the administration or use of certain countermeasures. Any requests for compensation must be filed within one year of the administration or use of the covered countermeasure. Requests for Benefits must be made to the Health Resources and Services Administration's (HRSA) Countermeasures Injury Compensation Program (http://www.hrsa.gov/cicp/) by filing a Request for Benefits Form and all required medical records and supporting documentation. Additional information on filing a Request for Benefits is available on the CICP's website at http://www.hrsa.gov/cicp/. Compensation may then be available for reasonable and necessary medical benefits, lost wages and/or death benefits to eligible individuals for certain injuries in accordance with regulations published by the Secretary of HHS (found at 42 CFR part 110).

If an individual suffers a serious physical injury or death from the administration or use of a covered countermeasure in this study, the individual, the individual's legal or personal representative, the administrator/executor of a deceased individual's estate, or certain survivors may request benefits from the CICP. A serious physical injury means an injury that warranted hospitalization (whether or not the person was actually hospitalized) or that led to a significant loss of function or disability. The CICP is the payer of last resort. This means that it only covers expenses or provides benefits that other third-party payers (such as health insurance, the Department of Veterans Affairs, or Workers' Compensation programs) do not have an obligation to pay.

If the Secretary of HHS does not make a final determination on the individual's request within 240 days, or if the individual decides not to accept the compensation, the injured individual or his representative may pursue a tort claim in the US District Court for the District of Columbia, but only if the claim involves willful misconduct and meets the other requirements for suit under the

DMID/NIAID/NIH 

Protocol 22-0020
Appendix B
23 May 2024

PREP Act. Any award is reduced by any public or private insurance or worker's compensation available to the injured individual. Awards for non-economic damages, such as pain, suffering, physical impairment, mental anguish, and loss of consortium are also limited. If the individual accepts compensation, or if there is no willful misconduct, then the individual does not have a tort claim that can be filed in a US Federal or a State court.

## 10. REFERENCES

1. Pan American Health Organization. Mpox (monkeypox) outbreak - 2022. (https://www.paho.org/en/mpox-monkeypox-outbreak-2022#:~:text=On%2023%20July%202022%2C%20the,of%20International%20Concern %20(PHEIC)).

- 2. Centers for Disease Control and Prevention. 2022 Mpox Outbreak Global Map. (https://www.cdc.gov/poxvirus/monkeypox/response/2022/world-map.html).
- 3. Outbreak News Today. England: Monkeypox case confirmed, Patient had recent travel history from Nigeria. (https://outbreaknewstoday.com/england-monkeypox-case-confirmed-patient-had-recent-travel-history-from-nigeria-68610/).
- 4. McCollum AM, Damon IK. Human monkeypox. Clin Infect Dis 2014;58(2):260-7. DOI: 10.1093/cid/cit703.
- 5. Grant R, Nguyen LL, Breban R. Modelling human-to-human transmission of monkeypox. Bull World Health Organ 2020;98(9):638-640. DOI: 10.2471/BLT.19.242347.
- 6. Gong Q, Wang C, Chuai X, Chiu S. Monkeypox virus: a re-emergent threat to humans. Virol Sin 2022. DOI: 10.1016/j.virs.2022.07.006.
- 7. Rimoin AW, Mulembakani PM, Johnston SC, et al. Major increase in human monkeypox incidence 30 years after smallpox vaccination campaigns cease in the Democratic Republic of Congo. Proc Natl Acad Sci U S A 2010;107(37):16262-7. DOI: 10.1073/pnas.1005769107.
- 8. World Health Organization. Emergence of monkeypox in West Africa and Central Africa, 1970-2017. Wkly Epidemiol Rec 2018;93(11):125-32. (https://www.ncbi.nlm.nih.gov/pubmed/29546750).
- 9. Centers for Disease Control and Prevention. Multistate outbreak of monkeypox--Illinois, Indiana, and Wisconsin, 2003. MMWR Morb Mortal Wkly Rep 2003;52(23):537-40. (https://www.ncbi.nlm.nih.gov/pubmed/12803191).
- 10. Erez N, Achdout H, Milrot E, et al. Diagnosis of Imported Monkeypox, Israel, 2018. Emerg Infect Dis 2019;25(5):980-983. DOI: 10.3201/eid2505.190076.
- 11. Yong SEF, Ng OT, Ho ZJM, et al. Imported Monkeypox, Singapore. Emerg Infect Dis 2020;26(8):1826-1830. DOI: 10.3201/eid2608.191387.
- 12. Rao AK, Schulte J, Chen TH, et al. Monkeypox in a Traveler Returning from Nigeria Dallas, Texas, July 2021. MMWR Morb Mortal Wkly Rep 2022;71(14):509-516. DOI: 10.15585/mmwr.mm7114a1.
- 13. Vaughan A, Aarons E, Astbury J, et al. Human-to-Human Transmission of Monkeypox Virus, United Kingdom, October 2018. Emerg Infect Dis 2020;26(4):782-785. DOI: 10.3201/eid2604.191164.
- 14. Hobson G, Adamson J, Adler H, et al. Family cluster of three cases of monkeypox imported from Nigeria to the United Kingdom, May 2021. Euro Surveill 2021;26(32). DOI: 10.2807/1560-7917.ES.2021.26.32.2100745.
- 15. Mauldin MR, McCollum AM, Nakazawa YJ, et al. Exportation of Monkeypox Virus From the African Continent. J Infect Dis 2022;225(8):1367-1376. DOI: 10.1093/infdis/jiaa559.
- 16. Yinka-Ogunleye A, Aruna O, Dalhat M, et al. Outbreak of human monkeypox in Nigeria in 2017-18: a clinical and epidemiological report. Lancet Infect Dis 2019;19(8):872-879. DOI: 10.1016/S1473-3099(19)30294-4.

DMID/NIAID/NIH 

17. Durski KN, McCollum AM, Nakazawa Y, et al. Emergence of Monkeypox - West and Central Africa, 1970-2017. MMWR Morb Mortal Wkly Rep 2018;67(10):306-310. DOI: 10.15585/mmwr.mm6710a5.

- 18. Constantino AK. Health officials confirm first U.S. case of monkeypox virus this year in Massachusetts. CNBC Health & Science, 2022.
- 19. Department of Health and Human Services. Determination that a public health emergency exists. (https://aspr.hhs.gov/legal/PHE/Pages/monkeypox-4Aug22.aspx).
- 20. Vollmar J, Arndtz N, Eckl KM, et al. Safety and immunogenicity of IMVAMUNE, a promising candidate as a third generation smallpox vaccine. Vaccine 2006;24(12):2065-70. DOI: 10.1016/j.vaccine.2005.11.022.
- 21. Frey SE, Wald A, Edupuganti S, et al. Comparison of lyophilized versus liquid modified vaccinia Ankara (MVA) formulations and subcutaneous versus intradermal routes of administration in healthy vaccinia-naive subjects. Vaccine 2015;33(39):5225-34. DOI: 10.1016/j.vaccine.2015.06.075.
- 22. Wilck MB, Seaman MS, Baden LR, et al. Safety and immunogenicity of modified vaccinia Ankara (ACAM3000): effect of dose and route of administration. J Infect Dis 2010;201(9):1361-70. DOI: 10.1086/651561.
- World Health Organization. Multi-country outbreak of mpox, External situation report #11. Emergency Situational Update. Geneva, Switzerland: December 1, 2022. (https://www.who.int/publications/m/item/multi-country-outbreak-of-mpox--external-situation-report--11---1-december-2022).
- 24. Hennessee I SV, McArdle CE, et al. . Epidemiologic and Clinical Features of Children and Adolescents Aged <18 Years with Monkeypox United States, May 17–September 24, 2022. MMWR Morb Mortal Wkly Rep 2022(71):1407–1411. DOI: http://dx.doi.org/10.15585/mmwr.mm7144a4.
- 25. Hutin W, R. J., Malfait, P., Pebody, R., Loparev, V. N., Ropp, S. L., Rodriguez, M., Knight, J. C., Tshioko, F. K., Khan, A. S., Szczeniowski, M. V., & Esposito, J. J. Outbreak of Human Monkeypox, Democratic Republic of Congo, 1996 to 1997. . Emerging Infectious Diseases 2001;7(3):434–438. DOI: https://doi.org/10.3201/eid0703.017311.
- 26. Ježek Z, Szczeniowski M, Paluku KM, Mutombo M. Human Monkeypox: Clinical Features of 282 Patients. The Journal of Infectious Diseases 1987;156(2):293-298. DOI: 10.1093/infdis/156.2.293.
- 27. US Food and Drug Administration. Summary Basis for Regulatory Action (https://www.fda.gov/media/131802/download).
- 28. Overton ET, Lawrence SJ, Wagner E, et al. Immunogenicity and safety of three consecutive production lots of the non replicating smallpox vaccine MVA: A randomised, double blind, placebo controlled phase III trial. PLoS One 2018;13(4):e0195897. DOI: 10.1371/journal.pone.0195897.
- 29. US Food and Drug Administration. Fact Sheet for Healthcare Providers Administering Vaccine: Emergency Use Authorization of JYNNEOS (Smallpox and Monkeypox Vaccine, Live, Non-replicating) for Prevention of Monkeypox Disease in Individuals Determined to Be at High Risk for Monkeypox Infection. 2022.
- 30. Elizaga ML VS, Marovich MA, Sato AH, Lawrence DN, Chaitman BR, Frey SE, Keefer MC; MVA Cardiac Safety Working Group. Prospective surveillance for cardiac adverse

DMID/NIAID/NIH 

- events in healthy adults receiving modified vaccinia Ankara vaccines: a systematic review. . PLoS One 2013;8(1):e54407. DOI: 10.1371/journal.pone.0054407.
- 31. Scriba TJ, Tameris, M., Mansoor, N., Smit, E., van der Merwe, L., Isaacs, F., Keyser, A., Moyo, S., Brittain, N., Lawrie, A., Gelderbloem, S., Veldsman, A., Hatherill, M., Hawkridge, A., Hill, A.V.S., Hussey, G.D., Mahomed, H., McShane, H. and Hanekom, W.A., . Modified vaccinia Ankara-expressing Ag85A, a novel tuberculosis vaccine, is safe in adolescents and children, and induces polyfunctional CD4+ T cells. . Eur J Immunol 2010;40:279-290. (https://doi.org/10.1002/eji.200939754).
- 32. Anywaine Z BH, Anzala O, Mutua G, Sirima SB, Eholie S, et al. . Safety and immunogenicity of 2-dose heterologous Ad26.ZEBOV, MVA-BN-Filo Ebola vaccination in children and adolescents in Africa: A randomised, placebo-controlled, multicentre Phase II clinical trial. PLoS Medicine 2022;19(1):e1003865. (https://doi.org/10.1371/journal.pmed.1003865).
- 33. Afolabi MO ID, Manno D, et al. Safety and immunogenicity of the two-dose heterologous Ad26.ZEBOV and MVA-BN-Filo Ebola vaccine regimen in children in Sierra Leone: a randomised, double-blind, controlled trial. Lancet Infect Dis 2022;22:110-122.
- 34. Suter M, Meisinger-Henschel C, Tzatzaris M, et al. Modified vaccinia Ankara strains with identical coding sequences actually represent complex mixtures of viruses that determine the biological properties of each strain. Vaccine 2009;27(52):7442-50. DOI: 10.1016/j.vaccine.2009.05.095.
- 35. Stittelaar KJ, Kuiken T, de Swart RL, et al. Safety of modified vaccinia virus Ankara (MVA) in immune-suppressed macaques. Vaccine 2001;19(27):3700-9. DOI: 10.1016/s0264-410x(01)00075-5.
- 36. Overton ET, Stapleton J, Frank I, et al. Safety and Immunogenicity of Modified Vaccinia Ankara-Bavarian Nordic Smallpox Vaccine in Vaccinia-Naive and Experienced Human Immunodeficiency Virus-Infected Individuals: An Open-Label, Controlled Clinical Phase II Trial. Open Forum Infect Dis 2015;2(2):ofv040. DOI: 10.1093/ofid/ofv040.
- 37. Greenberg RN, Overton ET, Haas DW, et al. Safety, immunogenicity, and surrogate markers of clinical efficacy for modified vaccinia Ankara as a smallpox vaccine in HIV-infected subjects. J Infect Dis 2013;207(5):749-58. DOI: 10.1093/infdis/jis753.
- 38. Overton ET, Lawrence SJ, Stapleton JT, et al. A randomized phase II trial to compare safety and immunogenicity of the MVA-BN smallpox vaccine at various doses in adults with a history of AIDS. Vaccine 2020;38(11):2600-2607. DOI: 10.1016/j.vaccine.2020.01.058.
- 39. von Sonnenburg F, Perona P, Darsow U, et al. Safety and immunogenicity of modified vaccinia Ankara as a smallpox vaccine in people with atopic dermatitis. Vaccine 2014;32(43):5696-702. DOI: 10.1016/j.vaccine.2014.08.022.
- 40. Greenberg RN, Hurley MY, Dinh DV, et al. A Multicenter, Open-Label, Controlled Phase II Study to Evaluate Safety and Immunogenicity of MVA Smallpox Vaccine (IMVAMUNE) in 18-40 Year Old Subjects with Diagnosed Atopic Dermatitis. PLoS One 2015;10(10):e0138348. DOI: 10.1371/journal.pone.0138348.
- 41. Cassimatis DC, Atwood JE, Engler RM, Linz PE, Grabenstein JD, Vernalis MN. Smallpox vaccination and myopericarditis: a clinical review. J Am Coll Cardiol 2004;43(9):1503-10. DOI: 10.1016/j.jacc.2003.11.053.

DMID/NIAID/NIH 

42. Department of Health and Human Services. 46.110 Expedited review procedures for certain kinds of research involving no more than minimal risk, and for minor changes in approved research.

(https://www.hhs.gov/ohrp/sites/default/files/ohrp/sachrp/mtgings/2013%20March%20Mtg/approvedexpeditedreviewcategories.pdf).

- 43. Sexson Tejtel SK, Munoz FM, Al-Ammouri I, et al. Myocarditis and pericarditis: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine 2022;40(10):1499-1511. DOI: 10.1016/j.vaccine.2021.11.074.
- 44. Pittman PR, Hahn M, Lee HS, et al. Phase 3 Efficacy Trial of Modified Vaccinia Ankara as a Vaccine against Smallpox. N Engl J Med 2019;381(20):1897-1908. DOI: 10.1056/NEJMoa1817307.
- 45. European Centre for Disease Prevention and Control. Outbreak of mpox caused by Monkeypox virus clade I in the Democratic Republic of the Congo. ECDC. (https://www.ecdc.europa.eu/en/news-events/outbreak-mpox-caused-monkeypox-virus-clade-i-democratic-republic-congo#:~:text=In%20the%20current%20epidemiological%20reports,in%20the%20DRC %20%5B6%5D).

DMID/NIAID/NIH 